# **Ablynx**

# ALX0061-C204

A Phase II Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-range Finding Study to Evaluate the Safety and Efficacy of ALX-0061 Administered Subcutaneously in Subjects with Moderate to Severe Active Systemic Lupus Erythematosus

# 28FEB2018

Statistical Analysis Plan

Final Version 1.0



# **TABLE OF CONTENTS**

| LIS | T OF A | BREVIATIONS | 6 |
|-----|-----------------|--------------------------------------------|----|
| 1 | INT | RODUCTION | 9 |
| 2 | ОВЈ | ECTIVES | 10 |
| 2. | 1 PRIM | IARY OBJECTIVE | 10 |
| 2. | | ONDARY OBJECTIVES | |
| 3 | INV | ESTIGATIONAL PLAN | 10 |
| 3. | 1 OVE | RALL STUDY DESIGN AND PLAN | 10 |
| | 3.1.1 | Sample Size | |
| | 3.1.2 | Blinding and Unblinding | |
| | 3.1.2. | | |
| | 3.1.2. | | |
| _ | 3.1.2. | | |
| | | DY ENDPOINTS | |
| | 3.2.1<br>3.2.2 | Primary Endpoint | |
| | | Secondary Endpoints | |
| 4 | GEN | ERAL STATISTICAL CONSIDERATIONS | 16 |
| 4. | 1 ANA | LYSIS POPULATIONS | 19 |
| | 4.1.1 | All Screened Population | 19 |
| | 4.1.2 | All Randomized Population | |
| | 4.1.3 | Modified Intent-to-Treat (mITT) Population | |
| | 4.1.4 | Per Protocol (PP) Population | |
| | 4.1.5 | Safety Population | |
| 5 | SUB | JECT DISPOSITION | 23 |
| 5. | 1 DISF | POSITION | 23 |
| 5. | 2 ANA | LYSIS POPULATIONS | 24 |
| 5. | 3 Pro | TOCOL DEVIATIONS | 24 |
| 6 | DEM | OGRAPHICS AND BASELINE CHARACTERISTICS | 24 |
| 6. | 1 DEM | OGRAPHICS | 24 |
| 6. | | ELINE DISEASE CHARACTERISTICS | |
| 6. | | ACCO USAGE | |
| 6. | | ical History | |
| 6. | 5 ADD | ITIONAL SCREENING/BASELINE ASSESSMENTS | 26 |
| 7 | TRE | ATMENTS AND MEDICATIONS | 26 |
| 7. | 1 <b>D</b> DTC | R AND CONCOMITANT MEDICATIONS | 26 |
| | | Prior Medications | |
| | 7.1.2 | Concomitant Medications | |
| 7. | – . – | DY TREATMENTS | |
| 8 | | CACY ANALYSIS | |
| 8. | 1 PRIM<br>8.1.1 | IARY EFFICACY ENDPOINT | |
| | 8.1.1<br>8.1.2 | Assumption Testing | |
| | 8.1.2<br>8.1.3 | Sensitivity Analysis | |
| | 8.1.4 | Subgroup Analysis | |
| | | DNDARY EFFICACY ENDPOINTS | |
| | 8.2.1 | mBICLA | |
| | 8.2.2 | BICLA | |
| | 8.2.3 | SRI | 36 |

| 8.2.4 | | |
|---|---|---|
| 8.2.5 | | |
| 8.2.6 | | |
| 8.2.7<br>8.2.8 | · | |
| 8.2.9 | | 38 |
| 8.2.1 | 0 BILAG-2004 Systems Tally | 38 |
| 8.2.1 | · | |
| 8.2.1. | | |
| 8.2.1. | | 39 |
| 8.2.1 | 4 Treatment Failure | 40 |
| 8.2.1 | | |
| 8.2.1 | | |
| 8.2.1 | | |
| 8.2.1 | | |
| 8.2.1<br>8.2.2 | | |
| 8.2.2 | | |
| 8.2.2. | | |
| 9 SA | AFETY ANALYSIS | 42 |
| 9.1 A | DVERSE EVENTS | |
| 9.1.1 | Incidence of Adverse Events | |
| 9.1.2 | and the state of t | |
| 9.1.3 | | |
| 9.1.4 | | |
| 9.1.5 | | |
| 9.1.6<br>9.1.7 | | |
| | LINICAL LABORATORY EVALUATIONS | |
| 9.2.1 | Haematology, Blood Chemistry, Lipid Profile and Coagulation | |
| 9.2.2 | | |
| 9.2.3 | | |
| 9.2.4 | | |
| 9.2.5 | INR | 47 |
| 9.2.6 | | |
| | ITAL SIGN MEASUREMENTS | |
| | HYSICAL EXAMINATION | |
| | LECTROCARDIOGRAM | |
| 9.6 O<br>9.6.1 | THER SAFETY DATA Tuberculosis Assessment | |
| 9.6.2 | | |
| | , | |
| 10 PH | HARMACOKINETICS (PK) | 49 |
| 11 PH | HARMACODYNAMICS (PD) | 51 |
| 12 IM | MUNOGENICITY | 51 |
| | VAILABLE DATA | |
| 12.1. | | |
| 12.1 | | |
| | UBGROUP ANALYSES | |
| 13 IN | ITERIM ANALYSIS | 55 |
| 14 D/ | ATA AND SAFETY MONITORING BOARD (DSMB) | 55 |
| 15 CH | HANGES IN THE PLANNED ANALYSIS | 55 |
| 16 RF | FERENCES | 56 |

| <b>17</b> | APPENDICES57 | 7 |
|---|---|---|
| 17 | '.1 Schedule of Study Procedures <sup>a</sup> | 58 |
| 17 | '.2 Dosing Schedule | 51 |
| 17 | '.3 BILAG-2004 | |
| _ | 17.3.1 BILAG-2004 Improvement (overall and individual): | <i>53</i> |
| _ | 17.3.2 BILAG-2004 Total Score: | |
| _ | 17.3.3 BILAG-2004 Systems Tally: | |
| - | 17.3.4 BILAG-2004 Flare Index: | 54 |
| - | 17.3.5 BILAG-2004 Scoring System: | 54 |
| | 17.3.5.1 Imputation of missing items | j |
| | 17.3.5.2 Constitutional | |
| | 17.3.5.3 Mucocutaneous | |
| | 17.3.5.4 Neuropsychatric | |
| | 17.3.5.5 Musculoskeletal | |
| | 17.3.5.6 Cardiorespiratory | |
| | 17.3.5.7 Gastrointestinal | |
| | 17.3.5.8 Ophthalmic | |
| | 17.3.5.9 Renal | |
| | 17.3.5.10 Hematological | |
| | '.4 SLEDAI-2K Scoring System | |
| | '.5 Treatment Failure Derivation Algorithm | |
| | 17.5.1 Cut-off date | |
| | 17.5.2 New / Increased dose Determination | <del>30</del> |
| | 17.5.3 Selection of Immunosuppressive Drugs: | 31 |
| | 17.5.4 Selection of anti-malarials Drugs | <del>3</del> 1 |
| | '.6 BILAG BASED COMPOSITE LUPUS ASSESSMENT (BICLA) | |
| | 7.7 SLE RESPONDER INDEX (SRI) | |
| | '.8 SELECTION OF NSAIDS | |
| | .9 SELECTION OF STEROIDS DRUGS AND DRUG EQUIVALENCE | |
| | '.10 Medical Outcome Survey Short Form 36 (SF-36) | |
| | .1128-JOINT COUNT | |
| | .12CLASI QUESTIONNAIRE | |
| | .13SLICC Score | |
| | .14Laboratory Parameters Precision Levels | |
| | '.15 Date Imputation (Medications and AEs) | |
| | 17.15.1 Adverse Events | |
| | 17.15.2 Prior/Concomitant Medications/Procedures | |
| 17 | 1.16 ANALYSIS VISIT / VISIT WINDOW | 96 |
| | '.17 Example of R code (MCP-Mod): | |
| | '.19Listing display/contents | |
| | .20CTCAE GRADES | |
| | .21 WORST ON-TREATMENT DEFINITION 1. '.22 STRATIFIED CMH 95%CI AND P-VALUE | |
| Ι/ | .223 KATIFIED CMIT 3370CI AND P-VALUE | <b>4</b> 7 |

# **LIST OF TABLES**

| Table 4-1: | Treatment Labels | . 17 |
|---|---|---|
| Table 4-2: | Actual Treatment Group | . 23 |
| Table 12-1: | ADA, mADA and Overall Subject Classification | |
| Table 12-2: | NAb Assay Classification | |
| Table 17-1: | Dosing schedule for Group 1 | |
| Table 17-2: | Dosing schedule for Group 2 | 61 |
| Table 17-3: | Dosing schedule for Group 3 | 62 |
| Table 17-4: | Dosing schedule for Group 4 | 62 |
| Table 17-5: | Dosing schedule for Group 5 | 62 |
| Table 17-6: | Musculoskeletal, Ophthalmic and Neuropsychiatric system organs - | |
| T 11 47 7 | Imputed values for Visitx | |
| Table 17-7: | | |
| T 11 47 0 | for Visit <sub>x</sub> | |
| | Prednisone Equivalence Table | |
| | Laboratory Precision Levels | |
| | Visit Windows (Post-Baseline) | |
| Table 17-11: | NCI CTCAE Grades | 127 |
| Table 17-12: | Worst on-treatment | 128 |
| | LIST OF FIGURES | |
| Figure 3-1: | Overview of the design of Study ALX0061-C204 | . 10 |
| Figure 8-1: | Graphical Representation of the Candidate models | 32 |

### **List of Abbreviations**

aCL anti-cardiolipin

ACR American College of Rheumatology

ADA Anti-drug antibodies

AE Adverse event

AESI Adverse event of Special Interest
AIC Akaike Information Criterion
ALT Alanine Aminotransferase
ANA Anti-nuclear Antibodies
ANCOVA Analysis of Covariance
AQL Above Quantification Limit

AST Aspartate Aminotransferase
ATC Anatomical Therapeutic Chemical

 $\beta_2$ -GPI anti- $\beta_2$ -glycoprotein I

BICLA BILAG-based composite lupus assessment

BILAG British Isles Lupus Assessment Group

BQL Below Quantification Limit
BST BILAG-2004 systems tally

CI Confidence interval

CLASI Cutaneous lupus erythematosus disease area and severity index

CMH Cochran-Mantel-Haenszel
CNS Central Nervous System

CRF Case Report Form
CRP C-reactive protein
CV Coefficient of variation
DM Data Management

DSMB Data and Safety Monitoring Board

ECG Electrocardiogram

eGFR Estimated glomerular filtration rate

EQ Equivocal

GGT Gamma Glutamyltransferase
HEENT Head, Ears, Eyes, Nose, Throat
HIV Human Immunodeficiency Virus

ICH International Council for Harmonisation

IL-6 Interleukin-6

INR International Normalized Ratio
IWRS Interactive Web Response System

Ablynx Statistical Analysis Plan, Final Version 1.0 ALX0061-C204 Date Issued: 28FEB2018

LA Lupus anti-coagulant

LOCF Last Observation Carried Forward

MACE Major Adverse Cardiac Events

mADA modified anti-drug antibodies

mBICLA modified BILAG-based composite lupus assessment

MCP-Mod Multiple Comparison Procedure – Modelling

MRD Minimal Required Dilution

MedDRA Medical Dictionary for Regulatory Activities

mITT modified Intent-to-Treat mSFI mSLEDAI-2K Flare Index

mSLEDAI-2K | modified systemic lupus erythematosus disease activity index 2000

mSRI modified systemic lupus erythematosus responder index

NAb Neutralizing antibody

NA Not Analyzed NC Not Calculable

NCI CTCAE

National Cancer Institute Common Terminology Criteria for Adverse

**Events** 

NRI Non-response imputation

NSAID Non-steroidal anti-inflammatory drug

PD Pharmacodynamics

PGA Physician's global assessment

PK Pharmacokinetics

PP Per Protocol
PT Preferred term
q2w Every 2 weeks
q4w Every 4 weeks

QTcB QT corrected Bazett Interval
QTcF QT corrected Fridericia Interval

RA Rheumatoid arthritis
s.c. Subcutaneous(ly)
SAE Serious adverse event
SAP Statistical analysis plan

sBST Simplified BILAG-2004 systems tally

SD Standard deviation

SDTM Study Data Tabulation Model

SE Standard error

SF-36 Short Form (36) Health Survey
SI International Standard Unit

Ablynx Statistical Analysis Plan, Final Version 1.0 ALX0061-C204 Date Issued: 28FEB2018

SIL-6R Soluble interleukin-6 receptor SLE Systemic lupus erythematosus

SLEDAI-2K Systemic lupus erythematosus disease activity index 2000

SLICC Systemic Lupus International Collaborating Clinics

SMQs Standardized MedDRA Queries

SOC System Organ Class

SRI Systemic lupus erythematosus responder index

TB Tuberculosis

TE Treatment Emergent

TEAE Treatment-emergent adverse events

TTP Thrombotic Thrombocytopenic Purpura

uMCP-1 Monocyte Chemotactic Protein-1 in urine

uCr urine creatinine

VAS Visual Analogue Scale

WHO-DD World Health Organization Drug Dictionary

#### 1 Introduction

Systemic lupus erythematosus (SLE) is a clinically heterogeneous disease that affects multiple organs, with the most common manifestations ranging from rash, fatigue and mucocutaneous and musculoskeletal conditions, to more severe renal and neurological manifestations. SLE is characterized by periods of active disease, alternated with temporary remission and relapses.

ALX-0061 has been developed by Ablynx as a new compound neutralizing proinflammatory activity in the Interleukin-6 (IL-6) pathway. Based on its mode of action, ALX-0061 is currently in development for the treatment of autoimmune diseases such as SLE and rheumatoid arthritis (RA).

This study is intended to evaluate the efficacy and safety of different dose regimens of ALX-0061 administered subcutaneously (s.c.) on top of standard of care to subjects with moderate to severe active, seropositive SLE. The selection of the doses used in this study was based on the results of study ALX0061-C102 in healthy volunteers (for pharmacokinetics [PK], safety and tolerability), study ALX-0061-1.1/10 in RA patients (for efficacy and pharmacological activity), and the exposure levels measured in preclinical toxicology studies (for safety margin calculation).

As this is an add-on therapy study, all subjects (including subjects in the placebo group) will receive standard of care treatment for SLE in line with their severity of disease and according the Investigator's clinical practice. Analysis of the placebo group will be of value in the assessment of whether or not any abnormalities observed were due to ALX-0061 or to study procedures, and will allow statistical comparison of efficacy between ALX-0061 and placebo.

This statistical analysis plan (SAP) has been created based on study Protocol version 3.0 dated 03-May-2016 and following the International Council for Harmonisation (ICH) quidelines.

# 2 Objectives

### 2.1 Primary objective

To assess the efficacy and safety of different dose regimens of ALX-0061 administered s.c. to subjects with moderate to severe active, seropositive SLE compared to placebo.

### 2.2 Secondary objectives

To assess the PK, pharmacodynamics (PD), immunogenicity, flare rate, steroid reduction and health-related quality of life, with different dose regimens of ALX-0061.

# 3 Investigational Plan

# 3.1 Overall Study Design and Plan

This is a multicenter, randomized, double-blind, placebo-controlled, dose-range finding Phase II study of ALX-0061 administered s.c. on top of standard of care, in subjects with moderate to severe active, seropositive SLE. Approximately 300 subjects will be randomized into 5 treatment groups in a 1:1:1:1:1 ratio (Placebo, ALX-0061 75 mg every 4 weeks [q4w], 150 mg q4w, 150 mg every 2 weeks [q2w] and 225 mg q2w). An overview of the study design is included in Figure 3-1.



Figure 3-1: Overview of the design of Study ALX0061-C204

At the Screening Visit, informed consent will be obtained from all subjects who are deemed potentially eligible for the study according to the protocol-specified inclusion and exclusion criteria, for enrolment in the study.

After obtaining oral and written informed consent, subjects will be screened according to the inclusion and exclusion criteria and will receive a unique subject identification number, assigned by Interactive Web Response System (IWRS).

After receipt of the approval by the eligibility review committee (see Protocol Section 3.4.1.1), subjects can be randomized.

At randomization, subjects will be reassessed and, if they meet the specified entry criteria, subjects will be allocated in a randomization to 1 of 5 treatment groups in a 1:1:1:1:1 ratio, and will receive a randomization number just prior to dosing according

to the randomization scheme. Randomization will be stratified by geographic region (North America, Latin America, Europe and Asia-Pacific).

Subjects will receive one of the following treatments:

- Placebo,
- ALX-0061 75 mg q4w,
- ALX-0061 150 mg q4w,
- ALX-0061 150 mg q2w,
- ALX-0061 225 mg q2w.

ALX-0061 s.c. or placebo s.c. injections, as applicable, will be administered via single-use pre-filled syringe by an appropriately licensed and authorized health professional.

At each administration, the subject will receive 2 s.c. injections in succession at a different quadrant in the abdominal region. As injections are to be performed q2w, the injections can be performed in an abdominal quadrant of choice. The dosing combinations are shown in Section 17.2.

Subjects and investigational staff will be blinded for treatment and dose. Subjects will be followed for efficacy through Week 48 and for safety through Week 58. Visits are planned every 2 weeks from randomization to Week 48 and then at follow-up at Week 58 [12 weeks after the last dose; last dose is at Week 46].

The schedule of assessment is included in Section 17.1.

#### 3.1.1 Sample Size

Up to approximately 300 subjects will be randomized over 5 treatment arms in a 1:1:1:1:1 ratio. Randomization will be stratified by geographic region.

Simulations were performed to evaluate the power of detecting a significant dose-response relationship, i.e., whether changes in ALX-0061 dose regimen lead to significant changes in mBICLA response rate at Week 24 by using the MCP-Mod methodology [1]. A set of 5 plausible candidate models containing both monotonous and non-monotonous exposure-response shapes was defined. For these models an estimated placebo response rate of 25%, and a difference in response rate between the ALX-0061 dose regimen with the largest response rate and placebo of 25% was assumed, taking into account a discontinuation rate of 15% (homogeneous over treatment arms). With this methodology a sample size of 60 subjects per arm will provide at least 85% power at a family-wise 5% significance level.

### 3.1.2 Blinding and Unblinding

### 3.1.2.1 Study Drug Administration Blinding

Since the 225 mg dose of ALX-0061 exceeds the volume that can be administered in a single injection, the placebo and ALX-0061 groups will have 2 different combinations of injections to ensure the double-blinded design. All subjects are to receive 2 injections in succession (syringe A containing 1 mL and syringe B containing 0.5 mL) at each dosing day, every 2 weeks. Syringes containing ALX-0061 or placebo are a visual match. When containing the active product, syringes A and B contain 150 mg and 75 mg of ALX-0061, respectively.

Therefore, there will be a total of 5 dosing combinations in the study, with 4 possible active dose regimens. These dosing combinations are shown in Section 17.2.

In order to protect the integrity of the data, ALX-0061 treatment assignment will be kept blinded for investigative sites, site monitors, subjects, vendors and PPD/Sponsor until the final database lock (including the Follow-up Visit 12 weeks after the last dosing).

Identification of Sponsor and vendor personnel who will have access to the unblinded data before final database lock, will be documented prior to their unblinding. The number of Sponsor personnel having access to the unblinded data will be limited.

### 3.1.2.2 Blinding of Potentially Unblinding Parameters

Given the pronounced effect of an anti-IL-6 compound on the acute phase reactants, the results of CRP and fibrinogen tests performed by the central laboratory will not be communicated to the investigational sites and PPD/Sponsor until after database lock and unblinding (unless in case of an alert). If an investigational site requests these data, it will be provided after the end of the study.

If the clinical condition of the subject warrants knowledge of the values of CRP or fibrinogen in order to provide appropriate medical care, the Investigator can request these assessments to be performed locally.

PK concentrations will be determined within Ablynx by dedicated personnel and will not be communicated to the investigational sites, PPD and Sponsor personnel (except for dedicated study personnel) until after the database lock and unblinding. The dedicated study personnel performing the analysis will be documented in the bioanalytical plan and unblinding forms according to Sponsor procedures. PK concentrations will be transferred to the immunogenicity study personnel to allow correct immunogenicity subject classification. The dedicated study personnel will also be documented in the unblinding forms according to Sponsor procedures.

sIL-6R concentrations will be determined within Eurofins and will not be communicated to the investigational sites and PPD/Sponsor until after the database lock and unblinding.

# 3.1.2.3 Emergency Unblinding

Code-breaking and unblinding in the event of medical emergencies can be done by the Investigator via the IWRS, which will be accessible 24 hours per day/7 days per week.

Unblinding by the Investigator should occur only in the event of an AE for which it is necessary to know the study treatment to determine an appropriate course of therapy for the subject.

If the Investigator must identify the treatment assignment of an individual subject, the Investigator or qualified designee is to call the IWRS. Unblinding performed by the IWRS at the request of the Investigator is to be reported to the Sponsor. When possible, the Investigator must first discuss options with the Medical Monitor.

Subjects for whom the code has been broken by the Investigator will have to discontinue treatment and all efforts must be made to conduct the Early Termination Visit and Follow-up Visit.

# 3.2 Study Endpoints

#### 3.2.1 Primary Endpoint

The primary endpoint is the percentage of subjects in the mITT population who achieved a response at Week 24 according to the modified British Isles Lupus Assessment Group (BILAG)-based Composite Lupus Assessment (mBICLA) score, see Section 17.6. Handling of missing data is described in Section 8.1.

### 3.2.2 Secondary Endpoints

The following endpoints are secondary endpoints (see Section 8.2, Section 17.3 to Section 17.12 for more details):

### **Efficacy Endpoints:**

- Composite endpoint mBICLA response rate at Week 4, Week 8, Week 12, Week 16, Week 20, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Composite endpoint BICLA response rate at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Composite endpoint Systemic lupus erythematosus Responder Index (SRI) response rate at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Composite endpoint SRI-5 response rate at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48
- Composite endpoint SRI-6 response rate at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Composite endpoint SRI-7 response rate at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Composite endpoint SRI-8 response rate at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48
- Composite endpoint modified SRI (mSRI) response rate at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Composite endpoint mSRI-5 response rate at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Composite endpoint mSRI-6 response rate at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Composite endpoint mSRI-7 response rate at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.

- Composite endpoint mSRI-8 response rate at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Actual and change from Baseline values in Systemic Lupus Erythematosus Disease activity index 2000 (SLEDAI-2K) score at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Actual and change from Baseline values in modified SLEDAI-2K (mSLEDAI-2K) score at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Number and percent of subjects with BILAG-2004 improvement (normal and enhanced) from Baseline at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Actual and change from Baseline values in BILAG-2004 Total Score at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Normal improvement in individual organ systems of the BILAG-2004 at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Number of BILAG-2004 systems with active/worsening disease, improving disease, or persistent minimal or no activity compared to previous visit (BILAG-2004 systems tally) at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Actual and change from Baseline values in Physician's Global Assessment (PGA) at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Actual and change from Baseline values in patient's global assessment at Week 24 and Week 48.
- Actual values and change from Baseline in efficacy laboratory parameters:
  - Proteinuria (as measured by spot urine protein to creatinine ratio) and estimated glomerular filtration rate (eGRF) at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
  - Serum creatinine at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48 and Follow-up.
- Shift from Baseline in urine sediment (present/not present) at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Proportion of treatment failures at Week 24 and at Week 48.
- Severe flare rate at Week 24 and at Week 48 using the following indexes:
  - BILAG-2004 Flare Index
  - mSLEDAI-2K Flare Index (mSFI)
- Mild/moderate flare rate at Week 24 and at Week 48 using the following indexes:
  - o BILAG-2004 Flare Index
  - o mSFI

- Actual values, change from baseline and percent change from Baseline in Prednisone Equivalent Total Daily Dose at Week 12, Week 24 and Week 48.
- Percent of subjects whose prednisone equivalent dose was >7.5 mg/day at Baseline and reduced to ≤7.5 mg/day during Weeks 40–48 without experiencing a mSFI-defined or BILAG-2004-defined flare (regardless of the severity of flare) after the first prednisone equivalent dose decrease.
- Percent of subjects whose prednisone equivalent dose was >7.5 mg/day at Baseline and reduced to ≤7.5 mg/day during Weeks 40-48 without experiencing a mSFI-defined or BILAG-2004-defined severe flare after the first prednisone equivalent dose decrease.
- Percent of subjects who are able to discontinue prednisone (or equivalent) before
  or on Week 48 without experiencing an mSFI-defined or BILAG-2004-defined
  flare (regardless of the severity of flare) after the first prednisone equivalent dose
  decrease.
- Percent of subjects who are able to discontinue prednisone (or equivalent) before
  or on Week 48 without experiencing an mSFI-defined or BILAG-defined severe
  flare after the first prednisone equivalent dose decrease.
- Actual values and change from Baseline in the physical and mental component scores of Short Form (36) Health Survey (SF-36) at Week 24 and at Week 48.
- Actual values and change from Baseline in 28 joint count swollenness and tenderness at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48.
- Actual values and change from Baseline in Cutaneous Lupus Erythematosus disease Area and Severity Index (CLASI) at Week 12, 24 and Week 48.

### Pharmacokinetic (PK) Endpoints:

Pharmacokinetic (PK) concentration at Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, and Week 48.

### **Pharmacodynamics Endpoints:**

- Actual values and percent change from baseline in the following Pharmacodynamic (PD) markers (including total sIL-6R, C-reactive protein [CRP], fibringen, anti-dsDNA (FARR), C3, C4 and CH50)
  - For sIL-6R: at Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48 and Follow-up.
  - For CRP, fibrinogen, anti-dsDNA (FARR), C3, C4 and CH50: at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48 and Follow-up.
- Shift from Baseline in Fibrinogen CTCAE grade category at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Follow-up and Worst on-treatment post-baseline visit.
- Actual values and percent change from Baseline in the following biomarkers at Week 8, Week 24 and Week 48.
  - Monocyte Chemotactic Protein-1 in urine (uMCP-1),
  - o uMCP-1/urine creatinine (uCr).

## **Immunogenicity Endpoints:**

- Overall subject classification based on ADA/mADA assays results.
- Overall subject classification based on NAb assay results.

### **Safety Endpoints:**

- Number of events as well as number and percent of subjects with Adverse Events
  (AEs), treatment-related AEs, Serious Adverse Events (SAEs), non-Serious AEs,
  treatment-related SAEs, AEs leading to treatment discontinuation and Adverse
  Events of Special Interest (AESI) categorized by System Organ Class (SOC),
  Preferred Term (PT) and Maximum Severity (where applicable).
- Actual values and change from Baseline in vital signs measurements at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48 and Follow-up.
- Actual values and change from Baseline in Electrocardiogram (ECG) values at Week 48.
- Actual values and change from Baseline in blood chemistry parameters (including liver enzymes and lipids), hematology parameters (including neutrophils and platelets) and coagulation parameters at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Follow-up and worst on-treatment.
- Number and percent of subjects with abnormal laboratory parameters of special interest at time post-Baseline.
- Shift from Baseline in laboratory parameters categorized with normal ranges or CTC grades at Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Follow-up and worst on-treatment post-Baseline.
- Number and percent of subjects for each pattern of anti-nuclear antibodies (ANA) at Screening and Week 24.
- Actual titres of ANA at Screening and Week 24.
- Actual values and change from Baseline in β2-glycoprotein I IgG, β2-glycoprotein I IgM, anti-cardiolipin IgA, anti-cardiolipin IgG, anti-cardiolipin IgM and anti-lupus at Week 24.

#### 4 General Statistical Considerations

Statistical analysis will be performed using SAS® Version 9.3 or higher on the Windows 7 platform. The Multiple Comparison Procedure – Modelling (MCP-Mod) procedure will be implemented using R version 3.1.0 (or higher) with the DoseFinding package version 0.9.15 (or higher) on the Windows 7 platform. SF-36 domains and components score will be derived by SF-36 v2 Scoring software.

Standardized and validated SAS macros from PPD will be used to set up table, listing, figure (TLF) formats (headers/footers and tabulation format) and tabulate the summaries (with the exception of the tables and figures programmed in R). All tables and listings will be independently validated using double programming; all figures will be independently validated manually.

#### **Treatment Labels**

The following treatment labels will be used in the Tables, Figures and Listings. Placebo will be presented first and then active treatment in increasing dosing received. An all active treatments combined group will be presented as an additional column for disposition, demographic and baseline characteristics, prior/concomitant medication, immunogenicity and safety outputs. Where applicable, in the listing, subjects who are randomized but not treated will be presented in a "Not Treated" column, which will be presented prior to the Placebo column.

**Table 4-1: Treatment Labels** 

| Treatment group | Treatment Label |
|---------------------|---------------------|
| Placebo | Placebo |
| ALX-0061 75 mg q4w | ALX-0061 75 mg q4w |
| ALX-0061 150 mg q4w | ALX-0061 150 mg q4w |
| ALX-0061 150 mg q2w | ALX-0061 150 mg q2w |
| ALX-0061 225 mg q2w | ALX-0061 225 mg q2w |
| All ALX-0061 | All ALX-0061 |

#### **Visit Naming Conventions**

For immunogenicity, Screening and Baseline assessments will be reported separately. The CRF visit label will be used to classify the assessments. All other assessments (including post Baseline immunogenicity) will be windowed (see Section 17.16).

The TLF shell Section 2.2.3 presents the visits labels convention that will be used in the Tables, Figures and Listings. For the Tables and Figures only scheduled post-Baseline visits will be displayed as per the schedule of events (see Section 17.1) in addition to the Baseline results, unless otherwise specified.

#### **Visit Windows**

The visit windows as defined in Section 17.16 will be applied to all parameters. For immunogenicity, both Screening and Baseline visits will be summarized separately and the CRF visit label will be used to classify the assessments.

# **Display of Data Summary and Analysis**

Continuous variables will be summarized using descriptive statistics, including the following: mean, standard deviation (SD) for demographics and Baseline disease characteristics summaries as well as for PK summaries, standard error (SE) for all PD and other summaries, median, minimum and maximum value; additional descriptive statistics will be provided for the summary of drug concentration, PD and ANA endpoints (see Section 9.2.6, Section 10 and Section 11). All minimum and maximum values will be displayed to the level of precision as the raw data, the quartiles (if applicable), mean and median will be displayed to one level of precision greater, and the SD and SE will be displayed to two additional levels of precision. For the safety and efficacy laboratory data, PD and immunogenicity data; the precision level of the raw data can be found in Section 17.14. Pharmacokinetic concentrations and descriptive statistics will be reported to 3 significant digits for values up to, but not including 1000. Values equal to and above 1000 will be reported as the value without decimal place.

95% confidence intervals (CIs) will be two-sided and displayed to the same level of precision as the statistic they relate to. If an estimate or a CI is not estimable, it will be

presented as 'NE'. If neither an estimate, nor its CI are estimable, it will be presented as simply 'NE', not displaying 'NE' twice.

The p-values will be two-sided and will be rounded to three decimal places. If a p-value is less than 0.001 it will be reported as '<0.001.' If a p-value is greater than 0.999 it will be reported as '>0.999.'

Categorical variables will be summarized using frequency counts and percentages. When count data are presented, the percent will be suppressed when the count is zero in order to draw attention to the non-zero counts. A row denoted 'Missing' will be included in count tabulations for demographics, Baseline characteristics and compliance to account for missing values. No percentages will be displayed on the 'Missing' rows and the percentages will be based on the number of non-missing observations. Unless otherwise specified, the denominator for all other percentages will be the number of subjects in that treatment within the specific analysis set of interest. Percentages will be displayed using one decimal place.

### Figures display

The TLF shell Section 2.2.7 presents the display that will be used in the Figures.

### Listing display/contents

See Section 17.19 for details on listings contents and display.

#### Baseline, study day and duration derivations

Baseline will be defined as the last non-missing assessment prior to the first dose. If there are multiple non-missing assessments collected on Day 1 where the time is not available, the assessment linked with the Baseline CRF Visit will be considered the baseline value. Where applicable, time will also be used to determine the pre/post Baseline assessment. Thus, the Baseline assessments for different variables may be collected at different times or on different days.

For post-Baseline visits, all visits including unscheduled visits are used to determine the analysis visit. For BILAG-2004, the visit mapping will be based on the date of assessments. If there are multiple results within the same visit windows, the non-missing assessment/sample closest to the planned study day will be selected for analysis. In case of ties, the first non-missing assessment after the target day will be selected for analysis. In case of ties on the same day with time not available, the assessment linked with the CRF visit will be selected for analysis.

For immunogenicity, Screening and Baseline assessments will be reported separately. The CRF visit label will be used to classify the assessments.

Calculations using dates (e.g. subject's age or relative day after the first dose of study drug) will adhere to the following conventions:

- Study days on or after the start day of study drug will be calculated as the difference between the date of interest (TARGET DATE) and the first date of dosing of study drug (DSTART) plus 1 day. The generalized calculation algorithm for relative day is the following:
  - If TARGET DATE ≥ DSTART then STUDY DAY = (TARGET DATE DSTART) + 1;
  - Else use STUDY DAY = TARGET DATE DSTART.

Statistical Analysis Plan, Final Version 1.0 Date Issued: 28FEB2018

Note that Study Day 1 is the first day of treatment of study drug. Study days on or before Day 1 are reflective of observations obtained during the Baseline/Screening period.

 Intervals that are presented in weeks will be transformed from days to weeks by using (without rounding) the following conversion formula:

$$WEEKS = DAYS / 7$$

• Intervals that are presented in months will be transformed from days to months by using (without rounding) the following conversion formula:

$$MONTHS = DAYS / 30.4375$$

# 4.1 Analysis Populations

### 4.1.1 All Screened Population

The all Screened population includes every subject who has signed informed consent.

The all Screened population will be used for summaries of disposition and associated listing. Listing of Informed Consent and Protocol Version will also use the all Screened population.

#### 4.1.2 All Randomized Population

The all Randomized population includes all subjects who have been randomized.

The all Randomized population will be used for listing of the subjects excluded from analysis populations as well as summarizing the number of subjects randomized in each country. Subjects will be summarized and listed based on the treatment they have been randomized to.

#### 4.1.3 Modified Intent-to-Treat (mITT) Population

The mITT population comprises all randomized subjects who received at least 1 administration of study drug. All subjects will be analyzed based on the treatment group they were randomized to regardless of the dosing regimen (dose and/or frequency for ALX-0061) received.

The mITT population will be used for summaries and analysis of demographics and Baseline characteristics, treatments and medications, secondary efficacy endpoints and will be the primary population for the analysis of the primary endpoint.

### 4.1.4 Per Protocol (PP) Population

The PP population consists of a subset of the mITT population, and excludes those subjects who have had a major protocol violation or deviation which might potentially impact the primary endpoint. All violations and deviations will be reviewed in a blinded fashion prior to database lock and classified as major or minor.

The Protocol Deviation Plan will contain all the information regarding the definitions of deviations, the frequency of meetings to be held by the study team to discuss any deviation related data, and the deviations to be used, which are also in the below categories. Protocol deviations will be reviewed on an ongoing basis throughout the trial.

Major protocol deviations are generally those which affect the general well-being and safety of the subject or have an impact on the scientific integrity of the study and will include the following violations (not an exhaustive list):

Missing primary endpoint at Week 24:

- o BILAG-2004 missing at Baseline and/or at Week 24.
- o SLEDAI-2K missing at Baseline and/or at Week 24.
- o PGA missing at Baseline and/or at Week 24.
- Failure to meet eligibility criteria.
- Incorrect treatment received:
  - o Incorrect dose received.
  - o Incorrect dosing regimen received.
- Criteria for study drug discontinuation met but the subject was not withdrawn from treatment.
- Intake of prohibited concomitant medications:
  - o Investigational or biological drug.
  - o Live, attenuated vaccine during the study or within 6 months after dosing.
  - o Intravenous immunoglobulins, cyclophosphamide or tacrolimus.
  - Therapy blocking the IL-6 pathway, such as but not limited to ALX-0061, sirukumab, tocilizumab, sarilumab, clazakizumab, olokizumab, or JAK inhibitors.

Based on the Protocol Deviation Plan, the following deviations reported into the CTMS and imported in the DV domain will lead to excluding the subject from the PP Population.

| Deviation Category | DVDECOD | DVTERM |
|---|---|---|
| Missing primary endpoint at Week 24 | Efficacy<br>Assessment<br>Deviation | Physician Global assessment not completed by the Investigator at baseline |
| | Deviation | Physician Global assessment not completed by the Investigator at Week 24 |
| | | (BILAG-2004 not completed at screening |
| | | or |
| | | BILAG-2004 2 not fully completed at screening:<br><specify and="" body="" items="" number<br="" or="" system="">missing&gt;)</specify> |
| | | <u>and</u> |
| | | (BILAG-2004 not completed at baseline |
| | | or |
| | | BILAG-2004 not fully completed at baseline:<br><specify and="" body="" items="" number<br="" or="" system="">missing&gt;)</specify> |
| | | BILAG-2004 not completed at Week 24 |
| | | BILAG-2004 not fully completed at Week 24:<br><specify and="" body="" items="" missing="" number="" or="" system="">.</specify> |

| <b>Deviation Category</b> | DVDECOD | DVTERM |
|---|---|---|
| Missing primary<br>endpoint at Week 24 | Efficacy<br>Assessment<br>Deviation | (SLEDAI not completed at screening or SLEDAI not fully completed at screening. Descriptor item <specify item(s)=""> missing) and (SLEDAI not completed at baseline or SLEDAI not fully completed at baseline. Descriptor item <specify item(s)=""> missing. SLEDAI not completed at week 24</specify></specify> |
| | | SLEDAI not fully completed at Week 24. Descriptor item <specify item(s)=""> missing.</specify> |
| | Other | The subject missed visit week 24 |
| | | Visit out of window: Week 24 was done <specify after="" before="" days=""> the planned visit date.</specify> |
| | | Where <specify after="" before="" days=""> is greater or equals to 14.</specify> |
| Failure to meet eligibility criteria. | Selection Criteria not met | Any |
| Incorrect treatment received | Treatment non-compliance | Any deviation recorded under "Kit number of study drug dispensed to subject at <specify visit=""> was not the same as kit number assigned by IRT.", where <specify visit=""> is Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 14, Week 16, Week 18, Week 20 or Week 22.</specify></specify> |
| | | for which (after unblinding) the dispensed kit number correspond to the incorrect treatment (e.g. kit number should correspond to Placebo but correspond to ALX0061) |
| Criteria for study<br>drug discontinuation<br>met but the subject<br>was not withdrawn<br>from treatment | Subject Not<br>Withdrawn as<br>per Protocol | Any deviations with a text started by "Before or at week 24" |
| Intake of prohibited concomitant medications | Prohibited concomitant medication | Any deviations with a text started by "Before or at week 24" |

| Deviation Category | DVDECOD | DVTERM |
|---|---|---|
| Undeclared/rejected IMP received | Treatment non-compliance | Any deviation recorded under "DOSING WITH UNDECLARED/REJECTED IP: DEVIATIONS TO THE STUDY DRUG CONDITIONS WHEN ADMINISTERED TO THE SUBJECT AT <specify visit="">." Where • for subjects randomized to ALX0061 75 or 150 mg q4w: visit is Baseline, Week 4, Week 8, Week 12, Week 16 or Week 20. • for subjects randomized to ALX0061 150 or 225 mg q2w: visit is Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 14, Week 16, Week 18, Week 20 or Week 22</specify> |

In addition, the following criteria will be programmed and subjects meeting this criterion will be excluded from the PP Population.

- For subjects randomized in the ALX-0061 75 mg q4w or ALX-0061 150 mg q4w:
   if ≥ 1 active dose has been missed between Baseline and Week 20 visit.
- For subjects randomized in the ALX-0061 150 mg q2w or ALX-0061 225 mg q2w: if ≥ 2 active doses missing between Baseline and Week 22 visit.

Subjects included in the PP population will be analyzed according to the randomized treatment. The PP population will be used as a supportive population for summaries and analyses of the primary endpoint.

### 4.1.5 Safety Population

The Safety population consists of all subjects who received at least 1 administration of study drug. All subjects will be classified based on the actual treatment group. This is the treatment group they were randomized to, except if the subject received a different dose regimen during the whole treatment period. In that case, the subject will be summarized based on the first treatment received. For subjects who received 150 mg as first dose, the dose administered at the following planned dosing visit (e.g. Week 2 if the first dose was administered at Baseline) will be considered as described in Table 4-2. For the subjects for which no dose was received at the planned dosing visit following the first dose (e.g. the subject discontinued, the visit was missed and no drug administered), the actual treatment group should be derived as follows:

- If the subject was randomized to 150 mg q2w or 150 mg q4w, the actual treatment will be set to be equal to the planned treatment
- If the subject was randomized to placebo, 75 mg q4w or 225 mg q2w, the actual treatment will be set to be 150 mg q4w.

**Table 4-2: Actual Treatment Group** 

| First Dose Received (ALX-0061)[a] | Second Dose Received (ALX-0061) <sup>[a]</sup> | Actual Treatment Group |
|---|---|---|
| 0 mg | Any | Placebo |
| 75 mg | Any | ALX-0061 75 mg q4w |
| 150 mg | 150 mg or 225 mg | ALX-0061 150 mg q2w |
| 150 mg | 0 mg or 75 mg | ALX-0061 150 mg q4w |
| 225 mg | Any | ALX-0061 225 mg q2w |

<sup>[</sup>a] first dose received should be at Baseline and second dose at Week 2.

The Safety population will be used for the summaries and analyses of the safety data as well as for the PK concentrations summaries and immunogenicity summaries.

### 5 Subject Disposition

#### 5.1 Disposition

Subject disposition will be summarized and listed for the all Screened population for each treatment group, "All ALX-0061" group and overall. A disposition of subjects includes the number of subjects who were screened, number of subjects who were randomized, number and percentage of subjects who were treated, number and percentage of subjects who discontinued from study during treatment period (i.e. have discontinued from the study and did not perform their Week 48 visit) and number and percentage of subjects who discontinued from the study during the follow-up period (i.e. have discontinued from the study but attended Week 48 visit). Percentages will be based on the number of subjects randomized. The reasons for discontinuation will also be summarized in this table. Percentages will be based on the number of subjects randomized.

The number of subjects randomized per country will be summarized for the all Randomized population.

A listing of screen failures will be provided.

Statistical Analysis Plan, Final Version 1.0 Date Issued: 28FEB2018

### 5.2 Analysis Populations

A summary of the analysis sets including the number and percentage of subjects for the following categories: subjects in the Safety population, subjects in the mITT population, and subjects in the PP population will be presented by treatment group, "All ALX-0061" group and overall. Percentage of subjects in the PP population will be based on the number of subjects in the mITT population.

A listing of subjects excluded from analysis populations will be provided.

#### 5.3 Protocol Deviations

The Protocol Deviation Plan document will contain all the information regarding the definitions of deviations, and the frequency of meetings to be held by the study team to discuss any deviation related data. All information held in that document will be updated as needed. General examples for major protocol deviations are provided in the PP population description, in Section 4.1.4 of this document. All major protocol deviations will be identified, and therefore the list of subjects excluded from the PP population will be finalized before database lock and unblinding.

A summary table of subjects per major protocol deviation category will be presented by treatment group, "All ALX-0061" group and overall and will be based on the mITT population.

Listing of protocol major deviations will be provided.

# 6 Demographics and Baseline Characteristics

Summaries for this section will be presented by treatment group, "All ALX-0061" group and overall using the mITT population.

# **6.1 Demographics**

The demographic characteristics consist of age (years), sex, race, and ethnicity. The Baseline characteristics consist of Baseline height (cm), Baseline weight (kg), Baseline body mass index (BMI)  $(kg/m^2)$  and geographic region. BMI is calculated as (body weight in kilograms) / (height in meters)<sup>2</sup>.

The following characteristics will be summarized using descriptive statistics.

- · Age (years),
- Baseline height (cm),
- Baseline weight (kg),
- Baseline BMI (kg/m²),

The number and percentage of subjects will be calculated for the following characteristics. Percentages will be based on the number of subjects in the mITT population and relevant treatment group with non-missing data.

- Age (18 to <45 years, 45 to <65 years),</li>
- Sex (Male, Female),
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, and Other),
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino),
- BMI (≤25 kg/m², > 25 kg/m²),
- Geographic region (North America, Latin America, Europe and Asia-Pacific),

Listings of demographics and Baseline characteristics will be provided. All CRF scheduled study visits dates will be displayed in a listing. In addition, the first subject first visit date and last subject last visit date will be provided in a listing.

#### 6.2 Baseline Disease Characteristics

The following baseline disease characteristics will be summarized using descriptive statistics.

- Baseline SLEDAI-2K score,
- Baseline BILAG-2004 total score,
- Baseline PGA score,
- Baseline CLASI activity score,
- Baseline CLASI damage score,
- · Baseline SF-36 physical component score,
- · Baseline SF-36 mental component score,
- Baseline 28-joint count total score Swollenness,
- Baseline 28-joint count total score Tenderness,
- Baseline Prednisone Equivalent Dose intake,
- Disease duration (months),
- Baseline SLICC damage score.

The number and percentage of subjects for the following baseline disease characteristics will also be reported. Percentages will be based on the number of subjects in the mITT population and the relevant treatment group with non-missing data.

- Baseline SLEDAI-2K score (< 10, ≥ 10),</li>
- At least one organ system with BILAG-2004 score A at Baseline (yes, no),
- At least two organ systems with BILAG-2004 score B at Baseline (yes, no),
- At least one BILAG-2004 score A or B at Baseline by organ system (yes, no),
- Baseline immunosuppressants intake (yes, no),
- Baseline corticosteroids intake (yes, no),
- Baseline Prednisone Equivalent Dose intake > 7.5 mg/day (yes, no),
- Baseline anti-dsDNA (FARR) ≥ 8 IU/mL (yes, no),
- Baseline SLEDAI-2K low complement item (yes, no),

- Baseline anti-malarial intake (yes, no).
- SLICC/ACR disease classification (None, SLICC, ACR, SLICC and ACR).
- Disease duration (< 6 months, 6 months to <1 year, 1 year to < 5 years and ≥ 5 years).</li>

Disease duration (months) is derived as the date of informed consent minus the date of diagnosis divided by 30.4375.

If the date of diagnosis is partial:

- If only the day is missing, the date will be imputed by the 15<sup>th</sup>;
- If only the day and month are missing, the date will be imputed by the 1<sup>st</sup> of July if the year of diagnosis is smaller than year of informed consent. If the year of diagnosis is the same as the year of informed consent then the day and month will not be imputed.

The SLICC damage score will be derived as described in Section 17.13. Individual responses to questions will be listed.

# 6.3 Tobacco Usage

Past and present tobacco usage will not be summarized but will be listed only.

# 6.4 Medical History

The number and percentage of subjects with any medical history will be summarized overall and for each predefined body system. Applicable body system codes include Dermatologic; Head, Eyes, Ears, Nose, Throat (HEENT); Respiratory; Cardiovascular; Gastrointestinal; Endocrine/Metabolic; Genitourinary; Neurologic; Blood/Lymphatic; Musculoskeletal; Hepatic; Allergy/Drug Sensitivity; Psychological/Psychiatric and Other. Percentages will be calculated based on number of subjects in the mITT population. Body system codes will be sorted in descending order of frequency based on the total of all treatment groups.

A listing of medical history will be provided.

### 6.5 Additional Screening/Baseline Assessments

Screening test results for Hepatitis B, Hepatitis C and human immunodeficiency virus (HIV) will be provided in data listing.

# 7 Treatments and Medications

# 7.1 Prior and Concomitant Medications

Summaries for this section will be presented by treatment group, "All ALX-0061" group and overall using the mITT population.

All medications (including SLE medications) used within a year of the date of informed consent through the end of the study (follow-up visit) will be collected on the CRF. SLE medications are recorded on the "SLE Medication" CRF page, while the other medications are recorded on the "Concomitant Medications" CRF page. All medications will be coded according to the latest World Health Organization Drug Dictionary (WHO-DD).

For the purpose of inclusion in prior and/or concomitant medication tables, incomplete medication start and stop dates will be imputed as described in Section 17.15.

SLE Prior/Concomitant Medications and Other Prior/Concomitant medications will be summarized and listed.

#### 7.1.1 Prior Medications

A prior medication is defined as any medication that is taken prior to the first dose of study drug.

#### **SLE Prior Medications**

The number and percentage of subjects with at least one prior SLE medication will be summarized by treatment group. The number and percentage of all prior SLE medications will be summarized by treatment group and listed by ATC level 4 and PT. Medications will be sorted in descending order of frequency of ATC 4 category based on the total of all treatment groups. Within each ATC 4 category, PTs will be sorted in descending order of frequency based on the total of all treatment groups.

#### **Other Prior Medications**

Other prior medications will be summarized similarly as prior SLE medications.

### 7.1.2 Concomitant Medications

A concomitant medication is defined as any medication that has a stop date that is on or after the date of first dose of study drug.

#### **Concomitant SLE Medications**

The number and percentage of subjects with at least one concomitant SLE medication will be summarized by treatment group. The number and percentage of all concomitant SLE medications will be summarized by treatment group and listed by ATC level 4 and PT. Medications will be sorted in descending order of frequency of ATC 4 category based on the total of all treatment groups. Within each ATC 4 category, PTs will be sorted in descending order of frequency based on the total of all treatment groups.

#### **Other Concomitant Medications**

Other concomitant medications will be summarized similarly as concomitant SLE medications.

### 7.2 Study Treatments

Extent of exposure and compliance will be summarized using descriptive statistics and frequency count by treatment group, and listed based on the Safety population.

### **Duration of Exposure (weeks):**

The duration of exposure is the number of weeks elapsed between the first and last dose (i.e. Date of last dose - date of first dose + 1 day, divided by 7).

The duration of exposure will be summarized by treatment group using descriptive statistics.

### **Actual Cumulative Dose (mg):**

The actual cumulative dose is the sum of all doses received (from syringes A and B); if a dose was administered but not complete, it will be assumed that 50% of the syringe content was administered. The actual cumulative dose (mg) will be summarized using descriptive statistics.

### **Compliance to Injections (%)**

Compliance to injections is the number of injections received regardless of the syringe type received (complete and incomplete) divided by the expected number of injections x 100. The expected number of injections is the expected number of injections up to the last available visit. For prematurely discontinued subjects, it corresponds to the expected number of injections up to last available assessment visit before discontinuation. The compliance to injections will be summarized by descriptive statistics; in addition the number and percentage of subjects with compliance to injections < 90%, between 90% and 110% and > 110% will be provided.

# **8 Efficacy Analysis**

The statistical inference will be 2-sided and performed at the 5% significance level, thereby providing 95% (2-sided) CIs. The MCP-Mod will be employed to address any multiplicity arising from the analysis of the primary endpoint using different models. Analyses will be performed on the secondary efficacy endpoints (see Section 8.2 for details) using 2-sided tests at 5% significance level. No adjustment for multiplicity for the secondary endpoints analysis will be performed as those analyses will be exploratory in nature. Statistical interpretation of the results will not be done on a single endpoint but will be based on the patterns of results.

Change from Baseline will be calculated as follows: post-Baseline value – Baseline value. Percent change from baseline will be (change from Baseline divided by Baseline value) x 100. For the changes from Baseline, only subjects with a value at both the Baseline visit and the specific post-Baseline visit will be included. Note that the post-Baseline visit value may be imputed, as described in Section 8.1 below.

All endpoints will be summarized by treatment group using descriptive statistics or frequency count and percentages.

For all secondary efficacy endpoints (excluding BILAG-2004 Systems Tally), the following inferential statistics will be provided:

- LSMeans, SE of the LSMeans and 95% CI of the change from Baseline for continuous endpoints from an analysis of covariance (ANCOVA) model or the Clopper Pearson 95% CI of the response rate/incidence will be provided by treatment group,
- LSMeans and 95% CI (from the ANCOVA) of the difference between each of the
  active treatment group versus the placebo group for continuous endpoints and
  difference and 95% CI (from the stratified CHM test) of the difference between
  each of the active treatment group versus the placebo group for binary endpoints.

In addition, p-values from the Cochran-Mantel-Haenszel (CMH) test stratified by geographic region [15] will be provided for the comparison of each active treatment group versus placebo group for the following endpoints and both Week 24 and Week 48 time points. Details for deriving the stratified CMH 95% CI and p-value can be found in Section 17.22.

- mBICLA response rate,
- mSRI response rate,
- Mild/moderate and severe mSFI-defined flare incidence rate (overall and split by intensity),
- Mild/moderate and severe BILAG-2004-defined flare incidence rate (overall and split by intensity),
- Treatment Failure incidence rate.

Unless otherwise specified, the mITT population will be the basis for all efficacy analyses. The PP population will be used for supportive summary and analysis of the primary endpoint. In addition, subgroup summary (see Section 8.1.4) will be performed for the primary endpoint based on the mITT population.

### 8.1 Primary Efficacy Endpoint

The primary endpoint is the mBICLA response rate at Week 24. The derivation of this endpoint is described in Section 17.6.

For the purpose of calculating the mBICLA response rate for the primary endpoint at Week 24, if mSLEDAI-2K is done but there are a few missing items in mSLEDAI-2K, the following imputation rule will be applied. If no more than 25% (including 25%) of the mSLEDAI-2K items are missing at Week 24 then the value will be imputed with the previous recorded value of the same item (last observation carried forward [LOCF] imputation). Baseline items (i.e. any records that occurred prior or on the first dose of study drug) will not be used to impute missing on-treatment items. If more than 25% of the items are missing then imputations rules will not be applied and mSLEDAI-2K score may be missing. Missing BILAG-2004 items will be imputed according to the specific rules described in Section 17.3.5.1.

Subjects will have mBICLA missing if any of the following is missing after the LOCF imputation for mSLEDAI-2K or after the imputation rules described in Section 17.3.5.1 have been applied for BILAG-2004 system organs scores:

- Missing BILAG-2004 at baseline or/and missing at Week 24, or
- Missing mSLEDAI-2K at baseline or/and missing at Week 24, or
- Missing PGA at baseline or/and missing at Week 24.

Subjects with missing mBICLA response at Week 24 including subjects who discontinued prior to Week 24 or who are confirmed treatment failures by a medical review (as described in Section 17.5) will be imputed as non-responders (i.e. non-response imputation approach [NRI]).

### 8.1.1 Primary Analysis

mBICLA response rates at Week 24 will be analyzed for dose-response using the MCP-Mod methodology [1, 11]. As the subjects are assigned to different dose schedules, the nominal doses included in the dose-response modelling will be as follows:

- Subjects randomized to Placebo will be assigned a dose of 0 mg,
- Subjects randomized to ALX-0061 75 mg q4w will be assigned a dose of 37.5 mg,
- Subjects randomized to ALX-0061 150 mg q4w will be assigned a dose of 75 mg,
- Subjects randomized to ALX-0061 150 mg q2w will be assigned a dose of 150 mg,
- Subjects randomized to ALX-0061 225 mg q2w will be assigned a dose of 225 mg.

The MCP-Mod method entails a unified strategy to the analysis of data from dose-response studies which combines multiple comparison and modelling techniques. The existence of several candidate parametric models is assumed and multiple comparison techniques are used to choose the model(s) most likely to represent the true underlying dose-response curve, while preserving the family-wise error rate. The selected model may further be used to guide the choice of adequate doses.

The MCP-Mod consists of the 2 major steps [11]: a multiple comparison step and a modelling step. The focus for the primary analysis will be on the MCP step. This step aims to establish evidence of a drug effect by testing for a statistically significant doseresponse signal for the clinical endpoint and patient population investigated in the study. This step will be performed using a multiple contrast test, adjusting for the fact that multiple candidate dose-response models are being considered.

The adjusted p-values for all models will be reported, with the primary objective being met if at least one of the values < 0.05.

Candidate models will be selected amongst the following types of parametric models. In these models, the following notation is used:

- d is the treatment dose,
- E(d) is the probability of a response at dose d,
- $E_0$  represents the probability of a response for the placebo treatment group,
- $E_0 + E_{max}$  is the maximum possible response probability,
- $ED_{50}$  is the dose that evokes a response of  $E_0 + E_{max}/2$ ,
- $\delta$ ,  $\delta_1$ ,  $\delta_2$ ,  $\epsilon$ ,  $\theta$  and scal are model-specific parameters.

$$E(d) = E_0 + \delta d$$

$$E(d) = E_0 + E_{max} \frac{d}{ED_{50} + d}$$

Logistic

$$E(d) = E_0 + \frac{E_{max}}{\left(1 + e^{\frac{ED_{50} - d}{\delta}}\right)}$$

Beta model

$$E(d) = E_0 + E_{max}B(\delta_1, \delta_2) \times \left(\frac{d}{scal}\right)^{\delta_1} \times \left(1 - \frac{d}{scal}\right)^{\delta_2}$$

where

$$B(\delta_1, \delta_2) = \frac{(\delta_1 + \delta_2)^{\delta_1 + \delta_2}}{\delta_1^{\delta_1} \times \delta_2^{\delta_2}}$$

scal is a fixed parameter.

The following parametrization will be used for the Emax, logistic and Beta models; plot of the models are included in Figure 8-1.

- **Emax model** with 80% of the maximum effect at 75 mg.
- **Logistic model** with 10% of the maximum effect at 37.5 mg and 90% effect at 150 mg.
- **1**<sup>st</sup> **Beta model** with 90% of the maximum effect at 75 mg and 70% of maximum effect at 150 mg, the maximum effect is reached at 37.5 mg dose and the maximal dose is 225 mg. The scale effect is 270 (1.2 times the maximal dose).
- **2<sup>nd</sup> Beta model** with 40% of the maximum effect at 37.5 mg and 70% of maximum effect at 75 mg, the maximum effect is reached at 150 mg dose and the maximal dose is 225 mg. The scale effect is 270 (1.2 times the maximal dose).

For all models E<sub>0</sub> will be set to 25% and E<sub>max</sub> will be set to 25%.



Figure 8-1: Graphical Representation of the Candidate models

The following steps [11] are used to determine the best dose response model and optimal dose using the DoseFinding package available in R. An example R code is provided in Section 17.17.

- Define the doses used in the study.
- Estimate the model parameters for each candidate model using the guesst function.
- Create the class object containing all the candidate models using the Mods function.
- Obtain asymptotic covariance matrix  $\hat{S}$ , which is required to perform the multiple contrast test, by using the **glm** function to apply a logistic regression (with response rate as response, dose level as factor, and no intercept). Note that the logistic regression is used here only to obtain  $\hat{S}$  from the design matrix which depends on nuisance parameters in the model when applied to non-normal data. Since the logistic regression model will be used, the candidate models are formulated on the logit scale.
- Perform the multiple contrast test using optimal trend contrasts (obtained from the optContr function). The optimal contrasts for non-normal data are calculated using the asymptotic covariance matrix obtained from the logistic regression model in the previous step. The optimal contrasts and asymptotic covariance matrices will be re-calculated for NRI per-protocol and observed case mITT analyses but will not be reported. A seed of 61204 will be defined to generate the results.

- If there are two or more significant models,
  - Model the data using the candidate model(s) for which the contrast test is significant with the MCPMod function.
  - Obtain fitted values as a weighted average of the response estimates from models identified as significant in the previous step. The weights are based on the Akaike Information Criterion (AIC) criterion and are calculated as follows:  $w_i = exp(-0.5AIC_i) / \sum_i (exp(-0.5AIC_i))$  where i=1,..., number of significant models [12].
  - The weighted average is calculated as

$$\bar{x}_{k} = \frac{\sum_{i=1}^{n} w_{i} \hat{x}_{i, k}}{\sum_{i=1}^{n} w_{i}}$$

where  $x_k$  is the weighted average of the fitted value for the logit transformed responder rate for dose k and  $\hat{x}_{i,k}$  is the fitted value for the transformed responder rate for model i at dose k.

A confidence interval will be calculated for  $x_k$  as  $x_k \pm Z_{\alpha/2} \times sd(\bar{x}_k)$ . A conservative estimate of the standard deviation of  $x_k$  will be used to calculate the confidence interval where

$$sd\left(\bar{x}_{k}\right) = \sum_{k} w_{i} \sqrt{var(\hat{x}_{i,k})}$$

is the upper bound for  $sd(x_k)$ ,  $Z_{\alpha/2}$  is the quantile from the normal distribution for confidence level  $1-\alpha$ , and  $var(\hat{x}_{i,k})$  is obtained by squaring the standard error of  $\hat{x}_{i,k}$  [12].

• If none of the models are significant, then no dose-response has been shown and no further steps will be undertaken.

The parameter estimates from the candidate models will be provided in a table (the **guesst** function will be applied to each candidate model to estimate the required model parameters, then the **Mods** function will be applied to combine all model parameters into a "matrix" and provide the parametrization described earlier, i.e.  $E_0$ ,  $E_{max}$ ,  $E_{D50}$ ,  $\delta$  etc.).

The following tables representing each step of the procedure will be provided; the analysis will be based on the mITT population. The multiple contrast test results will also be provided for the PP population.

- The asymptotic covariance matrix  $\hat{S}$  using the **glm** function.
- The optimal contrast for each model using the **optContr** function.
- The multiple contrast test (t-statistics and adjusted p-values) as well as the critical value (obtained from the MCPMod function), the AIC value for each model, and the corresponding weight.
- The estimated model parameters (for example  $E_0$ ,  $E_{max}$  and  $ED_{50}$  for the Emax model) on the logit scale for each model that is significant (obtained from the **MCPMod** function).
- The fitted values and confidence interval obtained as a weighted average of predicted values from the significant model(s) at each dose of interest.

For each model, the observed mean and associated CI of the response rate on the logit scale will be plotted alongside the candidate model and its confidence curve (logit scale)

against dose. The observed mean and associated CI of the response rate on the logit scale will also be plotted alongside the predicted values and corresponding confidence curves (logit scale) obtained from weighted averaging of the significant models, against dose.

The mBICLA response rates at Week 24 will be summarized by treatment group and presented for both the mITT and PP populations in the same table. Percentages will be derived based on the number of subjects in the analysis population and corresponding treatment group.

The tables will be programmed in SAS, and the figures will be produced using R (rtf package version 0.4-11). The SAS dataset (export format) containing the response rates will be imported into R using theSASxport package (version 1.5.3). The results from the MCP-Mod analyses will be exported from R in CSV format using the foreign package (version 0.8-67) and the CSV files will be imported into SAS using code generated by the foreign package.

The trial will be considered to have met its primary endpoint if at least one of the adjusted p-values is < 0.05.

# 8.1.2 Assumption Testing

No assumption testing of the dose-response model will be performed.

#### 8.1.3 Sensitivity Analysis

The sensitivity of results to missing data will be assessed with the use of observed case analysis, i.e. without applying the imputation rules for mSLEDAI-2K described in Section 8.1. The observed mBICLA response rates at Week 24 will be summarized by treatment group and presented for the mITT population. Percentages will be derived based on the number of subjects in the analysis population evaluated at Week 24 and corresponding treatment group.

In addition, to further evaluate the impact of the imputation of missing values, the multiple contrast test results from the primary endpoint analysis (MCP-Mod) will be provided as well using observed mBICLA responses on the mITT population, and the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% CI of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be also presented. 95% CI for the difference between each active treatment and placebo will be based on the CMH test stratified by geographic region. In addition, the associated p-value will be provided.

### 8.1.4 Subgroup Analysis

The primary endpoint will be summarized using frequency count and percentages by treatment groups on the mITT population for the following subgroups. Imputation rules from Section 8.1 will be applied to the data for subgroup analysis at Week 24.

- Age (18 to <45 years, 45 to <65 years),</li>
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, and Other),
- Geographic Region (Europe, Latin America, North America and Asia-Pacific),
- Baseline SLICC damage score (= 0 , > 0),
- Baseline BMI (≤ 25 kg/m², > 25 kg/m²),
- Baseline immunosuppressants intake (yes, no),
- Baseline corticosteroids intake (yes, no),
- Baseline SLEDAI-2K score ≥ 10 (yes, no),
- Baseline mSLEDAI-2K score ≥ 10 (yes, no),
- System Mucocutaneous with BILAG-2004 score A at Baseline (yes, no),
- System Musculoskeletal with BILAG-2004 score A at Baseline (yes, no),
- Baseline Prednisone Equivalent Dose intake > 7.5 mg/day (yes, no),
- Baseline anti-dsDNA (FARR) ≥ 8 IU/mL (yes, no),
- Baseline SLEDAI-2K low complement item (yes, no).

### 8.2 Secondary Efficacy Endpoints

All secondary efficacy endpoints (see Section 3.2.2) will be summarized and analyzed by planned treatment group, using the observed data (i.e. without applying the imputation rules for mSLEDAI-2K described in Section 8.1) in the mITT population. For continuous secondary efficacy endpoints, summary statistics include mean, SE, median, minimum and maximum, while for categorical secondary efficacy endpoints frequencies and proportions are provided. Definitions of endpoints are included in Section 17.3 to Section 17.13.

### 8.2.1 mBICLA

The number and percentage of subjects who are mBICLA responders will be presented for each post-Baseline visit (Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48) alongside the number of subjects evaluated at that visit. The mBICLA responder rate will be presented as percentage and derived based on the number of subjects who are evaluable at the visit.

Furthermore, at each post-Baseline visit, the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% CI of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be also presented. 95% CI for the difference between each active treatment and placebo will be based on the CMH test stratified by geographic region. In addition, at Week 24 and at Week 48, the associated p-value will be provided.

In addition, a line plot of the mBICLA response rate with the associated 95% CI will be provided by treatment group and visit.

The subgroup analysis from Section 8.1.4 will be repeated for mBICLA at Week 48. No imputation rules will be applied.

#### 8.2.2 BICLA

The number and percentage of subjects who are BICLA responders will be presented for each post-Baseline visit (Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48) alongside the number of

subjects evaluated at that visit. The BICLA responder rate will be presented as percentage and derived based on the number of subjects who are evaluable at the visit. Furthermore, at each post-Baseline visit, the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% CI of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be presented. 95% CI for the difference between active treatment and placebo will be based on the CMH test stratified by geographic region.

In addition, a line plot of the BICLA response rate with the associated 95% CI will be provided by treatment group and visit.

#### 8.2.3 SRI

The number and percentage of subjects who are SRI (see Section 17.7 for details) responders will be presented for each post-Baseline visit (Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48) alongside the number of subjects evaluated at that visit. The SRI responder rate will be presented as percentage and derived based on the number of subjects who are evaluable at the visit.

Furthermore, at each post-Baseline visit, the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be presented. 95% CI for the difference between active treatment and placebo will be based on the CMH test stratified by geographic region.

In addition, a line plot of the SRI response rate with the associated 95% CI will be provided by treatment group and visit.

Similar summaries and analyses will be presented for SRI-5, SRI-6, SRI-7 and SRI-8. For each cut-off, the number of assessable subjects will be displayed in these summaries; the number of assessable subjects is the number of subjects with Baseline SLEDAI-2K score greater than or equal to the cut-off point considered. For example, the cut-off for SRI is 4 and assessable subjects are subjects with Baseline SLEDAI\_2K score  $\geq$  4, the cut-off for SRI-5 is 5 and assessable subjects are subjects with Baseline SLEDAI-2K score  $\geq$  5 etc. The SRI responder rate will be presented as percentage and derived based on the number of assessable subjects who are evaluable at the visit.

### 8.2.4 mSRI

The number and percentage of subjects who are mSRI (see Section 17.7 for details) responders will be presented for each post-Baseline visit (Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48) alongside the number of subjects evaluated at that visit. The mSRI responder rate will be presented as percentage and derived based on the number of subjects who are evaluable at the visit.

Furthermore, at each post-Baseline visit, the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% CI of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be presented. 95% CI for the difference between active treatment and placebo will be based on the CMH test stratified by geographic region. In addition, at Week 24 and at Week 48, the associated p-value will be provided.

In addition, a line plot of the mSRI response rate with the associated 95% CI will be provided by treatment group and visit.

Similar summaries and analyses will be presented for mSRI-5, mSRI-6, mSRI-7 and mSRI-8. For each cut-off, the number of assessable subjects will be displayed in these summaries; the number of assessable subjects is the number of subjects with Baseline
mSLEDAI-2K score greater or equal to the cut-off point considered. The mSRI responder rate will be presented as percentage and derived based on the number of assessable subjects who are evaluable at the visit.

The same subgroups as for the primary endpoint (see Section 8.1.4) will also be used to summarize mSRI responders at Week 24 and 48 using frequency count and percentages by treatment group.

#### 8.2.5 **SLEDAI-2K**

The SLEDAI-2K score (see Section 17.4 for details) will be summarized at each visit (Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48).

In addition, at each post-Baseline visit, the change from Baseline will be modelled using an analysis of covariance (ANCOVA) model with treatment as factor and Baseline and geographic region as covariates. The LSMeans and SE of the LSMeans will be presented at each visit alongside the 95% CI. The difference in LSMeans between each of the active treatment group and placebo will be presented with the associated 95% CI.

#### 8.2.6 mSLEDAI-2K

The mSLEDAI-2K score (see Section 17.4 for details) will be summarized at each visit (Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48).

In addition, at each post-Baseline visit, the change from Baseline will be modelled using an ANCOVA model with treatment as factor and Baseline and geographic region as covariates. The LSMeans and SE of the LSMeans will be presented at each visit alongside the 95% CI. The difference in LSMeans between each of the active treatment group and placebo will be presented with the associated 95% CI.

#### 8.2.7 BILAG-2004 Improvement

#### **Normal Improvement:**

The number and percentage of subjects with normal improvement (see Section 17.3 for details) will be presented for each post-Baseline visit (Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48) alongside the number of subjects evaluated at that visit. The percentage of subjects with normal improvement will be presented and derived based on the number of subjects who are evaluable at the visit.

Furthermore, at each post-Baseline visit, the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% CI of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be presented. 95% CI for the difference between active treatment and placebo will be based on the CMH test stratified by geographic region.

### **Enhanced Improvement:**

The number and percentage of subjects with enhanced improvement (see Section 17.3 for details) will be presented for each post-Baseline visit (Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48) alongside the number of subjects evaluated at that visit. The percentage of subjects with enhanced improvement will be presented and derived based on the number of subjects who are evaluable at the visit.

Furthermore, at each post-Baseline visit, the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% CI of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be presented. 95% CI for the difference between active treatment and placebo will be based on the CMH test stratified by geographic region.

Subjects who meet the requirements for enhanced improvement also by definition meet the requirements for normal improvement and will therefore be counted as "responders" in both sets of presentations.

#### 8.2.8 BILAG-2004 Total Score

The BILAG-2004 total score (see Section 17.3 for details) will be summarized at each visit (Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48).

In addition, at each post-Baseline visit, the change from Baseline will be modelled using an ANCOVA model with treatment as factor and Baseline and geographic region as covariates. The LSMeans and SE of the LSMeans will be presented at each visit alongside the 95% CI. The difference in LSMeans between each of the active treatment group and placebo will be presented with the associated 95% CI.

## 8.2.9 BILAG-2004 Improvement by Individual Organ System

For each organ system (with at least 5 subjects in each treatment group with A or B score at Baseline), the number and percentage of subjects with normal improvement (see Section 17.3 for details) will be presented at each post-Baseline visit (Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48) alongside the number of subjects evaluated at that visit. The percentage of subjects with normal improvement will be presented and derived based on the number of subjects who are evaluable at the visit.

Furthermore, at each post-Baseline visit, the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% CI of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be also presented. 95% CI for the difference between active treatment and placebo will be based on the CMH test stratified by geographic region.

#### 8.2.10BILAG-2004 Systems Tally

Each organ system will be classified under active/worsening disease, improving disease, or persistent minimal or no activity (see Section 17.3 for details). For each subject the number of organ systems will be tallied within each category. Within the categories active/worsening disease and improving disease, the number and percentage of subjects with 1, 2, 3 and > 3 organ systems included will be summarized at each visit (Week 4, Week 8, week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48). For the persistent minimal or no activity category, the number and percentage of subjects with  $\leq$ 6, 7, 8 and 9 organ systems included will be summarized at each visit (Week 4, Week 8, week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48). Percentages will be

calculated based on the total number of subjects at the considered visit. Only subjects with non-missing assessments at Baseline and post-Baseline will be included in the summary.

#### 8.2.11PGA

The physician will make a mark between 0 ("very good") and 100 mm ("very bad") on the visual analogue scale (VAS) to indicate disease activity (independent of the subject's self-assessment).

The PGA score will be summarized at each visit (Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48).

In addition, at each post-Baseline visit, the change from Baseline will be modelled using an ANCOVA model with treatment as factor and Baseline and geographic region as covariates. The LSMeans and SE of the LSMeans will be presented at each visit alongside the 95% CI. The difference in LSMeans between each of the active treatment groups and placebo will be presented with the associated 95% CI.

#### 8.2.12 Patient's Global Assessment

The subject will make a mark between 0 ("very good") and 100 mm ("very bad") on the VAS to indicate disease activity.

The patient's global assessment of disease activity will be summarized at each visit (Week 24 and Week 48).

In addition, at each post-Baseline visit, the change from Baseline will be modelled using an ANCOVA model with treatment as factor and Baseline and geographic region as covariates. The LSMeans and SE of the LSMeans will be presented at each visit alongside the 95% CI. The difference in LSMeans between each of the active treatment groups and placebo will be presented with the associated 95% CI.

### 8.2.13Laboratory Efficacy Assessment

Summary tables presenting observed numeric values and changes from Baseline at each visit (Week 2 [blood chemistry parameters only], Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48 and Follow-up [blood chemistry parameters only]), will be provided for the following parameters (see Section 17.14 for the tests to be reported and units).

- Blood chemistry: Serum creatinine, eGFR
- Urinalysis: Proteinuria (urinary protein) as measured by spot urine protein to creatinine ratio.

In addition, at each post-Baseline visit, the change from Baseline will be modelled using an ANCOVA model with treatment as factor and Baseline and geographic region as covariates. The LSMeans and SE of the LSMeans will be presented at each visit alongside the 95% CI. The difference in LSMeans between each of the active treatment group and placebo will be presented with the associated 95% CI.

Active urine sediment (yes versus no) from the BILAG Renal CRF page will be summarized at each visit by way of shift table (i.e. summarizing the number of subjects who have [yes] or don't have [no] active urine sediment at Baseline and their shift at post-Baseline visit). The percentages will be based on the number of subjects with non-missing values at the Baseline and at the considered visit.

For urine protein/creatinine ratio, shift from Baseline at each post-Baseline visit and worst on-treatment using grade criteria below (Grade 0, Grade 1, Grade 2 and Grade 3) will be presented by treatment group.

- Grade 0: ≤ 17.0 g/mol (i.e. ≤0.15 g/g),
- Grade 1: > 17.0 g/mol to < 113.1 g/mol (i.e. > 0.15 g/g to < 1 g/g),</li>
- Grade 2:  $\geq 113.1$  g/mol to  $\leq 384.6$  g/mol (i.e.  $\geq 1.0$  g/g to  $\leq 3.4$  g/g),
- Grade 3: > 384.6 g/mol (i.e. > 3.4 g/g).

#### 8.2.14Treatment Failure

The number and percentage of subjects with treatment failure (see derivation details in Section 17.5) will be presented at Week 24 and at Week 48. The percentage of treatment failures will be also presented and derived based on the number of subjects in the mITT population.

Furthermore, at Week 24 and Week 48, the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% CI of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be presented. 95% CI for the difference between active treatment and placebo will be based on the CMH test stratified by geographic region. In addition, the associated p-value will be provided.

### 8.2.15BILAG-2004 Flare

The number of subjects with BILAG-2004 flare between Baseline and Week 24, and between Baseline and Week 48 (see Section 17.3 for details) will be presented by category (mild/moderate and severe). The percentage of subjects with BILAG-2004 flares will be presented and derived based on the number of subjects in the mITT population.

Furthermore, at Week 24 and Week 48, the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% CI of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be also presented for each flare category. 95% CI for the difference between active treatment and placebo will be based on the CMH test stratified by geographic region. In addition, the associated p-value will be provided.

# 8.2.16mSLEDAI-2K Flare (mSFI)

The number of subjects with mSLEDAI-2K flare between Baseline and Week 24, and between Baseline and Week 48 (see Section 17.4 for details) will be presented by category (mild/moderate and severe). The percentage of subjects with mSLEDAI-2K flares will be presented and derived based on the number of subjects in the mITT population.

Furthermore, at Week 24 and Week 48, the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% CI of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be also presented for each flare category. 95% CI for the difference between active treatment and placebo will be based on the CMH test stratified by geographic region. In addition, the associated p-value will be provided.

### 8.2.17 Prednisone Equivalent Total Daily Dose

The prednisone equivalent total daily dose at Week 12, Week 24 and Week 48 will be presented. The total daily dose at Baseline will be the sum of the Prednisone equivalent dose of steroids taken on the date the first dose of study drug was administered. The total daily dose will be derived as described in Section 17.9.

In addition, at each post-Baseline visit, the change from baseline and percent change from Baseline will be modelled using an ANCOVA model with treatment as factor and Baseline and geographic region as covariates. The LSMeans and SE of the LSMeans will be presented at each visit alongside the 95% CI. The difference in LSMeans between each of the active treatment groups and placebo will be presented with the associated 95% CI.

#### 8.2.18 Reduction Rate in Steroids Intake Without Severe Flare

The number and percentage of subjects whose prednisone equivalent dose was >7.5 mg/day at Baseline and  $\le 7.5$  mg/day between Week 40 to 48 without experiencing a severe mSFI-defined or severe BILAG-2004flare after the first decrease in prednisone equivalent dose and up to and including Week 48 cut-off date will be summarized. Percentages will be based on subjects in the mITT population whose prednisone equivalent dose was >7.5 mg/day at Baseline. The duration of flare assessment time which is starting from the date of first decrease in prednisone equivalent dose up to and including Week 48 cut-off date will be summarized.

Furthermore, the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% CI of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be presented. 95% CI for the difference between active treatment and placebo will be based on the CMH test stratified by geographic region. In addition, the associated p-value will be provided.

#### 8.2.19 Discontinuation Rate in Steroids Intake without Severe Flare

The number and percentage of subjects who are able to permanently discontinue prednisone (or equivalent) before or on Week 48 without experiencing a severe mSFI-defined or severe BILAG-2004-defined flare after the first decrease in prednisone equivalent dose and up to and including Week 48 cut-off date (see Section 17.5.1). Percentages will be based on subjects in the mITT population who took steroids at Baseline. The duration of flare assessment time which is starting from the date of first decrease in prednisone equivalent dose up to and including Week 48 cut-off date will be summarized.

Furthermore, the Clopper Pearson 95% CI of the incidence rate (expressed in percentage) and the 95% CI of the difference in incidence rate between each active treatment group and placebo (i.e. active treatment – placebo) will be also presented. 95% CI for the difference between active treatment and placebo will be based on the CMH test stratified by geographic region. In addition, the associated p-value will be provided.

Details of the derivation of prednisone equivalent dose can be found in Section 17.9.

# 8.2.20SF-36 Physical and Mental Component

SF-36 physical and mental component scores (see Section 17.10 for details) at Week 24 and at Week 48 will be summarized.

In addition, at each post-Baseline visit and for each component separately, the change from Baseline will be modelled using an ANCOVA model with Baseline and geographic region as covariates and treatment as factors. The LSMeans and SE of the LSMeans will be presented at each visit alongside the 95% CI. The difference in LSMeans between each of the active treatment group and placebo will be presented with the associated 95% CI.

#### 8.2.2128-Joint Count

The 28-Joint count swollenness and tenderness (see Section 17.11 for details) at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48 will be summarized.

In addition, at each post-Baseline visit and for 28-Joint count swollenness, tenderness separately, the change from Baseline will be modelled using an ANCOVA model with treatment as factor and Baseline and geographic region as covariates. The LSMeans and SE of the LSMeans will be presented at each visit alongside the 95% CI. The difference in LSMeans between each of the active treatment group and placebo will be presented with the associated 95% CI.

#### 8.2.22CLASI

The CLASI will be performed in interested sites having experience in this assessment. The CLASI activity and damage scores (see Section 17.12 for details) at Week 12, 24 and Week 48 will be summarized.

In addition, at each post-Baseline visit and for CLASI activity and damage scores separately, the change from Baseline will be modelled using an ANCOVA model with treatment as factor and Baseline and geographic region as covariates. The LSMeans and SE of the LSMeans will be presented at each visit alongside the 95% CI. The difference in LSMeans between each of the active treatment group and placebo will be presented with the associated 95% CI.

# 9 Safety Analysis

All safety summaries will be based on the Safety population and presented by treatment group and for the "All ALX-0061" group.

For laboratory parameters, vital signs and ECG, visits will be mapped to analysis visits using the rules defined in Section 17.16. Summaries will be based on those analysis visits.

Any abnormal laboratory test results, vital signs and/or ECG, including those that worsen from Baseline, believed to be clinically significant in the medical and scientific judgment of the investigator are recorded and analyzed along with other collected AEs or SAEs.

### **9.1 Adverse Events**

An AE is defined as any untoward medical occurrence in a subject enrolled into the study, regardless of its causal relationship to study drug. A treatment-emergent AE (TEAE) is defined as an AE that meets any of the following conditions:

- · begins on or after the first dose of study drug;
- begins before the first dose of study drug and worsens in severity on or after the first dose of study drug;
- begins on the first dose date of study drug and onset time is missing;
- onset date and end date are completely missing;
- onset date is completely missing and the end date is on or after the date of the first dose of study drug.

For the purpose of inclusion in TEAE tables, incomplete AE onset and end dates will be imputed as described in Section 17.15.

All AEs will be classified by System Organ Class (SOC) and PT according to the MedDRA version that is current at the time of the database lock.

An overview summary of the number of events, the subjects and percentage of subjects within the following categories will be provided by treatment group.

- Any TEAE,
- Any Severe TEAE
- Any study drug-related TEAE,
- Any TEAE leading to treatment discontinuation,
- Any serious TEAE,
- Any study drug-related serious TEAE,
- Any serious TEAE leading to treatment discontinuation,
- Any injection-site related TEAE,
- Any study drug-related injection-site related TEAE,
- · Any serious injection-site related TEAE,
- Any study drug-related serious injection-site related TEAE,
- Any TEAE of special interest,
- Any study drug-related TEAE of special interest,
- Any serious TEAE of special interest,
- Any study drug-related serious TEAE of special interest,
- Any TEAE leading to death.

A TEAE will be categorized as study drug-related if the relationship to the study drug is reported to be 'Possibly Related', or 'Related' as collected on the Adverse Events CRF page, or missing.

Tabulated listings for the following category will be provided:

- AE leading to death,
- SAE,
- AE leading to treatment discontinuation

In addition to the listing of all AEs, a listing for adverse events of interest will be provided.

TEAEs will be presented by SOC and PT and will be sorted in descending order from the SOC with the highest total incidence (that is, summed across all treatment groups) to the SOC with the lowest total incidence. If the total incidence for any two or more SOCs is equal, the SOCs will be presented in alphabetical order. Within each SOC, the PTs will be presented in the same manner as the SOC, i.e. in descending order from the PT with the highest total incidence.

## 9.1.1 Incidence of Adverse Events

Summaries of the number of TEAEs and the number and percentage of subjects with any TEAE will be provided by treatment group. The TEAEs will be presented by SOC and PT.

Similar summaries for subjects with any non-serious TEAE and for subjects with any serious TEAE will be provided.

At each level of subject summarization, a subject is counted once if the subject reported one or more events. Percentages will be calculated out of the number of subjects in the relevant treatment group.

### 9.1.2 Relationship of Adverse Events to Study Drug

Summaries of the number of study drug-related TEAEs and the number and percentage of subjects with any study drug-related TEAE will be provided by treatment group. The study drug-related TEAEs will be presented by SOC and PT.

At each level of subject summarization, a subject is counted once if the subject reported one or more events. TEAEs with missing relationship will be included in the summary of study drug-related TEAE and will be presented in the data listing with a missing relationship. Percentages will be calculated out of the number of subjects in the relevant treatment group.

### 9.1.3 Severity of Adverse Event

Summaries of number and percentage of subjects with any TEAE will be provided by treatment group and by severity (Mild, Moderate and Severe). The TEAEs will be presented by SOC, PT and severity.

At each level of subject summarization, a subject is counted once if the subject reported one or more events. If a subject reported multiple occurrences of the same TEAE, only the most severe will be presented. TEAEs with missing severity will be presented in tables under 'Missing' row and in the data listing with a missing severity. Percentages will be calculated out of the number of subjects in the relevant treatment group.

#### 9.1.4 Serious Adverse Events

Summaries of the number of serious TEAEs and the number and percentage of subjects with any serious TEAE will be provided by treatment group. These TEAEs will be presented by SOC and PT.

Summaries of the number of study drug-related serious TEAEs and the number and percentage of subjects with any study drug-related serious TEAE will be provided by treatment group. The study drug-related serious TEAEs will be presented by SOC and PT.

Summaries of number and percentage of subjects with any serious TEAE will be provided by treatment group and by severity (Mild, Moderate and Severe). The serious TEAEs will be presented by SOC, PT and severity.

### 9.1.5 Adverse Events Leading to Treatment Discontinuation

Summaries of the number of TEAEs leading to treatment discontinuation and the number and percentage of subjects with any TEAE leading to treatment discontinuation will be provided by treatment group. These TEAEs will be presented by SOC and PT. An AE leading to treatment discontinuation is an AE for which the action with regards to study drug was recorded as 'Drug withdrawn' on the CRF.

### 9.1.6 Adverse Event of Special Interest (AESI)

#### **Injection-site reaction**

An injection-site reaction is an AE that occurred at the location of the study drug administration. Using the start date and the location of the injection-site reaction (for TEAE recorded as injection-site reaction in the CRF and related to study drug administration), each injection-site reaction will be associated to the material injected at the site of the injection-site reaction (Placebo or ALX-0061) immediately prior to start of the AE.

Within each treatment group, study drug-related injection-site reactions will be summarized according to the material injected at the site of the ISR (i.e. ALX-0061 or

placebo). Summaries of the number of study drug-related injection-site reactions and the number and percentage of subjects with any study drug-related injection-site reaction will be provided by treatment group. These TEAEs will be presented by PT and will be sorted in descending order.

### Hypersensitivity

Summaries of the number and percentage of subjects with any hypersensitivity will be provided by treatment group and by severity (Mild, Moderate and Severe). These TEAEs will be presented by SOC and PT.

In addition, summary of treatment-emergent adverse event of hypersensitivity leading to treatment discontinuation will be provided and will present the number of treatment-emergent events of hypersensitivity leading to treatment discontinuation and the number and percentage of subjects with any treatment-emergent event of hypersensitivity leading to treatment discontinuation by treatment group. These TEAEs will be presented by SOC and PT.

**Note:** Hypersensitivity, Anaphylactic reaction and Angioedema Standardized MedDRA Queries (SMQs) with a narrow search will be used to determine hypersensitivity reactions (see Section 17.18).

Samples collected upon occurrence of serious and/or severe hypersensitivity reactions will be analyzed in the ADA and/or mADA assay (see Section 12) and optionally for the biomarkers tryptase and CH50. A listing of these serious and/or severe hypersensitivity adverse events will be presented, including ADA/mADA  $log_{10}(titer)$  and tryptase and CH50 test results.

#### Other AESI:

The Other Adverse Events of Special Interest are:

- Infections
- Serious Infections
- Opportunistic infections (excluding Tuberculosis [TB])
- Active TB
- Latent TB
- Herpes zoster infection
- Malignancies
- Lymphoma
- Gastrointestinal (GI) perforation
- Demyelinating disorder
- Major adverse cardiac events (MACE)

The number of treatment-emergent AESI and the number and percentage of subjects with any treatment-emergent AESI will be provided by treatment group for each of the AESI above.

**Note:** Search criteria for AESI are included in Section 17.18.

#### 9.1.7 Death

Summaries of the number of TEAEs leading to death and the number and percentage of subjects with any TEAE leading to death will be provided by treatment group. These TEAEs will be presented by SOC and PT and will be sorted in descending order for SOC

and PT. An AE leading to death is an AE for which the outcome was recorded as 'Death Related to Adverse Event' on the CRF.

# 9.2 Clinical Laboratory Evaluations

International Normalized Ratio (INR) (collected for subjects taking vitamin K antagonist) and Coombs' test (collected for all subjects) will be performed by local laboratories; other laboratory assessments will be performed by a central laboratory. All summaries will be based on the international system of units (SI) units provided by the central laboratory, no conversion will be done (see Section 17.14 for the tests to be reported and units).

Unless otherwise specified, if a laboratory value is reported using a non-numeric qualifier (e.g., less than [<] a certain value, or greater than [>] a certain value), the given numeric value will be used in the summary statistics, ignoring the non-numeric qualifier.

## 9.2.1 Haematology, Blood Chemistry, Lipid Profile and Coagulation

The following parameters will be summarized and displayed at the scheduled time points (see Section 17.1). For lipid profile parameters only fasting values will be summarized (i.e. if the sample was not marked as fasting, the associated results will not be used in the summary)

- Haematology: Leukocytes, Erythrocytes, Haemoglobin, Haematocrit, Platelets (recorded as Thrombocytes), Absolute Lymphocytes, Absolute Monocytes, Absolute Eosinophils, Absolute Basophils, Absolute Neutrophils, Mean Corpuscular Volume, Mean Corpuscular Haemoglobin and Mean Corpuscular Haemoglobin Concentration,
- Blood Chemistry: Total Bilirubin, Alkaline Phosphatase, Gamma Glutamyltransferase (GGT), Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Lactate Dehydrogenase, Creatine Phosphokinase, Urea, Total Protein, Albumin, Glucose, Inorganic Phosphate, Sodium, Potassium, Calcium and Chloride,
- Lipid Profile (fasting): Total Cholesterol, HDL-cholesterol, LDL/cholesterol, LDL/HDL-cholesterol ratio and Triglycerides
- Coagulation: activated Partial Prothrombin Time and Prothrombin Time.

Summary tables presenting observed numeric values and changes from Baseline (where applicable) will be provided for clinical laboratory tests with numeric values by treatment group for subjects in the Safety population.

Box plots of the change from Baseline at each post-Baseline visit will be presented for all central laboratory parameters by treatment group.

All relevant clinical laboratory tests will be classified as Low, Normal, and High according to the normal ranges; for selected lab parameters (see Section 17.20), directional National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events CTCAE grades) will be presented instead. These categorical data will be summarized in shift tables comparing the results (Low, Normal, High and for selected tests, Grade 0, Grade 1, Grade 2, Grade 3, Grade 4) at each post-Baseline visit with those at the Baseline visit. In addition, worst on-treatment post-Baseline excluding those taken more than 25 days after last dose of treatment will also be presented. Missing laboratory values will not be analysed in shift tables.

**Note:** Only patients consented under protocol version 3.0 (dated 16-May-2016) or subsequent protocol amendments have results for Creatine Phosphokinase test. This parameter will not be summarized separately.

### 9.2.2 Urinalysis

Proteinuria as measured by spot urine protein/creatinine ratio and urine sediment will be summarized as part of the efficacy endpoints.

### 9.2.3 Laboratory Parameters of Special Interest

The incidence rate of the following events will be provided by treatment group based on the Safety population. A subject will be counted in a category if he/she experienced the event at any time after the first dose of study drug up to 25 days after the last dose date. The percentage will be derived based on the number of subjects with at least one non-missing post-Baseline value for the considered parameter. If the criterion is based on change from Baseline, only subjects with non-missing Baseline results for the considered parameters will be considered in the table.

- Increase from Baseline in LDL Cholesterol ≥ 20 %,
- ALT > 3 x ULN and/or AST > 3 x ULN,
- Thrombocytopenia (platelets <100 x109/L),
- Neutropenia (absolute neutrophils count <0.500 x10<sup>9</sup>/L),
- Neutropenia (absolute neutrophils count 0.5-1.0 x10<sup>9</sup>/L),
- Neutropenia (absolute neutrophils count 1.0-1.5 x10<sup>9</sup>/L),
- Complement deficiency (C3, C4 or CH50 < LLN),</li>
- Increase from Baseline in proteinuria (protein / creatinine ratio) ≥ 20 %,
- Increase from Baseline in serum creatinine ≥ 26.52 μmol/L or ≥ 50 %,
- Urinary cast scored '4' from SLEDAI,
- Decrease from Baseline in eGFR ≥ 20 %,
- Hy's law: AST or ALT >3x ULN and total bilirubin > 2x ULN and alkaline phosphatase <2x ULN.</li>

#### 9.2.4 Coombs' test

Coombs' test results (positive and negative) will be summarized at the scheduled time points (see Section 17.1) by way of frequency count and percentages. Percentages will be based on the number of subjects who have no missing results.

#### 9.2.5 INR

INR test is locally performed for subjects taking Vitamin K antagonist at the scheduled time points (see Section 17.1). Subjects taking or not taking vitamin K antagonist at each visit is collected on the "Local Laboratory" CRF page.

INR will be classified as Low, Normal, and High according to the normal ranges. These categorical data will be summarized at Baseline and each post-Baseline visit. In addition worst on-treatment post-Baseline excluding those taken more than 25 days after last dose of treatment will also be presented (see Section 17.21 for definition of worst ontreatment). Percentages will be calculated based on the number of subjects for which the INR test was performed at the corresponding visit.

#### 9.2.6 Antibodies

### **Anti-nuclear Antibodies (ANA)**

At Baseline, frequency count and percentage of subjects with positive and negative results for ANA will be presented by treatment groups. For the subjects with positive ANA test results, the following summaries will be provided:

- Frequency count and percentages of subjects with each possible pattern of antibodies (atypical speckled, speckled, nucleolar, centromere and homogeneous, etc.); percentages will be based on the number of subjects with positive ANA results.
- Frequency count and percentages of subjects with titer below and above quantification limit; percentages will be based on the number of subjects with positive ANA results.
- Descriptive statistics (n, mean, median, SD, minimum, maximum, coefficient of variation [CV%], geometric mean, geometric SD, 5% and 95% percentiles). The descriptive statistics will only be provided if ≥ 20% of the subjects in the treatment group have positive ANA results.

The CV% is calculated as follows: CV% =  $\frac{SD}{mean} \times 100$ .

Geometric CV% is calculated as follows: Geometric CV% =  $100 \times \sqrt{(\exp(\sigma^2) - 1)}$ , where  $\sigma^2$  denotes the variance of the log-transformed values.

Geometric mean is calculated as follows:  $\mu_g = \exp\left(\frac{\sum_{i=1}^n \ln x_i}{n}\right)$  where  $x_i$  is the individual titer at current visit.

The Geometric SD is calculated as follows:  $\exp \sqrt{\frac{\sum_{i=1}^n (\ln x_i - \ln \mu_g)^2}{n}}$ 

For the descriptive statistics, the following rules will be used:

- Titres recorded as <1:80 or negative will be imputed as 40,
- Titres recorded as >1:1280 will be imputed as 1280,
- Titres recorded as 1:X where X is the dilution factor, will be converted to X (i.e. just the dilution factor).

# Other Antibodies:

The following antibody parameters will be summarized and displayed:  $\beta$ 2-glycoprotein 1 IgG,  $\beta$ 2-glycoprotein 1 IgM, anti-cardiolipin IgA, anti-cardiolipin IgG, anti-cardiolipin IgM and anti-lupus antibodies at Baseline and Week 24.

Summary tables presenting observed numeric values and changes from Baseline will be presented as well as the percentages of subjects below and above quantification limit (percentages will be based on the number of subjects with no missing data at the considered visit) for subjects in the Safety population.

### 9.3 Vital Sign Measurements

Summary tables presenting observed values at Baseline, each post-Baseline visit as well as changes from Baseline will be presented for all vital signs parameters (systolic blood pressure, diastolic blood pressure, temperature [converted to Celsius], pulse and weight [converted to kilogram]), by treatment group for subjects in the Safety population.

Statistical Analysis Plan, Final Version 1.0 Date Issued: 28FEB2018

Box plots of the change from Baseline at each post-Baseline visit will be presented for all vital signs parameters (systolic blood pressure, diastolic blood pressure, temperature, pulse and weight), by treatment group.

Temperature in degrees Fahrenheit will be converted to Celsius using the following formula:

Temperature (°C) = (Temperature (°F) - 32)  $\times$  5/9.

Weight in pounds will be converted to kilograms using the following formula:

Weight (kg) = Weight (lbs)  $\times$  0.4536.

# 9.4 Physical Examination

Abnormal findings in physical examinations will be listed. No summaries will be provided.

# 9.5 Electrocardiogram

A summary table presenting observed values at Baseline and at Week 48 and changes from Baseline will be provided for all ECG parameters (heart rate, RR interval, PR interval, QRS duration, QT interval, QT corrected Bazett (QTcB) and QT corrected Fridericia (QTcF)), by treatment group for subjects in the Safety population.

QT corrected Bazett and QT corrected Fridericia will be derived using the following formulae:

$$QTcB = \frac{QT}{\sqrt{RR}}$$

$$QTcF = \frac{QT}{\sqrt[3]{RR}}$$

#### 9.6 Other Safety Data

#### 9.6.1 Tuberculosis Assessment

TB assessments will be listed and not summarized.

#### 9.6.2 Pregnancy test

Pregnancy tests for females of childbearing potential will be listed.

# 10 Pharmacokinetics (PK)

PK analysis will be performed on the Safety population.

Drug concentrations will be summarized by treatment group using descriptive statistics (n, mean, median, SD, minimum, maximum, CV%, geometric mean, geometric SD, 5% and 95% percentiles). In general, geometric mean and the geometric SD will be derived from non-zero concentration values. These results will be tabulated by treatment group and visit (Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48).

The CV% is calculated as follows:  $CV\% = \frac{SD}{mean} \times 100$ .

Geometric mean is calculated as follows:  $\mu_g = \exp\left(\frac{\sum_{i=1}^n \ln x_i}{n}\right)$  where  $x_i$  is the individual drug concentration at current visit.

The Geometric SD is calculated as follows:  $\exp \sqrt{\frac{\sum_{i=1}^n (\ln x_i - \ln \mu_g)^2}{n}}$ 

Individual pharmacokinetic concentrations will be reported and listed in  $\mu g/mL$  (i.e. the concentrations reported as ng/mL will be converted to  $\mu g/mL$  by dividing the concentrations by 1000).

Individual pharmacokinetic concentrations below the limit of detection or below the quantification limit (BQL) will be reported as BQL. To compute descriptive statistics (i.e. mean [or median or geometric mean], SD, CV%, geometric SD, minimum, maximum, 5% and 95% percentiles), all BQL values will be treated as missing. When the total number of BQL values exceeds 1/3 of the total number of values at that time point, descriptive statistics will not be calculated. Descriptive statistics not calculated for the above reasons will be reported as not calculated (NC) in the associated table. In case the actual sampling time deviates more than allowed per study protocol from the nominal time (i.e. the sample should be prior to the dosing on that visit and within  $\pm 5$  days if the scheduled visit date, see Section 17.16), these samples will not be included in the calculation of descriptive statistics on pharmacokinetic concentrations and associated plots.

The following figures will be provided by treatment groups (linear and semi-logarithmic plots will be displayed on the same page):

- Spaghetti plot of Individual subjects concentration (linear scale) over time;
- Spaghetti plot of Individual subjects concentration (semi-logarithmic scale) over time;
- Mean and ± SE of concentration (linear scale) over time plot;
- Mean of concentration (semi-logarithmic scale) over time plot.
- Geometric mean ± geometric SD of concentration (linear scale) over time plot;
- Geometric mean of concentration (semi-logarithmic scale) over time plot.

For individual spaghetti plots, nominal sampling times are used, unless the actual time deviates more than allowed per study protocol. In that case the actual time is used.

A listing of the actual sampling times will be presented. Actual sample time that deviated from the protocol allowed window will not be assigned an analysis visit in the listing.

# 11 Pharmacodynamics (PD)

#### **Evaluations of PD**

The biomarkers results and percent change from Baseline will be summarized over time by treatment groups based on the Safety population using descriptive statistics (n, mean, median, SE, minimum, maximum, CV%, geometric mean, geometric SD, 5% and 95% percentiles [see Section 10 for details on CV%, geometric mean and geometric SD derivation]). To compute descriptive statistics (i.e. mean [or median or geometric mean], SD, CV%, geometric SD, minimum, maximum, 5% and 95% percentiles), all BQL values will be treated as missing. For percent change from baseline, CV%, geometric mean and geometric SD will not be provided. The biomarkers evaluated are:

- sIL-6R: at Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48 and Follow-up.
- CRP, Fibrinogen, anti-dsDNA (FARR), C3, C4 and CH50: at Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48 and Follow-up.
- uMCP-1 and uMCP-1/uCr: at Week 8, Week 24 and Week 48.

Finally, Fibrinogen will be classified according to NCI CTCAE. This categorical data will be summarized in shift tables comparing the results (Grade 0, Grade 1, Grade 2, Grade 3, Grade 4) at each post-Baseline visit (included worst on-treatment) with those at the Baseline visit. Worst on-treatment post-Baseline results exclude the samples taken more than 25 days after last dose of treatment (see Section 17.21 for definition of worst-on-treatment).

**Note:** during the study, the testing of anti-dsDNA was switched from ELISA assay to an FARR assay, therefore FARR assay will be used in the summaries, the ELISA assay results will only be listed. If results are recorded as '<' or '>', the same handling rules as the safety laboratory data will be used (see Section 9.2).

In addition, for each biomarker the following graphical representation will be provided by treatment group:

- Mean and ± SE of biomarkers results (linear scale) over time plot (all treatments on the same page);
- Mean of biomarkers results (semi-logarithmic scale) over time plot, (all treatments on the same page);

#### **Exposure-response Model(s)**

Exposure-response modelling will be described in a separate Data Analysis Plan, and will be performed under the responsibility of Ablynx NV. Results of this analysis will be provided in a separate Modelling and Simulation report. Pooled data from other studies might be included as well.

# 12 Immunogenicity

Samples for immunogenicity are collected for all subjects during the study.

The ADA assay will detect treatment emergent (TE) ADA as well as pre-existing antibodies (pre-Ab). However, using the ADA assay, sensitive detection of TE ADA might be defied in subjects presenting pre-Ab. Therefore, the mADA characterization assay will be implemented for subjects classified as equivocal ([EQ], TE ADA status remains uncertain due to presence of pre-Ab; no significant titer increase upon dosing) to enable

detection of TE ADA in presence of pre-Ab and will be implemented as additional tier after the conventional ADA assay.

The immunogenicity samples are evaluated to determine if they are positive or negative in the ADA assay (tiered analysis in screening and confirmatory assay); only samples confirmed as positive in the ADA assay are titrated and they are reported as  $\log_{10}(\text{titer})$ . Samples scoring negative in the ADA assay are not titrated and the respective titer is reported as  $< \log_{10}(\text{MRD})$  with Minimal Required Dilution (MRD) = 100, i.e.  $\log_{10}(\text{titer})$  <2.00.

Only subjects which are classified as "pre-Ab positive – equivocal" in the ADA assay will have their samples analyzed in the mADA assay; similarly to the ADA assay, only positive samples in the mADA assay (i.e. confirmed as positive) are titrated and are reported as log<sub>10</sub>(titer).

In addition, subjects presenting positive ADA samples, will have their samples (positive ADA samples) analyzed in the qualitative NAb assay (reported as the normalized assay result [i.e. ratio sample assay result/negative control assay result]). A subset of the available pre-dose samples will be analyzed in the NAb assay to evaluate the study-specific cut-point for the NAb assay. Subjects scoring negative in the NAb assay will be reported as 'neg' result.

- Subjects will be classified based on ADA assay results and mADA assay results (if applicable), separately, and will receive an overall subject classification as specified in the Table 12-1. No mADA subject classification will be attributed in case the subject was not analyzed in the mADA assay.
- Subjects will be classified based on their NAb pre-dose status and status on treatment as specified in the Table 12-2. Subjects with no positive ADA samples post-dose will be classified as 'Negative on treatment' by default.

No records will be reported for samples not evaluated in the mADA assay. Also, for samples not evaluated in the NAb assay (i.e., ADA negative samples), no records will be reported. These unavailable NAb records, for which the corresponding ADA record is negative, should be considered NAb negative in all further incidence calculations. Patients from which all time points are ADA negative should be classified per default as "Pre-dose neg – neg on treatment" in the NAb assay.

Table 12-1: ADA, mADA and Overall Subject Classification

| ADA Assay | mADA Assay | Overall Subject Classification |
|---------------------|---------------------|--------------------------------|
| Classification | Classification | |
| MISSING | | MISSING |
| PRE-AB NEG - TE NEG | | PRE-AB NEG - TE NEG |
| PRE-AB NEG - TE POS | | PRE-AB NEG - TE POS |
| PRE-AB NEG - TE | | PRE-AB NEG - TE INCONCLUSIVE |
| INCONCLUSIVE | | |
| PRE-AB POS - TE NEG | | PRE-AB POS - TE NEG |
| PRE-AB POS - TE POS | | PRE-AB POS - TE POS |
| PRE-AB POS - TE | | PRE-AB POS - TE INCONCLUSIVE |
| INCONCLUSIVE | | |
| PRE-AB POS – EQ | PRE-AB NEG - TE POS | PRE-AB POS - TE POS |
| | PRE-AB POS - TE POS | PRE-AB POS - TE POS |
| | PRE-AB NEG - TE NEG | PRE-AB POS – EQ |
| | PRE-AB POS - EQ | PRE-AB POS – EQ |
| | PRE-AB POS - TE NEG | PRE-AB POS – EQ |
| | PRE-AB NEG - TE | PRE-AB POS - TE INCONCLUSIVE |
| | INCONCLUSIVE | |

| ADA Assay<br>Classification | mADA Assay<br>Classification | Overall Subject Classification |
|---|---|---|
| | PRE-AB POS - TE<br>INCONCLUSIVE | PRE-AB POS - TE INCONCLUSIVE |

#### Table 12-2: NAb Assay Classification

| NAb assay classification |
|--------------------------------|
| Pre-dose Neg, Neg on treatment |
| Pre-dose Neg, Pos on treatment |
| Pre-dose Pos, Neg on treatment |
| Pre-dose Pos, Pos on treatment |

#### 12.1 Available data

The following parameters will be summarized by treatment group:

- · ADA subject classification
- mADA subject classification (based on subset of subjects)
- Overall subject classification per subject (based on ADA and/or mADA analysis)
- NAb subject classification (based on subset of subjects)

Note that, for immunogenicity, screening and baseline visits are derived based on the CRF visit label.

#### 12.1.1 ADA and mADA

The following 2 populations will be defined and used where specified in the summary statistics:

- **Pre-Ab negative population**: includes all the subjects who had all their available pre-dose titers (Screening and/or Baseline) reported as <2.00.
- **Pre-Ab positive population**: includes all the subjects with at least one pre-dose log<sub>10</sub>(titer) reported as a numeric value equal to or above 2.00.

### **ADA Subject Classification:**

The incidence rate (number and percentage of subjects) of pre-Ab status (negative, positive and total) versus treatment-emergent ADA status (TE negative, TE positive, TE inconclusive and equivocal) will be presented by treatment group and by all ALX-0061 treated subjects. The percentages will be based on the number of subjects within each treatment group, excluding the subjects who are classified as missing.

In addition, the incidence rate of pre-Ab status (negative, positive and total) versus treatment-emergent ADA/mADA positive status (TE negative, TE positive, TE inconclusive and equivocal) will be presented for both the pre-Ab negative and positive populations. The percentages will be based on the number of subjects within each treatment group in the subpopulations (i.e., pre-Ab negative and pre-Ab positive), excluding the subjects who are classified as missing.

The following subject categories will be used in the table:

- Pre-Ab Negative TE Negative
- Pre-Ab Negative TE Positive

- Pre-Ab Negative TE inconclusive,
- Pre-Ab Positive TE Negative,
- Pre-Ab Positive TE Positive,
- Pre-Ab Positive Equivocal,
- Pre-Ab Positive TE inconclusive,
- Total Pre-Ab Negative ("Pre-Ab Negative TE Negative", "Pre-Ab Negative TE Positive" and "Pre-Ab Negative TE inconclusive"),
- Total Pre-Ab Positive ("Pre-Ab Positive TE Negative", "Pre-Ab Positive TE Positive", "Pre-Ab Positive Equivocal" and "Pre-Ab Positive TE inconclusive"),
- Total TE Negative ("Pre-Ab Negative TE Negative" and "Pre-Ab Positive TE Negative"),
- Total TE Positive ("Pre-Ab Negative TE Positive" and "Pre-Ab Positive TE Positive"),
- Total TE inconclusive ("Pre-Ab Negative TE Inconclusive" and "Pre-Ab Positive TE Inconclusive"),
- Missing
- TE Positive within Pre-Ab Negative population
- TE Positive within Pre-Ab Positive population

#### mADA Subject Classification:

Similar summary (as for the ADA subject classification) will be provided for the mADA subject classification with exception that subjects will not be classified as missing.

### ADA/mADA Overall Subject Classification:

Similar summary (as for the ADA subject classification) will be provided for the overall subject classification.

#### 12.1.2NAb

The incidence rate of pre-dose status (negative, positive) versus NAb status on treatment (negative on treatment, positive on treatment) will be presented by treatment group. The percentages will be based on the number of subjects within each treatment group. For the pre-dose negative and pre-dose positive population, the percentages are based on the number of subjects within each treatment group in the subpopulation.

The following NAb subject categories will be used:

- Pre-dose negative negative on treatment
- Pre-dose negative positive on treatment
- Pre-dose positive negative on treatment
- Pre-dose positive positive on treatment
- Total Pre-dose Negative
- Total Pre-dose Positive

- Total negative on treatment
- Total positive on treatment
- Positive on treatment within Pre-dose negative population
- Positive on treatment within Pre-dose positive population

# 12.2 Subgroup analyses

The incidence rate of pre-Ab status (negative, positive and total) versus treatment-emergent ADA/mADA status (TE negative, TE positive, TE inconclusive and equivocal) will be presented by treatment group for the following subgroups. The percentages will be based on the number of subjects within each treatment group and subgroup, excluding the subjects who are classified as missing.

In addition, for the following subgroups, the incidence rate of pre-Ab status (negative, positive and total) versus treatment-emergent ADA/mADA positive status (TE positive) will be presented for both the pre-Ab negative and positive populations. The same classifications will be used as the ones outlined above (see ADA subject classifications).

- Injection-site reaction
  - No injection-site reaction
  - o At least 1 injection-site reaction
- · Hypersensitivity reaction
  - No hypersensitivity reaction
  - At least 1 hypersensitivity reaction

### 13 Interim Analysis

No interim analysis is planned for the study.

# 14 Data and Safety Monitoring Board (DSMB)

The Data and Safety Monitoring Board (DSMB) is an independent committee. None of the members are participating in the study. The major function of this committee is to monitor the safety of the subjects participating in the ALX-0061 clinical program by periodically reviewing unblinded safety data. They advise concerning continuation, modification or termination of study. The DSMB meets every 6 months to review the study data. PPD provides the blinded SDTM datasets to the company responsible to organize the DSMB.

The DSMB charter and DSMB SAP define and document the content of the safety summaries, the DSMB's role and responsibilities, and the general procedures (including communications).

# 15 Changes in the Planned Analysis

The following points are changes in analysis from the protocol.

- Primary endpoint: sensitivity analysis was added using the observed case data.
- SRI definition was updated by adding that a subject will be deemed to be nonresponder at any time point after treatment failure (including the premature discontinuation from study treatment) has been determined.

- Treatment failure definition was harmonized to exclude early discontinuation as the protocol was including early discontinuation in some of the references of treatment failure but not all, therefore early discontinuation was added to the following endpoints definitions:
  - BICLA and mBICLA
  - o SRI and mSRI
- Subgroup analyses for secondary endpoints (except mSRI at Week 24 and 48) and safety endpoints were not included.
- Subgroup summaries for mBICLA at Week 48 were added.
- Inferential statistics were added for all secondary endpoints.
- PK population was removed and Safety population was used instead.
- QTcB and QTcF were added in the list of ECG endpoints.
- Percent Change from Baseline in Daily Prednisone or Equivalent now includes Week 12 (in addition to Week 24 and Week 48).
- Change from Baseline in Daily Prednisone or Equivalent to Week 12, 24 and 48 was added.
- SE was used instead of SD for secondary endpoints (excluding PK and ANA data) and safety endpoints summaries.
- Shift tables from Baseline in NCI CTCAE or Ablynx defined grades for selected laboratory parameters (AST, ALT, serum Creatinine, eGFR, GGT, Total Cholesterol, Leukocytes, Absolute Lymphocytes, Absolute Neutrophils, Platelets, Fibrinogen and Proteinuria as measured by spot urine protein to creatinine ratio) were included.
- The following laboratory parameters have been added to the list of endpoints (and will be derived):
  - o Fasting LDL/HDL-cholesterol ratio
  - o UCr
- The following parameters will not be summarized:
  - o Plasma cells
  - o T-helper 17
  - o T regulatory cells

# 16 References

- Bretz, F., J.C. Pinheiro, and M. Branson. Combining multiple comparisons and modeling techniques in dose-response studies. Biometrics, 2005. 61(3): p. 738-48.
- 2. Isenberg, D.A., et al. BILAG 2004. Development and initial validation of an updated version of the British Isles Lupus Assessment Group's disease activity index for patients with systemic lupus erythematosus. Rheumatology, 2005. 44(7): p. 902-6.
- 3. Yee, C.S., et al. Numerical scoring for the BILAG-2004 index. Rheumatology, 2010. 49(9): p. 1665-9.
- 4. Yee, C.S., et al. BILAG-2004 index captures systemic lupus erythematosus disease activity better than SLEDAI-2000. Annals of the rheumatic diseases, 2008. 67(6): p. 873-6.

Statistical Analysis Plan, Final Version 1.0 Date Issued: 28FEB2018

- Gladman, D.D., D. Ibanez, and M.B. Urowitz. Systemic lupus erythematosus disease activity index 2000. The Journal of rheumatology, 2002. 29(2): p. 288-91.
- Uribe AG, et al. The Systemic Lupus Activity Measure-revised, the Mexican Systemic Lupus Erythematosus Disease Activity Index (SLEDAI), and a modified SLEDAI-2K are adequate instruments to measure disease activity in systemic lupus erythematosus. The Journal of rheumatology, 2004 Oct; 31(10): p. 1934-1940.
- 7. Illei, G.G., et al. Tocilizumab in systemic lupus erythematosus: data on safety, preliminary efficacy, and impact on circulating plasma cells from an open-label phase I dosage-escalation study. Arthritis and rheumatism, 2010. 62(2): p. 542-52.
- 8. Szepietowski, J.C., et al. Phase I, randomized, double-blind, placebo-controlled, multiple intravenous, dose-ascending study of sirukumab in cutaneous or systemic lupus erythematosus. Arthritis and rheumatism, 2013. 65(10): p. 2661-71.
- 9. Luijten, K.M., et al. The Systemic Lupus Erythematosus Responder Index (SRI); a new SLE disease activity assessment. Autoimmunity reviews, 2012. 11(5): p. 326-9.
- 10. Petri, M., J. Buyon, and M. Kim. Classification and definition of major flares in SLE clinical trials. Lupus, 1999. 8(8): p. 685-91.
- 11. Pinheiro J.C., Bornkamp B., Glimm E. and Bretz F. (2014) Model-based dose finding under model uncertainty using general parametric models, Statistics in Medicine, 33, 1646–1661.
- 12. Buckland, S. T., Burnham, K. P. and Augustin, N. H. (1997). Model selection an integral part of inference, Biometrics, 53, 603–618
- 13. Cresswell, L., et al. Numerical scoring of the Classic BILAG index. Rheumatology (Oxford). 2009 Dec; 48(12): 1548–1552.
- 14. Yee CS, Gordon C, Isenberg DA et al. The BILAG-2004 systems tally-a novel way of representing the BILAG-2004 index scores longitudinally. Rheumatology 2012; 51:2099-105.
- 15. Mehrotra DV. Railkar R. Minimum risk weights for comparing treatments in stratified binomial trials. Statistics in Medicine Vol 19 pp. 811-825, 2000.

# 17 Appendices

57

# 17.1 Schedule of Study Procedures<sup>a</sup>

| Study Period | Screening | Base-<br>line<br>(Day) | | | | | | | | | Trea | | | nd As<br>ek ± | | | ıt Pe | riod | | | | | | | | | Early<br>Termination<br>Visit | Follow-up<br>(± 2 weeks) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Visit | Within<br>28 days<br>prior to<br>baseline | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 | 26 | 28 | 30 | 32 | 34 | 36 | 38 | 40 | 42 | 44 | 46 | 48 | Within<br>3 weeks<br>after last<br>dosing | 12 weeks<br>after last<br>dosing |
| Written informed consent | × | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Demographics,<br>medical history | х | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Physical examination | × | х | | | | | | х | | | | | | х | | | | | | x | | | | | | х | х | х |
| Vital signs <sup>b</sup> | X | Х | х | х | Х | Х | Х | Х | | Х | | Х | | Х | | Х | | х | | х | | х | | Х | | Х | х | х |
| 12-lead ECG <sup>c</sup> | X | | | | | | | | | | | | | | | | | | | | | | | | | Х | х | |
| Screening Hep B,<br>Hep C, HIV <sup>d</sup> | x | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| IGRA test | X | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Chest radiograph <sup>e</sup> | X | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| TB evaluation <sup>f</sup> | | | | | | | | | | | | | | | | | | | | | | | | | | | | $\rightarrow$ |
| Review of entry<br>criteria | х | х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Prior medication | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Concomitant medication | | - | | | | | | | | | | | | | | | | | | | | | | | | | | > |
| Randomization | | X | | | | | | | | | | | | | | | | | | | | | | | | | | |
| ANA, LA, aCL,<br>β <sub>2</sub> -GPI <sup>g</sup> | x | | | | | | | | | | | | | х | | | | | | | | | | | | | | |
| Study drug allocation<br>and administration | | х | x | x | х | х | х | х | х | х | х | х | х | х | x | X | x | х | х | х | х | х | х | х | х | | | |
| SLEDAI-2K | X | X | | х | | Х | | Х | | х | | Х | | Х | | х | | х | | х | | х | | Х | | Х | x | |
| BILAG-2004 | X | X | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | x | |
| Physician's Global<br>Assessment | | х | | x | | х | | х | | х | | х | | х | | X | | x | | x | | х | | х | | х | х | |
| Patient's Global<br>Assessment | | х | | | | | | | | | | | | х | | | | | | | | | | | | х | х | |
| SF-36 | | Х | | | | | | | | | | | | Х | | | | | | | | | | | | Х | Х | |
| 28 joint count | Х | X | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | Х | |
| CLASI h | | X | | | | | | Х | | | | | | х | | | | | | | | | | | | х | x | |

| Study Period | Screening | Base-<br>line<br>(Day) | | | | | | | | | Trea | | | nd As<br>ek ± | | | | riod | | | | | | | | | Early<br>Termination<br>Visit | Follow-up<br>(± 2 weeks) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Visit | Within<br>28 days<br>prior to<br>baseline | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 | 26 | 28 | 30 | 32 | 34 | 36 | 38 | 40 | 42 | 44 | 46 | 48 | Within<br>3 weeks<br>after last<br>dosing | 12 weeks<br>after last<br>dosing |
| SLICC/<br>ACR damage score | | х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Adverse events <sup>i</sup> | | | | | | | | | | | | | | | | | | | | | | | | | | | | $\rightarrow$ |
| Clinical laboratory<br>analyses <sup>j</sup> | х | х | х | х | | х | | х | | х | | х | | х | | х | | х | | х | | x | | х | | х | х | × |
| Urinalysis | Х | Х | | Х | | Х | | Х | | х | | Х | | х | | Х | | х | | х | | Х | | Х | | х | x | |
| Pregnancy test<br>(serum at<br>screening/urine at<br>other visits) | х | х | | | | | | х | | | | | | х | | | | | | | | | | | | х | х | х |
| PK <sup>k</sup> | | х | х | Х | Х | Х | Х | Х | | Х | | х | | Х | | Х | | Х | | Х | | х | | Х | | Х | Х | |
| PD biomarker<br>(sIL-6R) <sup>k,</sup> | | х | | х | | х | | х | | x | | | | x | | | | х | | | | x | | | | х | х | х |
| PD biomarker<br>(others) <sup>k,l</sup> | х | х | | х | | х | | х | | х | | х | | х | | х | | х | | х | | х | | х | | х | × | х |
| Exploratory<br>biomarkers <sup>m</sup> | | х | | | | х | | | | | | | | х | | | | | | | | | | | | х | х | |
| Immunogenicity k,i | х | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | Х | | х | | Х | | Х | | Х | х | X |
| Local lab analyses<br>(Direct Coombs) <sup>n</sup> | х | х | | х | | х | | х | | х | | х | | х | | х | | х | | х | | x | | х | | х | х | |

If assessments are planned at the same time, following guidance should be followed: 1) ECG and vital signs should be assessed prior to blood sampling, 2) Patient assessments (patient's global assessment and SF-36) should occur prior to physician's assessments, 3) Study drug should be dosed after all other assessments have been performed.

b Vital signs (assessment after 5 min in supine position): including height, weight, blood pressure, pulse and temperature. Height measurement is only required at the screening visit.

<sup>&</sup>lt;sup>c</sup> To be performed after 5 min in supine position.

<sup>&</sup>lt;sup>d</sup> Lab tests for hepatitis B will be done according to the guidelines [2].

e If a chest radiograph has not been performed within 12 weeks prior to screening as part of standard of care, a chest radiograph must be performed during the screening period. In case local regulations do not allow radiographs during the study, a radiograph as part of standard of care should be available prior to screening.

If TB is suspected at any time during the study, chest radiography and IGRA or a comparable local practice test should be performed.

<sup>&</sup>lt;sup>g</sup> Lupus anti-coagulant (LA), anticardiolipin (aCL) and anti- $\beta_2$ -glycoprotein I ( $\beta_2$ -GPI) antibodies will be evaluated at screening and Week 24. Anti-nuclear antibodies (ANA) will be evaluated at screening only.

- The CLASI will be performed in interested sites having experience in this assessment.
- In case of acute or delayed severe/serious hypersensitivity reactions, an additional blood sample should be collected as soon as possible after the start of the event.
- On dosing days, blood sampling will be performed pre-dose. Subjects will be fasted for at least 10h at baseline and Weeks 4, 8, 12, 24, 36 and 48 and/or the Early Termination Visit for assessment of fasting serum lipids. Samples will be assessed by a central laboratory.
- K On dosing days, PK, PD biomarker and immunogenicity samples will be taken predose.
- CRP, fibrinogen, anti-dsDNA, C3, C4, CH50.
- <sup>m</sup> Urine samples for uMCP-1 will be collected in all subjects. Blood samples for immunophenotyping will be collected in a subset of subjects (at selected sites based on qualification).
- Parameters to be assessed by the local laboratory include Direct Coombs and INR (INR for subjects on vitamin K antagonist only). INR will be performed at Weeks 0, 2, 4, 8, and 12, and every 4 weeks (or more frequent if considered necessary by Investigator) thereafter up to Week 48 (or Early Termination Visit), and Follow-Up Visit.

# 17.2 Dosing Schedule

### Placebo (Group 1)

Syringe A with placebo (1 mL) q2w starting at Week 0 (Day 1), up to and including Week 46.

Syringe B with placebo (0.5 mL) q2w starting at Week 0, up to and including Week 46.

Table 17-1: Dosing schedule for Group 1

| | | | | | | | | | | | Vis | sit (\ | Veel | (s) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 | 26 | 28 | 30 | 32 | 34 | 36 | 38 | 40 | 42 | 44 | 46 |
| Placebo<br>1 mL | X | Х | X | X | X | X | X | X | Х | X | X | X | X | Х | Х | Х | X | Х | X | Х | X | X | X | Х |
| Placebo<br>0.5 mL | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | Х | Х | Х | X | Х |
| ALX<br>1 mL | | | | | | | | | | | | | | | | | | | | | | | | |
| ALX<br>0.5 mL | | | | | | | | | | | | | | | | | | | | | | | | |

### 75 mg q4w (Group 2)

Syringe A with placebo (1 mL) q2w starting at Week 0, up to and including Week 46.

Syringe B with ALX-0061 (0.5 mL) q4w at Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40 and 44, and syringe B with placebo (0.5 mL) q4w at Weeks 2, 6, 10, 14, 18, 22, 26, 30, 34, 38, 42 and 46.

Table 17-2: Dosing schedule for Group 2

| | | | | | | | | | | | Vis | sit (\ | Veel | ks) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 | 26 | 28 | 30 | 32 | 34 | 36 | 38 | 40 | 42 | 44 | 46 |
| Placebo<br>1 mL | X | X | Х | X | X | X | Х | X | X | X | X | Х | Х | X | X | Х | Х | X | X | X | X | X | X | X |
| Placebo<br>0.5 mL | | Х | | X | | Х | | X | | X | | Х | | Х | | Х | | Х | | X | | X | | X |
| ALX<br>1 mL | | | | | | | | | | | | | | | | | | | | | | | | |
| ALX<br>0.5 mL | Х | | Х | | Х | | Х | | Х | | X | | Х | | Х | | Х | | Х | | Х | | Х | |

# 150 mg q4w (Group 3)

Syringe A with ALX-0061 (1 mL) q4w at Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40 and 44, and syringe A with placebo (1 mL) q4w at Weeks 2, 6, 10, 14, 18, 22, 26, 30, 34, 38, 42 and 46.

Syringe B with placebo (0.5 mL) q2w starting at Week 0, up to and including Week 46.

Table 17-3: Dosing schedule for Group 3

| | | | | | | | | | | | Vis | sit (\ | Veel | ks) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 | 26 | 28 | 30 | 32 | 34 | 36 | 38 | 40 | 42 | 44 | 46 |
| Placebo<br>1 mL | | Х | | X | | Х | | Х | | X | | Х | | Х | | Х | | Х | | X | | Х | | Х |
| Placebo<br>0.5 mL | Х | Х | Х | X | Х | Х | Х | Х | Х | X | X | X | X | Х | X | Х | Х | Х | Х | X | X | X | X | Х |
| ALX<br>1 mL | Х | | Х | | Х | | Х | | Х | | X | | X | | X | | Х | | Х | | X | | Х | |
| ALX<br>0.5 mL | | | | | | | | | | | | | | | | | | | | | | | | |

# 150 mg q2w (Group 4)

Syringe A with ALX-0061 (1 mL) q2w starting at Week 0, up to and including Week 46. Syringe B with placebo (0.5 mL) q2w starting at Week 0, up to and including Week 46.

Table 17-4: Dosing schedule for Group 4



# 225 mg q2w (Group 5)

Syringe A with ALX-0061 (1 mL) q2w starting, at Week 0, up to and including Week 46. Syringe B with ALX-0061 (0.5 mL) q2w starting at Week 0, up to and including Week 46.

Table 17-5: Dosing schedule for Group 5

| | | | | | | | | | | | Vis | sit (\ | Veel | (s) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 2 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 | 26 | 28 | 30 | 32 | 34 | 36 | 38 | 40 | 42 | 44 | 46 |
| Placebo | | | | | | | | | | | | | | | | | | | | | | | | |
| 1 mL | | | | | | | | | | | | | | | | | | | | | | | | |
| Placebo | | | | | | | | | | | | | | | | | | | | | | | | |
| 0.5 mL | | | | | | | | | | | | | | | | | | | | | | | | |
| ALX | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| 1 mL | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ | ^ |
| ALX | V | Х | | Х | Х | Х | V | Х | V | V | V | V | V | V | V | Х | V | V | V | V | Х | V | V | Х |
| 0.5 mL | X | Α | X | ^ | ^ | Α | X | ^ | X | X | X | X | Χ | X | X | ^ | X | X | X | X | X | X | X | ^ |

#### 17.3 BILAG-2004

The BILAG-2004 [2-4] is a comprehensive composite clinical index that has been developed based on the principle of a physician's intention to treat using a nominal consensus approach. In the index, the nine systems (not organs) considered are: constitutional, mucocutaneous, neuropsychiatric, musculoskeletal, cardiorespiratory, gastrointestinal, renal, ophthalmic and haematological. Disease activity in each of the nine systems is categorized into five levels (Grades A-E). For the assessment of the BILAG-2004 scores, Coombs' test from local laboratory assessments will be used and all other laboratory parameters will be from the central laboratory. The BILAG-2004 version dated 2009 (latest validated version) will be used.

### 17.3.1BILAG-2004 Improvement (overall and individual):

BILAG-2004 improvement will be evaluated as normal and enhanced improvement and as improvement by individual organ system score.

- Normal improvement: all A scores at Baseline improved to B/C/D, and all B scores improved to C or D.
- **Enhanced improvement**: all A scores at Baseline improved to B/C/D, and all B scores improved to C or D and no worsening between consecutive visits from Baseline up to considered visit. For enhanced improvement if no more than one consecutive score is missing in visit(s) between the Baseline and the visit of interest for a considered organ system and no worsening is observed at the prior and subsequent visits it is assumed that the missing score is the same as the one at the prior visit.
- Improvement by individual organ system score: For each organ system, an
  improvement is defined as an A score at Baseline improved to B/C/D or a B score
  improved to C or D.

#### 17.3.2BILAG-2004 Total Score:

BILAG total score is derived by assigning the following value to each grade [3] and summing the scores over all organ systems:

- A = 12,
- B = 8,
- C = 1,
- D/E = 0.

#### 17.3.3BILAG-2004 Systems Tally:

BILAG-2004 system tally (BST) [14] is derived by classifying changes in the BILAG-2004 index system scores, using counts of systems with specified transitions in scores. It records the number of systems in which activity increased, decreased or remained the same between two consecutive visits and expresses this as a tally. It has the following six components:

- Major deterioration: change from grade B/C/D/E to A or grade D/E to B
- *Minor deterioration*: change from grade C to B
- **Persistent significant activity**: no change from grade A or B
- Major improvement: change from grade A to C/D or grade B to D
- Minor improvement: change from grade A to B or grade B to C

Persistent minimal or no activity: change from grade C/D/E to C/D/E

BST was further simplified into three components (simplified BILAG-2004 systems tally, sBST) by grouping major deterioration, minor deterioration and persistent activity into a single group, and major improvement with minor improvement into a separate group. The simplified version of the BST will be used in the study.

- Active/worsening disease: systems with major deterioration, minor deterioration or persistent significant activity
- Improving disease: systems with major improvement or minor improvement
- Persistent minimal or no activity.

#### 17.3.4BILAG-2004 Flare Index:

Using the BILAG-2004 score, severe and mild/moderate flares are defined as follows:

- Severe flare defined as a new A score in any system of the BILAG-2004 index following a B, C, D or E score at the previous assessment.
- Mild/moderate flare defined as a new B score following a C, D or E score at the previous assessment.

Flares will be evaluated from Baseline up to Week 24 and from Baseline up to Week 48.

# 17.3.5BILAG-2004 Scoring System:

The BILAG-2004 scoring system is based on the physician's intention to treat.

| Grade | Definition |
|---|---|
| A | Severe disease activity requiring any of the following treatment: |
| | <ol> <li>Systemic high dose oral corticosteroids (equivalent to Prednisolone &gt; 20 mg/day)</li> </ol> |
| | 2. Intravenous pulse corticosteroids (equivalent to pulse |
| | methylprednisolone ≥ 500 mg) |
| | <ol><li>Systemic immunomodulators (include biologicals, immunoglobulins and plasmapheresis)</li></ol> |
| | 4. Therapeutic high dose anticoagulation in the presence of high dose |
| | corticosteroids or immunomodulators (e.g. warfarin with target INR 3 - |
| | 4) |
| В | Moderate disease activity requiring any of the following treatment: |
| | <ol> <li>Systemic low dose oral corticosteroids (equivalent to prednisolone ≤ 20</li> </ol> |
| | mg/day) |
| | Intramuscular or intra-articular or soft tissue corticosteroids injection |
| | (equivalent to methylprednisolone < 500 mg) |
| | 3. Topical corticosteroids |
| | 4. Topical immunomodulators |
| | 5. Antimalarials or thalidomide or prasterone or acitretin |
| | 6. Symptomatic therapy (e.g. NSAIDs for inflammatory arthritis) |
| C | Mild disease |
| D | Inactive disease but previously affected |
| E | System never involved |

The following 9 systems are evaluated as follow: constitutional, mucocutaneous, neuropsychiatric, musculoskeletal, cardiorespiratory, gastrointestinal, renal, ophthalmic and haematology.

If the answer to the question "Has the subject ever had any previous involvement of this system (prior to the past 4 weeks)" is answered as No, then

the organ system is graded at E. If the answer is missing then the organ system is graded at D.

The following imputation for missing items will be used prior to determining the score for each system.

# 17.3.5.1 Imputation of missing items

For the <u>Constitutional, Cardiorespiratory, Gastrointestinal, Mucocutaneous, Musculoskeletal, Ophthalmic and Neuropsychiatric</u> system organs, the following algorithm will be used for missing items:

- Step 1: If the current involvement is "NO", the missing items will be imputed as "NOT PRESENT".
- Step2:
  - For assessments performed prior or on the first dose of study drug, the missing items will be imputed by the previous last non-missing items (therefore the baseline score will be derived using the last non-missing items across all assessments performed prior or on the first dose of study drug).
  - For post-baseline assessments, if the current involvement is "YES", the missing items will be imputed if the previous and next values are as described in Table 17-6 as well as the rules for Week 48 described further below.

Table 17-6: Constitutional, Cardiorespiratory, Gastrointestinal, Mucocutaneous, Musculoskeletal, Ophthalmic and Neuropsychiatric system organs - Imputed values for Visitx

| Visit <sub>x-1</sub> | Visit <sub>x</sub> | Visit <sub>x+1</sub> |
|---|---|---|
| Not present | Not present | Not present |
| Not present | New | Same, Improving or Worse |
| Not present | Not present | New |
| New, Same, Improving or Worse | Improving | Not present |
| New, Same, Improving or Worse | Same | Same, Improving or Worse |
| New, Same or Worse | | New |
| Improving | Not present | New |

For the <u>Hematology and Renal</u> system organs, the following algorithm will be used for missing items:

- For characters items (TTP, evidence of active hemolysis, Coombs' test positive, accelerated hypertension, nephrotic syndrome, active urinary sediment and active nephritis) items:
  - Step 1: If the current involvement is "NO", TTP will be imputed as "NOT PRESENT" and the other items will be imputed as "NO".
  - o Step 2:
    - For assessments performed prior or on the first dose of study drug, the
      missing items will be imputed by the previous last non-missing items
      (therefore the baseline score will be derived using the last non-missing
      items across all assessments performed prior or on the first dose of
      study drug).
    - For post-baseline assessments, if the current involvement is "YES", the missing items will be imputed if the previous and next values are as

described in Table 17-6 for TTP items and Table 17-7 for the other items as well as the rules for Week 48 described further below.

Table 17-7: Hematological and Renal system organs (excluding TTP) - Imputed values for Visit<sub>x</sub>

| Visit <sub>x-1</sub> | Visit <sub>x</sub> | Visit <sub>x+1</sub> |
|----------------------|--------------------|----------------------|
| Yes | Yes | Yes or No |
| No | Yes | Yes |
| No | No | No |

• For numeric items (hemoglobin (g/dL), total white cell count (x 10<sup>9</sup>/L), neutrophils (x 10<sup>9</sup>/L), lymphocytes (x 10<sup>9</sup>/L), platelets (x 10<sup>9</sup>/L), systolic blood pressure, diastolic blood pressure, urine protein-creatinine ratio (mg/mmol), creatinine (plasma/serum) (umol/L) and GFR (calculated) (mL/min/1.73 m²)), LOCF will be used. Post-baseline results will not be imputed with baseline (or pre-baseline values). If week 4 have missing results those will not be imputed if there are no unscheduled results available on the BILAG page that have been assessed after the 1<sup>st</sup> dose of study drug.

At Week 48 (or the last visit performed), the values at Week 44 (or the visit prior to the last visit performed) will be used to impute the missing values as follow:

- If the previous value is "NEW" then the missing value will be imputed with "SAME".
- If the previous value is "IMPROVING", "SAME", "WORSE" or "NOT PRESENT", the missing value will be imputed with the value from the previous visit (i.e. "SAME" if the previous visit has a value of "SAME").
- If the previous visit value is missing, no imputation will be performed.

### 17.3.5.2 Constitutional

# Category A:

Pyrexia recorded as 2 (same), 3 (worse) or 4 (new) AND

Any 2 or more of the following recorded as 2 (same), 3 (worse) or 4 (new):

Weight loss

Lymphadenopathy/splenomegaly

Anorexia

### Category B:

Pyrexia recorded as 2 (same), 3 (worse) or 4 (new) OR

Any 2 or more of the following recorded as 2 (same), 3 (worse) or 4 (new):

Weight loss

Lymphadenopathy/splenomegaly

Anorexia

BUT do not fulfil criteria for Category A

### **Category C**

Pyrexia recorded as 1 (improving) OR

One or more of the following recorded as > 0:

Weight loss

Lymphadenopathy/Splenomegaly

Anorexia

BUT does not fulfil criteria for category A or B

# **Category D**

Previous involvement

# **Category E**

No previous involvement

### 17.3.5.3 Mucocutaneous

### **Category A**

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Skin eruption - severe

Angio-oedema - severe

Mucosal ulceration - severe

Panniculitis/Bullous lupus - severe

Major cutaneous vasculitis/thrombosis

### **Category B**

Any Category A features recorded as 1 (improving) OR

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Skin eruption - mild

Panniculitis/Bullous lupus - mild

Digital infarcts or nodular vasculitis

Alopecia - severe

# **Category C**

Any Category B features recorded as 1 (improving) OR

Any of the following recorded as > 0:

Angio-oedema - mild

Mucosal ulceration - mild

Alopecia - mild

Periungual erythema/chilblains

Splinter haemorrhages

#### **Category D**

Previous involvement

### **Category E**

No previous involvement

# 17.3.5.4 Neuropsychatric

#### **Category A**

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Aseptic meningitis

Cerebral vasculitis

Demyelinating syndrome

Myelopathy

Acute confusional state

**Psychosis** 

Acute inflammatory demyelinating polyradiculoneuropathy

Mononeuropathy (single/multiplex)

Cranial neuropathy

Plexopathy

Polyneuropathy

Status epilepticus

Cerebellar ataxia

### **Category B**

Any Category A features recorded as 1 (improving) OR

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Seizure disorder

Cerebrovascular disease (not due to vasculitis)

Cognitive dysfunction

Movement disorder

Autonomic disorder

Lupus headache - severe unremitting

Headache due to raised intracranial hypertension

### **Category C**

Any Category B features recorded as 1 (improving)

### **Category D**

Previous involvement

#### **Category E**

No previous involvement

#### 17.3.5.5 Musculoskeletal

### **Category A**

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Severe Myositis

Severe Arthritis

# **Category B**

Any Category A features recorded as 1 (improving) OR

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Mild Myositis

Moderate Arthritis/Tendonitis/Tenosynovitis

# **Category C**

Any Category B features recorded as 1 (improving) OR

Any of the following recorded as > 0:

Mild Arthritis/Arthralgia/Myalgia

# **Category D**

Previous involvement

# Category E

No previous involvement

# 17.3.5.6 Cardiorespiratory

# **Category A**

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Myocarditis/Endocarditis + Cardiac failure

Arrhythmia

New valvular dysfunction

Cardiac tamponade

Pleural effusion with dyspnoea

Pulmonary haemorrhage/vasculitis

Interstitial alveolitis/pneumonitis

Shrinking lung syndrome

Aortitis

Coronary vasculitis

### **Category B**

Any Category A features recorded as 1 (improving) OR

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Pleurisy/Pericarditis

Myocarditis - mild

# Category C

Any Category B features recorded as 1 (improving)

### **Category D**

Previous involvement

# Category E

No previous involvement

# 17.3.5.7 Gastrointestinal

# **Category A**

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Peritonitis

Lupus enteritis/colitis

Intestinal pseudo-obstruction

Acute lupus cholecystitis

Acute lupus pancreatitis

# **Category B**

Any Category A feature recorded as 1 (improving) OR

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Abdominal serositis and/or ascites

Malabsorption

Protein losing enteropathy

Lupus hepatitis

### **Category C**

Any Category B features recorded as 1 (improving)

### Category D

Previous involvement

### Category E

No previous involvement

# 17.3.5.8 Ophthalmic

# **Category A**

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Orbital inflammation/myositis/proptosis

Keratitis - severe

Posterior uveitis/retinal vasculitis - severe

Scleritis - severe

Retinal/choroidal vaso-occlusive disease

Optic neuritis

Anterior ischaemic optic neuropathy

### **Category B**

Any Category A features recorded as 1 (improving) OR

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Keratitis - mild

Anterior uveitis

Posterior uveitis/retinal vasculitis - mild

Scleritis - mild

# **Category C**

Any Category B features recorded as 1 (improving) OR

Any of the following recorded as > 0:

**Episcleritis** 

Isolated cotton-wool spots (cytoid bodies)

# **Category D**

Previous involvement

#### **Category E**

No previous involvement

#### 17.3.5.9 Renal

For Proteinuria, only urine protein-creatinine ratio will be used in calculation of the grades. Abnormal laboratory values will be used for scoring only if they are due to SLE.

### Category A

# Two or more of the following providing 1, 4 or 5 is included:

- 1. Deteriorating proteinuria (severe) defined as
  - (a) urine protein-creatinine ratio > 100 mg/mmol that has not decreased (improved) by  $\ge 25\%$ ;
- 2. Accelerated hypertension
- 3. Deteriorating renal function (severe) defined as
  - (a) plasma creatinine > 130  $\mu$ mol/L and having risen to > 130% of previous value; **or**
  - (b) eGFR < 80 ml/min per 1.73 m<sup>2</sup> and having fallen to < 67% of previous value; or
  - (c) eGFR < 50 ml/min per 1.73 m², and last time was > 50 ml/min per 1.73 m² or was not measured.
- 4. Active urinary sediment
- 5. Histological evidence of active nephritis within last 3 months
- 6. Nephrotic syndrome
### **Category B**

One of the following:

- 1. One of the Category A feature
- 2. Proteinuria (that has not fulfilled Category A criteria)
  - (a) urine protein-creatinine ratio  $\geq$  50 mg/mmol that has not decreased (improved) by  $\geq$  25%; **or**
- 3. Plasma creatinine > 130  $\mu mol/L$  and having risen to  $\geq$  115% but  $\leq$  130% of previous value

# **Category C**

One of the following:

- 1. Mild/Stable proteinuria defined as
  - (a) urine protein-creatinine ratio > 25 mg/mmol but has not fulfilled criteria for Category A & B;
- 2. Rising blood pressure (providing the recorded values are > 140/90 mm Hg) which has not fulfilled criteria for Category A & B, defined as
  - (a) systolic rise of ≥ 30 mm Hg; and
  - (b) diastolic rise of ≥ 15mm Hg

### Category D

Previous involvement

# **Category E**

No previous involvement

# 17.3.5.10 Hematological

Abnormal laboratory values will be used for scoring only if they are due to SLE.

# **Category A**

Thrombotic Thrombocytopenic Purpura (TTP) recorded as 2 (same), 3 (worse) or 4 (new) **OR** 

Any of the following:

Haemoglobin < 8 g/dL

White cell count  $< 1.0 \times 10^9/L$ 

Neutrophil count  $< 0.5 \times 10^9/L$ 

Platelet count  $< 25 \times 10^9/L$ 

# **Category B**

TTP recorded as 1 (improving)  $\mathbf{OR}$ 

Any of the following:

Haemoglobin 8 - 8.9 g/dL

White cell count 1 - 1.9  $\times$  10 $^{9}/L$ 

Neutrophil count  $0.5 - 0.9 \times 10^9/L$ 

Platelet count 25 - 49 x 109/L

Evidence of active haemolysis

# **Category C**

Any of the following:

Haemoglobin 9 - 10.9 g/dL

White cell count 2 -  $3.9 \times 10^9/L$ 

Neutrophil count 1 - 1.9 x 10<sup>9</sup>/L

Lymphocyte count  $< 1.0 \times 10^9/L$ 

Platelet count 50 - 149 x 109/L

Isolated Coombs' test positive

# **Category D**

Previous involvement

# **Category E**

No previous involvement

# 17.4 SLEDAI-2K Scoring System

The SLEDAI-2K [5] is a one-page weighted scale for 24 items (seizure, psychosis, organic brain syndrome, visual disturbance, cranial nerve disorder, lupus headache, cerebrovascular accident, vasculitis, arthritis, myositis, urinary casts, haematuria, proteinuria, pyuria, rash, alopecia, mucosal ulcers, pleurisy, pericarditis, low complement, increased DNA binding, fever, thrombocytopenia, leukopenia). The manifestations felt to be most commonly contributing to disease activity are included and scored based on the presence or absence within 30 days prior to the evaluation. The score can range from 0-105 and reflects all aspects of disease activity. Results from central laboratory will be used in the SLEDAI-2K scoring by the investigator.

SLEDAI-2K weighted scoring sheet can be found below.

Enter weight in SLEDAI-2K Score column if descriptor is present at the time of the visit or in the **preceding 30 days**.

| SLEDAI 2K | | Descriptor | Definition |
|---|---|---|---|
| Weight | SCORE | | |
| 8 | | Seizure | Recent onset, exclude metabolic, infectious or drug causes. |
| 8 | _ | Psychosis | Altered ability to function in normal activity due to severe disturbance in the perception of reality. Include hallucinations, incoherence, marked loose associations, impoverished thought content, marked illogical thinking, bizarre, disorganized, or catatonic behavior. Exclude uremia and drug causes |
| 8 | | Organic brain<br>syndrome | Altered mental function with impaired orientation, memory, or other intellectual function, with rapid onset and fluctuating clinical features, inability to sustain attention to environment, plus at least 2 of the following: perceptual disturbance, incoherent speech, insomnia or daytime drowsiness, or increased or decreased psychomotor activity. Exclude metabolic, infectious, or drug causes. |
| 8 | _ | Visual<br>disturbance | Retinal changes of SLE. Include cytoid bodies, retinal hemorrhages, serous exudate or hemorrhages in the choroid, or optic neuritis. Exclude hypertension, infection, or drug causes. |
| 8 | | Cranial nerve<br>disorder | New onset of sensory or motor neuropathy involving cranial nerves. |
| 8 | | Lupus<br>headache | Severe, persistent headache; may be migrainous, but must be nonresponsive to narcotic analgesia. |
| 8 | | CVA | New onset of cerebrovascular accident(s). Exclude arteriosclerosis. |
| 8 | _ | Vasculitis | Ulceration, gangrene, tender finger nodules, periungual infarction, splinter hemorrhages, or biopsy or angiogram proof of vasqulitis. |
| 4 | | Arthritis | $\geq$ 2 joints with pain and signs of inflammation (i.e., tenderness, swelling or effusion). |

| SLEDAI 2K | | Descriptor | Definition |
|---|---|---|---|
| Weight | SCORE | | |
| 4 | | Myositis | Proximal muscle aching/weakness, associated with elevated creatine phosphokinase/aldolase or electromyogram changes or a biopsy showing myositis. |
| 4 | | Urinary casts | Heme-granular or red blood cell casts. |
| 4 | — | Hematuria | >5 red blood cells/high power field. Exclude stone, infection or other cause. |
| 4 | | Proteinuria | >0.5 gram/24 hours |
| 4 | | Pyuria | >5 white blood cells/high power field. Exclude infection. |
| 2 | | Rash | Inflammatory type rash. |
| 2 | | Alopecia | Abnormal, patchy or diffuse loss of hair. |
| 2 | | Mucosal ulcers | Oral or nasal ulcerations. |
| 2 | | Pleurisy | Pleuritic chest pain with pleural rub or effusion, or pleural thickening. |
| 2 | P | Pericarditis | Pericardial pain with at least 1 of the following:<br>rub, effusion, or electrocardiogram or<br>echocardiogram confirmation. |
| 2 | | Low<br>complement | Decrease in CH50, C3, or C4 below the lower limit of normal for testing laboratory |
| 2 | | Increased<br>DNA binding | Increased DNA binding by Farr assay above normal range for testing laboratory. |
| 1 | | Fever | >38° C. Exclude infectious cause. |
| 1 | | Thrombocytop<br>enia | <100,000 platelets / $\times 10^9 / L$ , exclude drug causes. |
| 1 | | Leukopenia | $<$ 3,000 white blood cells / $\times 10^9 / \text{L},$ exclude drug causes. |

TOTAL SCORE:

### Imputation of missing data for Baseline Score:

For assessments performed prior or on the first dose of study drug, the missing items will be imputed by the previous last non-missing items (therefore the baseline score will be derived using the last non-missing items across all assessments performed prior or on the first dose of study drug).

## **Modified SLEDAI-2K (mSLEDAI-2K):**

An mSLEDAI-2K index [6] will be derived from the standard index by omitting 1 of the standard items (low complement). An anti-IL-6R compound strongly decreases production of acute phase reactants, including complement [7, 8]. Therefore, the complement (C3/C4) values (parameters of the low complement item in the SLEDAI-2K index) may be decreased due to decreased production while effect on complement consumption (relevant for disease activity evaluation) cannot be assessed.

# mSLEDAI-2K Flare Index (mSFI):

Using the mSLEDAI-2K score [10], severe and mild/moderate flares are defined as follows. The flares will be assessed at Week 24 (i.e. from Baseline to the end of Week 24 visit window as defined in Section 17.16) and at Week 48 (i.e. from Baseline to the end of Week 48 visit window as defined in Section 17.16).

- Severe flare defined as:
  - Change from Baseline in mSLEDAI-2K > 12, or
  - New/worse central nervous system (CNS) SLE, vasculitis (captured in SLEDAI-2K), nephritis, myositis (captured in SLEDAI-2K), Platelets < 60 000, haemolytic anaemia with Haemoglobin < 7 mg/dL, requiring doubling (compared to baseline) or an increase to a dose > 0.5 mg/kg/day prednisone, or
  - Hospitalization for SLE, or
  - o Increase of Prednisone equivalent dose to a dose > 0.5 mg/kg/day, or
  - o New or increased immunosuppressive, or
  - Increase of PGA from Baseline and PGA > 83.3 (using a 100 VAS).
- · Mild/moderate flare defined as:
  - o Change from Baseline in mSLEDAI-2K ≥ 3, or
  - o New/worse skin, stomatitis, serositis, arthritis, fever, or
  - Increase in prednisone equivalent dose to a dose ≤ 0.5 mg/kg/day, or
  - o Added non-steroidal anti-inflammatory drug (NSAID)/Plaquenil, or
  - o Increase from Baseline in PGA of  $\geq$  33.3 (using a 100 VAS).

The following items of the mSFI will be derived programmatically:

- Change from Baseline in mSLEDAI-2K ≥ 3
- Change from Baseline in mSLEDAI-2K > 12,
- Prednisone Equivalent Dose > 0.5 mg/kg/day (weight will be derived from the weight assessed at the visit prior to or on the medication start date; if the weight is missing, LOCF principle will be applied; see Section 17.9 for details on how Prednisone Equivalent Dose is derived at Week 24 and Week 48),
- Increase in Prednisone Equivalent Dose to a dose ≤ 0.5 mg/kg/day,
- Added non-steroidal anti-inflammatory drug (NSAID)/Plaquenil (anti-malarial),
- Increase of PGA from Baseline and PGA > 83.3 (using a 100 VAS),
- Increase from Baseline in PGA of ≥ 33.3 (using a 100 VAS),
- New/worse skin is defined as any items (except "mucosal ulceration") recorded as 3 (worse) or 4 (new) in system "mucocutaneous" of BILAG-2004 index or new score >0 recorded or increase of score from Baseline in "rash" and "alopecia" items of SLEDAI-2K index,
- New/worse stomatitis is defined as any "Mucosal ulceration severe" or "Mucosal ulceration Mild" items recorded as 3 (worse) or 4 (new) in system "mucocutaneous" of BILAG-2004 index or new score > 0 recorded or increase of score from Baseline in "mucosal ulcers" items of SLEDAI-2K index,
- New/worse serositis is defined as any "Pleurisy/pericarditis", "Cardiac tamponade" or "Pleural effusion with dyspnoea" items recorded as 3 (worse) or 4 (new) in system 'Cardiorespiratory" of BILAG-2004 or new score > 0 recorded or increase of score from Baseline in "Pleurisy" and "Pericarditis" items of SLEDAI-2K index,

- New/worse arthritis is defined as any "Arthritis (severe)", "Arthritis (moderate)/
  Tendonitis/ Tenosynovitis" or "Arthritis (mild)/ Arthralgia/ Myalgia" items
  recorded as 3 (worse) or 4 (new) in system "Musculoskeletal" of BILAG-2004 or
  new score > 0 recorded or increase of score from Baseline in "Arthritis" item of
  SLEDAI-2K index,
- New/worse fever is defined as any "Pyrexia documented > 37.5 °C" item recorded as 3 (worse) or 4 (new) in system "constitutional" of BILAG-2004 index or new score > 0 recorded or increase of score from Baseline in "Fever" item of SLEDAI-2K index.

The following items will be medically reviewed to determine if they meet the criteria of severe mSFI flare.

- New/worse central nervous system (CNS) SLE, vasculitis (captured in SLEDAI-2K), nephritis, myositis (captured in SLEDAI-2K), Platelets < 60 000, haemolytic anaemia with Haemoglobin < 7 mg/dL, requiring doubling (compared to baseline) or > 0.5 mg/kg/day prednisone, and
- · New or increased immunosuppressive, and
- Hospitalization for SLE.

PPD Programming and Biostatistics will provide medical monitor with a listing of study drugs (restricted to immunosuppressives, anti-malarials and systemic corticosteroids with prednisone equivalent dose and changes post-Baseline) for their review (data fields will be agreed and documented in the Data Validation Manual and/or the Medical Manual). The listing will be programmed based on the analysis datasets and approved SAP. The medical monitor team will review the listings on an agreed frequency for sufficiently clean subjects. The outcome of the review will be included in subsequent delivery of the listings by PPD Programming and Biostatistics and will be used to derive flare in the analysis datasets. Prior to database lock (during soft lock process), a medical review on the final listing will be performed to confirm the subjects who experience severe flare based on the 3 criteria listed under medical review.

## 17.5 Treatment Failure Derivation Algorithm

A subject is deemed a treatment failure prior to a certain analysis visit (for example prior to week 24) if any of the following criteria are met and the corresponding date of the event is prior to the cut-off date (see Section 17.5.1).

- New or increased immunosuppressives or anti-malarials (see Section 17.5.3 and Section 17.5.4)
- Non-protocol allowed increased oral, intravenous or intramuscular corticosteroids (see Section 17.9 for selection of the corticosteroids drugs);

During blinded targeted medical review prior to database lock, the criteria above will be evaluated. The medication and corresponding start date will be identified. PPD Programming and Biostatistics will provide medical monitor with a listing of prior and concomitant medications recorded on the SLE medication page (restricted to immunosuppressives, anti-malarials and systemic corticosteroids with prednisone equivalent dose and changes post-Baseline) for their review (data fields will be agreed and documented in the Data Validation Manual and/or the Medical Manual). The listing will be programmed based on the analysis datasets and approved SAP. The medical monitor team will review the listings on an agreed frequency for clean subjects. The outcome of the review will be included in subsequent delivery of the listings by PPD Programming and Biostatistics and will be used to derive treatment failure in the analysis datasets. Prior to database lock (during soft lock process), a medical review on the final listing will be performed to confirm the subjects who are treatment failure.

#### 17.5.1Cut-off date

The cut-off date is defined as the latest of the following assessment/sample dates for the analysis visit considered. For subjects who discontinue from the study before the analysis visit considered, the cut-off date is defined as the latest of the following assessment/sample dates prior to the analysis visit considered (for example, for a subject who discontinued at Week 16 (last assessment=Week 16), the treatment failure should still be evaluated from baseline up to Week 16). In case no assessment is available and subject is still on treatment for the analysis visit considered, the cut-off date is defined as the upper bound of visit window for that visit (see Section 17.16). In case of partial start date for medications, the start date is imputed as per Section 17.15.

- BILAG-2004 assessment date for constitutional system
- BILAG-2004 assessment date for mucocutaneous system
- BILAG-2004 assessment date for neuropsychiatric system
- BILAG-2004 assessment date for musculoskeletal system
- BILAG-2004 assessment date for cardiorespiratory system
- BILAG-2004 assessment date for gastro intestinal system
- BILAG-2004 assessment date for ophthalmic system
- BILAG-2004 assessment date for renal system
- BILAG-2004 assessment date for hematological system
- SLEDAI-2K assessment date
- PGA assessment date

### 17.5.2New / Increased dose Determination

New/increase intake of steroids, immunosuppressive or anti-malarial drugs are defined as new records in the concomitant SLE medication page with either a new PT in the

• L01XC

same category or the same PT but with a total daily dose (i.e. dose times frequency) higher than the previous record of the same drug.

If an immunosuppressive, steroid or anti-malarial drug is interrupted or decreased due to an AE and re-started at the same dose as before the interruption, then it should not be considered as a treatment failure during the medical review.

# 17.5.3 Selection of Immunosuppressive Drugs:

The following ATC codes will be used to select immunosuppressive drugs from the CRF.

L04AX
 L04AA

• L04AD • L04AB • M01CX

L01AA
 L01XX

# 17.5.4 Selection of anti-malarials Drugs

The following ATC codes will be used to select anti-malarial drugs (including Plaquil) from the CRF.

P01BA

## 17.6 BILAG based Composite Lupus Assessment (BICLA)

BICLA responders are defined as subjects who meet all of the following criteria:

- BILAG-2004 normal improvement: all A scores at Baseline improved to B, C or D, and all B scores improved to C or D.
- 2. No worsening in disease activity: no new BILAG-2004 A scores and  $\leq 1$  new increase to B.
- 3. No worsening of total SLEDAI-2K score from Baseline.
- 4. No significant deterioration (< 10 % worsening from Baseline) in PGA.
- 5. No treatment failure (including the premature discontinuation from study treatment).

A subject will be deemed to be non-responder at any time point after treatment failure has been determined.

The date associated with premature discontinuation from treatment will be the date of last dose of treatment + 1 day, i.e. if criteria 1, 2, 3 and 4 are met prior to or on the date of last dose of treatment and there is no treatment failure prior to or on the date of last dose of treatment, the subject will be BICLA responder.

#### **Modified BICLA:**

A modified BICLA (mBICLA) will be derived from BICLA by using the mSLEDAI-2K instead of SLEDAI-2K.

mBICLA responders are defined as subjects who meet all of the following criteria:

- 1. BILAG-2004 normal improvement: all A scores at Baseline improved to B, C or D, and all B scores improved to C or D.
- 2. No worsening in disease activity: no new BILAG-2004 A scores and  $\leq$  1 new increase to B.
- 3. No worsening of total mSLEDAI-2K score from Baseline.
- 4. No significant deterioration (< 10 % worsening from Baseline) in PGA.
- 5. No treatment failure (including the premature discontinuation from study treatment).

A subject will be deemed to be non-responder at any time point after treatment failure has been determined.

The date associated with premature discontinuation from treatment will be the date of last dose of treatment + 1 day, i.e. if criteria 1, 2, 3 and 4 are met prior to or on the date of last dose of treatment and there is no treatment failure prior to or on the date of last dose of treatment, the subject will be mBICLA responder.

## 17.7 SLE Responder Index (SRI)

The composite index SRI enables quantification of decrease and increase in disease activity in a broad spectrum of manifestations thereby offering a comprehensive assessment of SLE disease status [9].

SRI combines advantages from three validated measurement tools:

- · SLEDAI covers global disease improvement,
- BILAG covers organ specific disease worsening or improvement, and
- PGA is used as a validity and safety net for items that were not addressed by the other two indices.

The composite SRI criteria for response are:

- SLEDAI-2K: ≥ 4 point reduction.
- BILAG-2004: no new A domain score and no more than 1 new increase to B.
- PGA: no worsening (<10% increase from Baseline).</li>

When all 3 criteria are met, the subject is a responder according to the SRI at that time point, i.e., a clinically meaningful improvement of disease is detected.

A subject will be deemed to be a non-responder at any time point after treatment failure (including the premature discontinuation from study treatment) has been determined. This criterion is also applicable for SRI-5, SRI-6, SRI-7, SRI-8 and their modified version.

# **SRI-5:**

The composite SRI-5 criteria for response are:

- SLEDAI-2K: ≥ 5 point reduction.
- BILAG-2004: no new A domain score and no more than 1 new increase to B domain score.
- PGA: no worsening (<10% increase from Baseline).

Only subjects with Baseline SLEDAI-2K  $\geq$  5 will be considered for the derivation of that endpoint.

#### **SRI-6:**

The composite SRI-6 criteria for response are:

- SLEDAI-2K: ≥ 6 point reduction.
- BILAG-2004: no new A domain score and no more than 1 new increase to B domain score.
- PGA: no worsening (<10% increase from Baseline).</li>

Only subjects with Baseline SLEDAI-2K  $\geq$  6 will be considered for the derivation of that endpoint.

## **SRI-7:**

The composite SRI-7 criteria for response are:

- SLEDAI-2K: ≥ 7 point reduction.
- BILAG-2004: no new A domain score and no more than 1 new increase to B domain score.

• PGA: no worsening (<10% increase from Baseline).

Only subjects with Baseline SLEDAI-2K  $\geq$  7 will be considered for the derivation of that endpoint.

### **SRI-8:**

The composite SRI-8 criteria for response are:

- SLEDAI-2K: ≥ 8 point reduction.
- BILAG-2004: no new A domain score and no more than 1 new increase to B domain score.
- PGA: no worsening (<10% increase from Baseline).

Only subjects with Baseline SLEDAI-2K  $\geq$  8 will be considered for the derivation of that endpoint.

#### **Modified SRI (mSRI):**

The mSRI will be assessed using the modified (excluding the low component item) version of the SLEDAI-2K as a criterion.

### mSRI-5:

The mSRI-5 will be assessed using the modified (excluding the low component item) version of the SLEDAI-2K as a criterion. Only subjects with Baseline mSLEDAI-2K  $\geq$  5 will be considered for the derivation of that endpoint.

#### **mSRI-6:**

The mSRI-6 will be assessed using the modified (excluding the low component item) version of the SLEDAI-2K as a criterion. Only subjects with Baseline mSLEDAI-2K  $\geq$  6 will be considered for the derivation of that endpoint.

#### mSRI-7:

The mSRI-7 will be assessed using the modified (excluding the low component item) version of the SLEDAI-2K as a criterion. Only subjects with Baseline mSLEDAI-2K  $\geq$  7 will be considered for the derivation of that endpoint.

## mSRI-8:

The mSRI-8 will be assessed using the modified (excluding the low component item) version of the SLEDAI-2K as a criterion. Only subjects with Baseline mSLEDAI-2K  $\geq$  8 will be considered for the derivation of that endpoint.

### 17.8 Selection of NSAIDS

The following ATC codes will be used to select NSAIDs from the SLE medication CRF page.

- M01AB
- M01AE
- M01AH
- M01AC

# 17.9 Selection of Steroids drugs and Drug Equivalence

The following ATC codes will be used to select steroids drugs from the CRF. Only systemic corticosteroids will be considered for the assessment of treatment failure. Systemic corticosteroids are corticosteroids with a route of administration of oral, intramuscular and intravenous.

H02AB

Total daily dose will be derived using the frequency and the corresponding dose recorded in CRF (i.e. if a subject takes a dose of 5 mg at a frequency of twice a day, their total daily dose will be 10 mg) and will be converted to Prednisone equivalent using the equivalence Table 17-8 below.

**Table 17-8: Prednisone Equivalence Table** 

| Glucocorticoid | Approximate equivalent dose (mg) | Conversion factor |
|---|---|---|
| Cortisone | 25 | 0.20 |
| Hydrocortisone | 20 | 0.25 |
| Methylprednisolone, | 4 | 1.25 |
| Methylprednisolone Sodium Succinate, | | |
| Methylprednisolone Acetate | | |
| Prednisolone | 5 | 1.00 |
| Prednisone | 5 | 1.00 |
| Triamcinolone | 4 | 1.25 |
| Triamcinolone Acetonide | | |
| Betamethasone | 0.70 | 7.15 |
| DIPROSPAN /00582101/ | | |
| Dexamethasone | 0.75 | 6.67 |
| Deflazacort | 6 | 0.83 |
| Meprednisone | 4 | 1.25 |

- Dixon JS. Second-line Agents in the Treatment of Rheumatic Diseases. Informa Health Care, 1991. (456).
- Meikle AW and Tyler FH. Potency and duration of action of glucocorticoids. Am J of Med 1977;63;200.
- Webb R, Singer M. Oxford Handbook of Critical Care. Oxford; New York: Oxford University Press, 2005.
- Nayak S, Acharjya B. Deflazacort versus other glucocorticoids: A comparison. Indian J Dermatol 2008;53:167-70

The total daily dose of steroids is the sum of all Prednisone equivalent doses taken by the subject on the date of the visit of interest. For example, if the subject takes steroid every other day, it will be assumed that the steroid was taken every day and the dose recorded on the CRF will be halved.

- **Week 12:** total daily dose is the sum of the Prednisone equivalent doses for all steroids that have a start date (included imputed date) prior to or on the latest assessment date for Week 12 for assessments defined in Section 17.5.1 and have a stop date on or after the same cut-off date.
- **Week 24**: total daily dose is the sum of the Prednisone equivalent doses for all steroids that have a start date (included imputed date) prior to or on the cut-off date for treatment failure at Week 24 and have a stop date on or after the same cut-off date.
- Week 48: total daily dose is the sum of the Prednisone equivalent doses for all steroids that have a start date (included imputed date) prior to or on the cut-off date for treatment failure at Week 48 and have a stop date on or after the same cut-off date.
- Week 40 to Week 48: total daily dose is the average of Prednisone equivalent doses adjusted by their duration within the period of interest (Week 40 to Week 48) for all steroids that meet one of the following conditions. The start of the Week-40-to-Week-48 period is defined as the earliest of the dates of the BILAG-2004, SLEDAI-2K and PGA assessments that fall within the Week 40 visit window. The end of theWeek-40-to-Week-48 period is defined as the cut-off date for treatment failure at Week 48 (Section 17.5.1).
  - A start date (included imputed date) prior to or on the start of the Week-40-to-Week-48 period and have a stop date on or after the end of the Week-40-to-48-period; or
  - A start date (included imputed date) between the start of the Week-40-to-Week-48 period and the end of the Week-40-to-Week-48 period; or
  - A stop date (included imputed date) between the start of the Week-40-to-Week-48 period and the end of the Week-40-to-Week-48 period.

For each steroid the daily dose (expressed as Prednisone equivalent dose) will be multiplied by the number of days within the period (week 40-48) that the subject was treated with steroid (end date of interest – start date of interest + 1) and divided by the number of days within the period (the end of the Week 40 to Week 48 period to the start of the Week 40 to Week 48 period + 1 day). The average daily doses by steroid will then be summed to get the total daily dose for each subject.

## 17.10 Medical Outcome Survey Short Form 36 (SF-36)

The SF-36 consists of 36 items that can be summarized into 8 domains: physical functioning, role limitations due to physical health problems (role-physical), bodily pain, general health, vitality, social functioning, role limitations due to emotional problems (role-emotional), and mental health. Two summary measures, the physical component summary and the mental component summary, can be derived based on these domain scores.

The domain scores for the SF-36 questionnaire will be derived based on the responses collected for the 36 questions directly in the CRF. In order to derive SF-36 domain scores based on the questionnaire, the SF-36 v2 Scoring software will be used (the handling of missing data with regards to the derivation of the domain and component score will be performed by the software). The handling and the implementation of the derived scores into the datasets will be described in the Datasets Specification document.

The following options will be selected in the software to derive the domains scores.

**Survey:** SF-26 v2 **Recall period:** 4 weeks **T-Scores:** 2009 US T-Scores

Benchmarks: None

Missing data Estimation (MDE) Method: Maximum data recovery Additional Component Scores Using Alternative Method: No

### 17.1128-Joint Count

Twenty-eight joints will be assessed separately for tenderness and swollenness (a score of 1 for a joint denotes a presence of tenderness or swollenness). The sum will be derived to create a total score (ranging from 0 to 28; where the highest score indicate all 28 joints are swollen/tender, respectively). If any joint assessment is missing, the LOCF imputation will be performed at a joint level.

## 17.12CLASI Questionnaire

The CLASI will be performed in interested sites having experience in this assessment.

The CLASI consists of two scores, i.e., one for damage and one for activity:

- Activity is scored based on erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and nonscarring alopecia.
- Damage is score based on dyspigmentation and scarring, including scarring alopecia.

Subjects are asked whether dyspigmentation due to SLE lesions usually remains visible for more than 12 months, which is considered to be permanent and resulting in doubling of the dyspigmentation score. The scores are calculated by addition of the different subscores for clinical symptoms.

The CLASI is designed as a table where the rows represent anatomical areas and the columns represent major clinical symptoms. The extent of involvement for each of the skin symptoms is documented according to specific anatomic areas taking into account the worst affected lesion within that area for each symptom.

| | activity | | dama | | |
|---|---|---|---|---|---|
| Anatomical Location | Erythema | Scale/<br>Hypertrophy | Dyspigmentation | Scarring/<br>Atrophy/<br>Pannicuitis | Anatomical Location |
| | 0-absent<br>1-pink; faint erythema<br>2-red;<br>3-dark red;<br>purple/violaceous/<br>crusted/ hemorrhagic | 0-absent;<br>1-scale<br>2-verrucous/<br>hypertrophic | 0-absent,<br>1-dyspigmentaton | 0 - absent<br>1 - scarring<br>2 - severely<br>atrophic scarring<br>or panniculitis | |
| Scalp | 3 | | | See below | Scalp |
| Ears | | | | | Ears |
| Nose (incl. malar area) | 9 7 | | | 2 | Nose (incl. malar area) |
| Rest of the face | | | 1 | | Rest of the face |
| V-area neck (frontal) | | | 1 | | V-area neck (frontal) |
| Post, Neck &/or shoulders | | | | | Post, Neck &/or shoulde |
| Chest | | | | - | Chest |
| Abdomen | | | | | Abdomen |
| Back, buttocks | 9 9 | | 1 | 4 | Back, buttocks |
| Arms | | | 1 | - | Arms |
| Hands | | | 1 | | Hands |
| Legs | | | 1 | | Legs |
| Feet | | | 1 | | Feet |
| 0-absent;<br>1-lesion or ulceration | | 0- dyspigmentation usually lasts less than<br>12 months<br>1- dyspigmentation usually lasts at least<br>12 months | | | |
| Alopecia Recent Hair loss (within the last 30 days / as 1-Yes 0-No Divide the scalp into four quits the line connecting the hi | uadrants as shown. The | | to coexist in | n one lesion, plane. The dividing line | between frontal and occip |
| Alopecia (clinically not obviously scarred) | | Scarring of the scalp (judged clinically) | | | |
| 0-absent<br>1-diffuse; non-inflammatory<br>2-focal or patchy in one quadrant;<br>3-focal or patchy in more than one quadrant | | | 0- absent<br>3- in one quadrant<br>4- two quadrants<br>5- three quadrants<br>6- affects the whole sk | ull | |

# 17.13SLICC Score

The SLICC damage score is derived by summing the individual score for each symptom/event present as described in the below scoring sheet.

| Item | Score |
|---|---|
| Ocular (either eye, by clinical assessment) | |
| Any cataract ever | 1 |
| Retinal change or optic atrophy | 1 |
| Neuropsychiatric | |
| Cognitive impairment (e.g., memory deficit, difficulty with | 1 |
| calculation, poor concentration, difficulty in spoken or written | |
| language, impaired performance level) or major psychosis | |
| Seizures requiring therapy for 6 months | l<br> |
| Cerebrovascular accident ever (score 2 if >1) | 1 (2 |
| Cranial or peripheral neuropathy (excluding optic) | 1 |
| Transverse myelitis | 1 |
| Renal | - 1 |
| Estimated or measured glomerular filtration rate <50% | 1 |
| Proteinuria ≥3.5 gm/24 hours | |
| or | 3 |
| End-stage renal disease (regardless of dialysis or transplantation) | 3 |
| Pulmonary | 3 |
| Pulmonary hypertension (right ventricular prominence, or loud P2) Pulmonary fibrosis (physical and radiograph) | î |
| Shrinking lung (radiograph) | i |
| Pleural fibrosis (radiograph) | i |
| Pulmonary infarction (radiograph) | i |
| Cardiovascular | |
| Angina or coronary artery bypass | 1 |
| Myocardial infarction ever (score 2 if >1) | 1 (2 |
| Cardiomyopathy (ventricular dysfunction) | 1 |
| Valvular disease (diastolic, murmur, or systolic murmur >3/6) | 1 |
| Pericarditis for 6 months, or pericardiectomy | 1 |
| Peripheral vascular | |
| Claudication for 6 months | 1 |
| Minor tissue loss (pulp space) | 1 |
| Significant tissue loss ever (e.g., loss of digit or limb) (score 2 if >1 | 1 (2 |
| site) | |
| Venous thrombosis with swelling, ulceration, or venous stasis | 1 |
| Gastrointestinal | |
| Infarction or resection of bowel below duodenum, spleen, liver, or | 1 (2 |
| gall bladder ever, for cause any (score 2 if >1 site) | |
| Mesenteric insufficiency | 1 |
| Chronic peritonitis | 1 |
| Stricture or upper gastrointestinal tract surgery ever | 1 |
| Musculoskeletal | |
| Muscle atrophy or weakness | ı |
| Deforming or erosive arthritis (including reducible deformities, | 1 |
| excluding avascular necrosis) | 140 |
| Osteoporosis with fracture or vertebral collapse (excluding avascular | 1 |
| necrosis) | 104.100 |
| Avascular necrosis (score 2 if >1) | 1 (2 |
| Osteomyelitis | 1 |
| Skin | :14:1 |
| Scarring chronic alopecia | 1 |
| Extensive scarring or panniculum other than scalp and pulp space | 1 |
| Skin ulceration (excluding thrombosis) for >6 months | 1 |
| Premature gonadal failure | ! |
| Diabetes (regardless of treatment) | 1.7 |
| Malignancy (exclude dysplasia) (score 2 if >1 site) | 1 (2 |

# **17.14Laboratory Parameters Precision Levels**

Table 17-9 described the precision level to be applied to the laboratory parameters in the summary statistics. Only the laboratory tests to be summarized are included in the table.

**Table 17-9: Laboratory Precision Levels** 

| Laboratory Parameter | SI Unit | Precision | LLOQ | ULOQ |
|---|---|---|---|---|
| Pro | CHEMISTRY | (raw) | | |
| Total Bilirubin | umol/mL | 2 | 2.5 | |
| Alkaline Phosphatase | U/L | 0 | 2.5 | |
| GGT | U/L | 0 | | |
| AST | U/L | 0 | | |
| ALT | U/L | 0 | | |
| Lactate Dehydrogenase | U/L | 0 | | |
| Creatine Phosphokinase | U/L | 0 | | |
| Urea | mmol/L | 2 | | |
| Total Protein | g/L | 1 | | |
| Albumin | g/L | 1 | | |
| Glucose | mmol/L | 2 | | |
| Inorganic Phosphate | mmol/L | 2 | | |
| Sodium | mmol/L | 0 | | |
| Potassium | mmol/L | 1 | | |
| Calcium | mmol/L | 2 | | |
| Chloride | mmol/L | 0 | | |
| | ID PROFILE | 0 | | |
| Total Cholesterol | mmol/L | 2 | | |
| HDL-cholesterol | mmol/L | 2 | | |
| LDL-cholesterol | mmol/L | 2 | | |
| LDL/HDL-cholesterol ratio <sup>[d]</sup> | 1 | 2 | | |
| Triglycerides | mmol/L | 2 | | |
| | EMATOLOGY | | | |
| Leukocytes (White Blood Cells) | 10 <sup>9</sup> /L | 1 | | |
| Erythrocytes (Red Blood Cells) | 10 <sup>12</sup> /L | 2 | | |
| Haemoglobin | | 0 | | |
| Haematocrit | g/L<br>% | 1 | | |
| | 10 <sup>9</sup> /L | 0 | | |
| Thrombocytes (Platelets) Absolute Lymphocytes | 10 <sup>9</sup> /L | 1 | | |
| | 10°/L | 1 | | |
| Absolute Monocytes Absolute Eosinophils | 10°/L<br>10°/L | 1 | | |
| | <del>'</del> | | | |
| Absolute Basophils | 10 <sup>9</sup> /L | 1 1 | | |
| Absolute Neutrophils | 10 <sup>9</sup> /L<br>fL | 1 | | |
| Mean Corpuscular Volume (MCV) | | | | |
| Mean Corpuscular Haemoglobin (MCH) | pg<br>g/dl | 1 1 | | |
| Mean Corpuscular Haemoglobin | g/dL | 1 | | |
| Concentration (MCHC) | AGULATION | | | |
| activated Partial Prothrombin Time | sec | 1 | | |
| (aPTT) | 300 | 1 | | |
| Prothrombin Time (PT) | sec | 1 | | |
| INR [b] | 330 | 2 | | |
| | EROLOGY | | | |
| ANA Titer | TITER | 0 | 80 | 1280 |
| β <sub>2</sub> Glycoprotein IgG | SGU U/mL | 0 | 9 | 150 |
| β <sub>2</sub> Glycoprotein IgM | SMU U/mL | 0 | 9 | 150 |
| aCL IgA | APL U/mL | 0 | 9 | 150 |
| aCL IgA | GPL U/mL | 0 | 9 | 150 |
| aCL IgM | MPL U/mL | 0 | 9 | 150 |
| LA [c] | sec | 1 | 2 | 300 |
| En · · | 350 | | | 500 |

| Laboratory Parameter | SI Unit | Precision<br>(raw) | LLOQ | ULOQ |
|---|---|---|---|---|
| | EFFICACY PARAMETERS | | | |
| Serum Creatinine | μmol/L | 1 | | |
| eGFR [a] | mL/min/1.73 m <sup>2</sup> | 1 | | |
| Proteinuria | g/mol | 1 | | |
| E | XPLORATORY BIOMARKERS | | | |
| uMCP-1 | pg/mL | 1 | 29.8 | |
| uCr | pg/mol | 1 | | |
| | PD BIOMARKERS | | | |
| sIL-6R | mg/mL | 2 | | |
| CRP | mg/L | 1 | | |
| Fibrinogen | mg/dL | 0 | | |
| anti-dsDNA [FARR] | IU/mL | 1 | 1 | |
| C3 | mg/dL | 0 | | |
| C4 | mg/dL | 0 | 6 | |
| CH50 | U | 0 | | |

<sup>[</sup>a] eGFR is derived based on the modification of the diet in renal disease (MDRD) formula, i.e. eGFR =  $175 \times (\text{Serum creatinine [mg/dL]})^{-1.154} \times (\text{Age})^{-0.203} \times (0.742 \text{ if female}) \times (1.212 \text{ if African})$ 

<sup>[</sup>b] For subjects on vitamin K antagonist only.
[c] DRVVT: Dilute Russell Viper Venom Time.

<sup>[</sup>d] Derived from LDL and HDL-cholesterol.

## 17.15 Date Imputation (medications and AEs)

#### 17.15.1 Adverse Events

Incomplete Start Date

Missing day and month

- If the year is the **same** as the year of the first dosing date, then the day and month of the first dosing date will be assigned to the missing fields.
- If the year is **prior to** the year of first dosing date, then December 31 will be assigned to the missing fields.
- If the year is **after** the year of first dosing, then January 1 will be assigned to the missing fields.

Missing day only

- If the month and year are the **same** as the year and month of first dosing date, then the first dosing date will be assigned to the missing day.
- If either the year of the partial date is **before** the year of the first dosing date or the years of the partial date and the first dosing date are the same but the month of partial date is **before** the month of the first dosing date, then the last day of the month will be assigned to the missing day.
- If either the year of the partial date is **after** the year of the first dosing date or the years of the partial date and the first dose date are the same but the month of partial date is **after** the month of the first dosing date, then the first day of the month will be assigned to the missing day.

Missing day, month, and year

• No imputation is needed, the corresponding AE will be included as TEAE if end date of AE is after the first dose date or the end date is also missing.

If the stop date is not missing, and the imputed start date is after the stop date, the start date will be imputed by the stop date.

Incomplete Stop Date

Missing day and month

• The missing day and month will be imputed as the 31st of December.

Missing day only

• The missing day will be assigned as the last day of the month.

If the imputed stop date is before the start date, then the imputed stop date will be equal to the start date.

Partially missing AE start and end dates will be imputed in the derived dataset for AEs and will only be used to derived treatment emergent flag.

#### 17.15.2 Prior/Concomitant Medications/Procedures

Partially missing start/stop dates for prior/concomitant medications and partially missing start dates for prior/concomitant procedures will be imputed in the derived dataset for prior/concomitant medications/procedures.

Partially missing prior/concomitant medication/procedure start dates will be imputed by the earliest possible date given the non-missing field(s) of the date.

Partially missing prior/concomitant medication stop dates will be imputed by the latest possible date given the non-missing field(s) of the date.

If the start date is completely missing and end date is not prior to the first dose, then the medication will be classified as both prior and concomitant. If the start date is completely missing and the end date is prior to the first dose of study drug, then the medication will be classified as prior. Medications for which the start and end dates are missing will be classified as both prior and concomitant.

For the purpose of determining treatment failure, flare and deriving Prednisone Equivalent Doses the following additional imputation rules will be implemented in the following order before the above rules are derived. Those imputation rules are only for the medications recorded on the SLE medications eCRF page.

• If the start date and the stop date of a medication are identical and only month/year are known, the start date will be imputed as the first of the month and the stop date will be imputed as the last day of the month.

If, for a patient, the stop date of a medication is partial (only month and year known) and in the same month there is a partial start date for a different medication (or dose) coded to the same preferred term, the stop date is imputed as the 14th of the month and the start date is imputed to the 15th of the month (so the medications do not overlap).

# 17.16 Analysis Visit / Visit Window

Table 17-10 provides the study day ranges to be applied to the assessment/sample collection date to derive the analysis visits. The following considerations are to be followed when deriving the analysis visits.

- All visits including unscheduled visits are used to determine the analysis visits.
- For BILAG-2004, the visit mapping will be based on the date of assessments.
- For immunogenicity, Screening and Baseline assessments will be reported separately. The CRF visit label will be used to classify the assessments.
- If there are multiple results within the same visit windows, the non-missing assessment/sample closest to the planned study day will be selected for analysis. In case of ties on the same day with time not available, the assessment linked with the CRF visit will be selected for analysis.

**Table 17-10: Visit Windows (Post-Baseline)** 

| Analysis Visit | Planned<br>Day | Efficacy | Systolic/Dias<br>tolic Blood<br>Pressure,<br>Temperature | PK | Central<br>laboratory | Direct<br>Coombs,<br>Urinalysis,<br>Immunogeni<br>city, PD | Other Safety<br>Parameters |
|---|---|---|---|---|---|---|---|
| Week 2 | 15 | | [8; 22] | [10;20] | [8; 22] | 0.077 . 2 | [8; 22] |
| Week 4 | 29 | [16; 43] | [23; 36] | [24;34] | [23; 43] | [16; 43] | [23; 36] |
| Week 6 | 43 | | [37; 50] | [38; 48] | | | [37; 50] |
| Week 8 | 57 | [44; 71] | [51; 64] | [52; 62] | [44; 71] | [44; 71] | [51; 64] |
| Week 10 | 71 | | [65; 78] | [66; 76] | | | [65; 78] |
| Week 12 | 85 | [72; 99] | [79; 99] | [80; 90] | [72; 99] | [72; 99] | [79; 99] |
| Week 16 | 113 | [100; 127] | [100; 127] | [108; 118] | [100; 127] | [100; 127] | [100; 127] |
| Week 20 | 141 | [128; 155] | [128; 155] | [136; 146] | [128; 155] | [128; 155] | [128; 155] |
| Week 24 | 169 | [156; 183] | [156; 183] | [164; 174] | [156; 183] | [156; 183] | [156; 183] |
| Week 28 | 197 | [184; 211] | [184; 211] | [192; 202] | [184; 211] | [184; 211] | [184; 211] |
| Week 32 | 225 | [212; 239] | [212; 239] | [220; 230] | [212; 239] | [212; 239] | [212; 239] |
| Week 36 | 253 | [240; 267] | [240; 267] | [248; 258] | [240; 267] | [240; 267] | [240; 267] |
| Week 40 | 281 | [268; 295] | [268; 295] | [276; 286] | [268; 295] | [268; 295] | [268; 295] |
| Week 44 | 309 | [296; 323] | [296; 323] | [304; 314] | [296; 323] | [296; 323] | [296; 323] |
| Week 48 | 337 | [324; 351] | [324; 351] | [332; 342] | [324; 351] | [324; 351] | [324; 351] |
| Follow-up | 85* | | [26; 106] | | [26; 106] | [26; 106] | [26; 106] |

#### Notes:

- For Week 2 to Week 48, Study day is calculated from the day of the first dose of study drug administration (Day 1 is the day of first administration). For Week 2 to Week 48, if the assessment /sample date is less than or equal to 25 days after the last dose of treatment, the assessment will be mapped to the corresponding analysis visit.
  - For Week 2 to Week 48, if the assessment/sample date is more than 25 days after the last dose of treatment, the assessment will be mapped to Follow-up visit.
- Early Termination visit will be flagged in listings, by adding a symbol after the Visit Name in the Analysis Visit column and associated footnote will be added.
- \* For Follow-up, the study day is based on the date of last dose (Day 1 is the day after last administration).
- For PK sampling, the samples need to be taken prior to the study drug injection.

## 17.17 Example of R code (MCP-Mod):

```
# load add-on package DoseFinding for MCP-Mod functionalities
library(DoseFinding)
# define doses to be used in models
doses <- c(0, 37.5, 75, 150, 225)
# calculate guesstimates for model parameters of set of 5 candidate models
nmodels <- 5
ndoses <- length(doses)</pre>
betascaling <- 1.2
emax1 <- guesst(d=75,p=0.8,model="emax")
logistic1 <- guesst(d=c(37.5,150),p=c(0.1,0.9),model="logistic")
beta1 <- guesst(d=c(75,150), p=c(0.9,0.7), scal=betascaling*225, dMax=37.5,
Maxd=225, model="betaMod")
beta2 <- guesst(d=c(37.5,75), p=c(0.4,0.7), scal=betascaling*225, dMax=150,
Maxd=225, model="betaMod")
# create "Mods" class object of the set of candidate models
models <- Mods(linear=NULL, emax=emax1, logistic=logistic1,
betaMod=rbind(beta1,beta2), addArqs=list(scal=betascaling*doses[ndoses]),
doses=doses, placEff=25, maxEff=25, direction="increasing")
# plot the models
plot(models)
# example mBICLA response proportion for different groups
rrObs <- c(0.2,0.316667,0.55,0.4333333,0.3833333)
# logistic regression (on logit scale) without intercept to obtain covariance matrix
logfit <- glm(rrObs~as.factor(doses)-1, family=binomial, weights=rep(60,5))</pre>
# optimum contrast
contMat <- optContr(models, w=1)</pre>
muHat <- coef(logfit)
S <- vcov(logfit)
# multiple contrast test from the optimal trend contrasts
mcpModTest <- MCTtest(doses, rrObs, S=S, models=models, type="general")
# t-statistics with adjusted p-values
mcpModTest$tStat
# Calculate the functions for the candidate models using pre-specified parameters
qfit <- MCPMod(doses, rrObs, S=S, models=models, type = "general", Delta = 0.2,
selModel = "aveAIC")
# create a sequence of dose values used to predict the response for a range of dose
sq <- seq(0,max(doses),length=11)</pre>
# get predicted values for this sequence of doses
pred <- predict(gfit, doseSeq=sq, predType="Is-means")</pre>
```

Statistical Analysis Plan, Final Version 1.0 Date Issued: 28FEB2018

# pull out weights from model object
modWeights <- gfit\$selMod</pre>

# model averaged predictions - this is just matrix multiplication of predicted values from each significant candidate model multiplied by weights pred <- do.call("cbind", pred)%\*%modWeights

# 17.18Search criteria for adverse events of special interest

Search criteria for AESIs are either MedDRA PT clusters or SMOs. The SMOs and the individual PTs for the PT clusters are provided below.

#### **Infections**

Abdominal abscess Abdominal hernia gangrenous Abdominal infection Abdominal lymphadenopathy Abdominal sepsis

Abdominal wall abscess

Abdominal wall

infection

Abortion infected

Abscess

Abscess bacterial Abscess fungal Abscess intestinal Abscess jaw Abscess limb Abscess neck Abscess of external auditory meatus Abscess of eyelid Abscess of salivary

gland Abscess oral Abscess rupture Abscess soft tissue Abscess sweat gland Acanthamoeba

Acanthamoeba keratitis

Acariasis Acarodermatitis

infection

Acid fast bacilli infection Acinetobacter

bacteraemia Acinetobacter infection

Acinetobacter test

positive Acne pustular Acquired

immunodeficiency

syndrome

Acrodermatitis chronica

atrophicans Actinomyces test

positive

Actinomycosis Actinomycotic abdominal infection

Actinomycotic pulmonary infection Actinomycotic skin

infection

Acute endocarditis Acute focal bacterial

nephritis

Acute haemorrhagic conjunctivitis Acute hepatitis B Acute hepatitis C Acute HIV infection Acute pulmonary histoplasmosis Acute sinusitis Acute tonsillitis

Adenopathy syphilitic

Adenoviral conjunctivitis Adenoviral

Adenoiditis

haemorrhagic cystitis Adenoviral hepatitis

Adenoviral upper respiratory infection Adenovirus infection Adenovirus test

Adenovirus test

positive Adiponectin increased

abscess

Administration site Administration site

cellulitis

Administration site

infection

Adrenal gland abscess

Adrenal gland tuberculosis Adrenalitis

Aeromona infection Aeromonas test

positive

African trypanosomiasis AIDS cholangiopathy AIDS dementia

complex

AIDS related complex

AIDS related complication AIDS retinopathy Air-borne transmission Alcaligenes infection Allescheriosis Alopecia syphilitic Alpha haemolytic

streptococcal infection Alphaviral infection Alphavirus test

Alphavirus test positive Alternaria infection Alveolar osteitis American

trypanosomiasis Amniotic cavity

infection

Amniotic infection syndrome of Blane

Amoeba test

Amoeba test positive

Amoebiasis

Amoebic brain abscess

Amoebic colitis Amoebic dysentery Amoebic lung abscess Amoebic skin ulcer Anal abscess

Anal candidiasis Anal chlamydia

infection

Anal fistula infection

Anal fungal infection Anal infection Anal tinea

Angina gangrenous Angiostrongylus

infection

Anicteric leptospirosis

Anisakiasis Anogenital warts Anorectal cellulitis Anorectal human

papilloma virus

infection

Anorectal infection Anorectal infection

bacterial Anthrax Anthrax sepsis

Antifungal treatment

Antimicrobial susceptibility test Antimicrobial susceptibility test intermediate Antimicrobial susceptibility test susceptibility test susceptibility test susceptibility test

resistant Antimicrobial susceptibility test

sensitive

Aortic aneurysm

syphilitic

Aortitis salmonella Aortitis syphilitic Aphthovirus test

positive

Apical granuloma Appendiceal abscess

**Appendicitis** 

Appendicitis perforated Application site abscess

Application site cellulitis

Application site folliculitis Application site infection

Application site pustules Arachnoiditis Arboviral infection Arbovirus test positive Arenaviral

haemorrhagic fever Arenavirus test positive

Argentine

haemorrhagic fever Arteriosclerotic

gangrene

Arteriovenous fistula

site infection

Arteriovenous graft site

abscess

Arteriovenous graft site

infection

Arteritis infective Arthritis bacterial

Arthritis fungal Arthritis gonococcal Arthritis helminthic

Arthritis infective

Arthritis reactive Arthritis rubella Arthritis salmonella

Arthritis viral

Arthropod infestation Arthropod-borne

disease Ascariasis Aspergilloma Aspergillosis oral Aspergillus infection Aspergillus test

Aspergillus test positive Astrovirus test positive

Asymptomatic bacteriuria

Asymptomatic HIV

infection

Asymptomatic viral

hepatitis

Atypical mycobacterial

infection

Atypical mycobacterial lower respiratory tract

infection

Atypical mycobacterial

lymphadenitis

Atypical mycobacterial

pneumonia Atypical mycobacterium pericarditis Atypical

mycobacterium test

positive

Atypical pneumonia Avian influenza Babesiosis

Bacillary angiomatosis Bacillus bacteraemia Bacillus infection Bacillus test positive

Bacteraemia Bacterascites Bacterial abscess

central nervous system

Bacterial allergy

Bacterial dacryocystitis Bacterial diarrhoea Bacterial disease

carrier

Bacterial food poisoning

Bacterial infection Bacterial iritis

Bacterial labyrinthitis Bacterial pericarditis Bacterial prostatitis Bacterial pyelonephritis

Bacterial rhinitis
Bacterial sepsis
Bacterial test

Bacterial test positive Bacterial toxaemia Bacterial tracheitis Bacterial translocation Bacterial vaginosis

Bacteriuria
Bacteriuria in
pregnancy
Bacteroides
bacteraemia

Bacteroides infection Bacteroides test

positive

Balamuthia infection Balanitis candida Balanoposthitis Balanoposthitis infective

Balantidiasis Bartholin's abscess

Bartholin's abscess
Bartonella test positive

Bartonellosis

Bed bug infestation Beta haemolytic streptococcal infection Bifidobacterium

infection

Bifidobacterium test

positive Bile culture

Bile culture positive Biliary abscess Biliary sepsis

Biliary tract infection Biliary tract infection

bacterial

Biliary tract infection cryptosporidial Biliary tract infection

fungal

Biliary tract infection

helminthic

Biliary tract infection

viral

BK virus infection

Black piedra

Bladder candidiasis Bladder diverticulitis Blastocystis infection

Blastomycosis Blebitis Blepharitis Blister infected Blood bactericidal

activity

Blood beta-D-glucan

abnormal

Blood beta-D-glucan

decreased

Blood beta-D-glucan

increased Blood culture

Blood culture positive Blood HIV RNA

Blood HIV RNA below

assay limit Blood HIV RNA decreased Blood HIV RNA increased Body tinea

Bolivian haemorrhagic

fever

Bone abscess

Bone tuberculosis Borderline leprosy Bordetella infection Bordetella test

Bordetella test positive Borrelia infection

Borrelia test

Borrelia test positive

Botryomycosis Botulism

Boutonneuse fever Bovine pustular stomatitis virus

infection

Bovine tuberculosis Brain abscess Brain empyema Breast abscess

Breast cellulitis Breast discharge

infected

Bronchiectasis

Bronchiolitis Bronchitis

Bronchitis bacterial Bronchitis fungal Bronchitis haemophilus

Bronchitis moraxella

Bronchitis pneumococcal Bronchitis viral

Bronchoalveolar lavage

abnormal

Bronchopneumonia Bronchopulmonary aspergillosis

Bronchopulmonary

aspergillosis allergic

Bronchoscopy abnormal Brucella sepsis Brucella test

Brucella test positive

Brucellosis Bubonic plague Bulbar poliomyelitis Bullous impetigo Burkholderia cepacia

complex infection Burkholderia cepacia

complex sepsis

Burkholderia gladioli

infection

Burkholderia infection Burkholderia mallei

infection Burkholderia

pseudomallei infection Burkholderia test

positive Burn infection Bursitis infective Bursitis infective staphylococcal

Calicivirus test positive

Campylobacter gastroenteritis Campylobacter infection

Campylobacter sepsis Campylobacter test

positive

Candida cervicitis

Candida

endophthalmitis
Candida infection
Candida nappy rash
Candida osteomyelitis
Candida pneumonia
Candida retinitis
Candida sepsis
Candida test

Candida test positive

Candiduria Capillariasis Capillaritis Capnocytophaga

infection

Capnocytophaga test

positive Carbuncle

Cardiac granuloma Cardiac infection Cardiac valve abscess

Cardiac valve vegetation

Cardiovascular syphilis

Carditis

Cat scratch disease Catheter culture Catheter culture

positive

Catheter site abscess

Catheter site cellulitis
Catheter site infection
Catheter site pustule
Catheter site warmth
Cavernous sinus
thrombosis
Cellulitis
Cellulitis enterococcal

Cellulitis enterococcal
Cellulitis gangrenous
Cellulitis laryngeal
Cellulitis of male
external genital organ
Cellulitis orbital
Cellulitis pasteurella
Cellulitis pharyngeal
Cellulitis staphylococcal
Cellulitis streptococcal
Central nervous system
abscess

Central nervous system enteroviral infection Central nervous system fungal infection Central nervous system

infection

Central nervous system inflammation

Central nervous system viral infection
Cerebral aneurysm ruptured syphilitic
Cerebral aspergillosis
Cerebral fungal

infection

Cerebral malaria Cerebral sarcoidosis Cerebral septic infarct Cerebral toxoplasmosis

Cervicitis

Cervicitis gonococcal Cervicitis human papilloma virus

Cervicitis mycoplasmal Cervicitis streptococcal

Cervicitis trichomonal Cervix warts Cestode infection

Chancroid Chest wall abscess Chikungunya virus

infection

Chlamydia test

Chlamydia test positive Chlamydial cervicitis Chlamydial infection Chlamydial pelvic inflammatory disease Cholangitis infective Cholecystitis infective

Cholera

Cholesteatoma

Cholesterol granuloma Choriomeningitis lymphocytic

Chorioretinitis
Choroid tubercles

Choroiditis

Chromoblastomycosis
Chronic gastritis
Chronic hepatitis
Chronic hepatitis B
Chronic hepatitis C
Chronic pulmonary
histoplasmosis
Chronic recurrent

multifocal osteomyelitis

Chronic sinusitis
Chronic tonsillitis
Citrobacter infection
Citrobacter sepsis

positive

Clitoris abscess Clonorchiasis Clostridial infection

Citrobacter test

Clostridium bacteraemia Clostridium colitis Clostridium difficile

colitis

Clostridium difficile

infection

Clostridium difficile

sepsis

Clostridium test Clostridium test

positive

CNS ventriculitis Coccidioides encephalitis Coccidioidomycosis

Colitis herpes Colon gangrene Colonic abscess Colorado tick fever Colorado tick fever virus test positive Colostomy infection Community acquired

infection

Condyloma latum Congenital condyloma

Congenital cytomegalovirus

infection

Congenital hepatitis B

infection

Congenital herpes simplex infection Congenital HIV

infection

Congenital infection Congenital malaria Congenital pneumonia Congenital rubella

infection

Congenital syphilis Congenital syphilitic

encephalitis

Congenital syphilitic

meningitis

Congenital syphilitic osteochondritis Congenital toxoplasmosis

Congenital tuberculosis Congenital varicella

infection

Congo-Crimean haemorrhagic fever Conjunctivitis

Conjunctivitis bacterial

Conjunctivitis chlamydial Conjunctivitis

gonococcal neonatal

Conjunctivitis tuberculous Conjunctivitis viral Corneal abscess

Corneal endotheliitis
Corneal infection
Corona virus infection
Coronavirus test

positive

infection Corynebacterium sepsis Corynebacterium test

Corynebacterium

Corynebacterium test positive Cow pox

Coxiella infection Coxiella test positive Coxsackie carditis Coxsackie endocarditis Coxsackie myocarditis Coxsackie pericarditis Coxsackie viral disease

of the newborn Coxsackie viral infection

Coxsackie virus test Coxsackie virus test

positive

Cranial nerve infection Creutzfeldt-Jakob

disease Cronobacter bacteraemia

Cronobacter infection Cronobacter necrotising

enterocolitis Cronobacter test

positive

Cross infection Croup infectious

Cryptococcal cutaneous

infection

Cryptococcal fungaemia Cryptococcosis Cryptococcus test Cryptococcus test

positive

Cryptosporidiosis

infection CSF culture

CSF culture positive CSF immunoglobulin G

index **CSF** 

leukocyte/erythrocyte

**CSF** 

leukocyte/erythrocyte

ratio increased

CSF measles antibody

positive

CSF virus identified CSF virus no organisms

observed Culture Culture cervix

Culture cervix positive

Culture positive Culture stool

Culture stool positive

Culture throat

Culture throat positive Culture tissue specimen

Culture tissue specimen positive

Culture urine

Culture urine positive

Culture wound

Culture wound positive Cutaneous anthrax

Cutaneous

coccidioidomycosis Cutaneous Iarva

migrans Cutaneous leishmaniasis Cutaneous sporotrichosis

Cutaneous tuberculosis

Cyclitis

Cyclosporidium infection

Cystitis

Cystitis bacterial Cystitis erosive Cystitis escherichia

Cystitis glandularis Cystitis gonococcal Cystitis haemorrhagic

Cystitis helminthic Cystitis interstitial

Cystitis klebsiella Cystitis noninfective

Cystitis pseudomonal Cystitis radiation Cystitis ulcerative

Cystitis viral Cytomegalovirus chorioretinitis

Cytomegalovirus colitis

Cytomegalovirus

duodenitis Cytomegalovirus

enteritis

Cytomegalovirus enterocolitis Cytomegalovirus

gastritis

Cytomegalovirus gastroenteritis Cytomegalovirus gastrointestinal

infection

Cytomegalovirus

hepatitis

Cytomegalovirus

infection

Cytomegalovirus mononucleosis Cytomegalovirus mucocutaneous ulcer Cytomegalovirus myelomeningoradiculiti

Cytomegalovirus myocarditis Cytomegalovirus oesophagitis Cytomegalovirus pancreatitis Cytomegalovirus pericarditis Cytomegalovirus

syndrome

Cytomegalovirus test Cytomegalovirus test

positive

Cytomegalovirus urinary tract infection Cytomegalovirus

viraemia

Dacryoadenitis

acquired

Dacryocanaliculitis Dacryocystitis Deltaretrovirus test

positive Demodicidosis Dengue fever Dental caries Dental fistula Dental gangrene

Dermatitis infected
Dermatomyositis
Dermatophytosis
Dermo-hypodermitis
Device related infection
Device related sepsis
Diabetic foot infection
Diabetic gangrene
Diaphragmatic hernia

gangrenous Diarrhoea infectious

Diarrhoea infectious neonatal Diphtheria

Diphtheria carrier Diphyllobothriasis Direct infection transmission Disseminated cryptococcosis Disseminated cytomegaloviral

infection
Disseminated
tuberculosis
Diverticulitis
Douglas' abscess
Dracunculiasis
Dural abscess

Dysentery
Ear infection
Ear infection bacterial
Ear infection fungal
Ear infection

staphylococcal
Ear infection viral
Ear lobe infection
Ear tuberculosis

Ebola disease Ebola Reston virus

infection

Ebola virus test positive Echinococciasis Echo virus infection Echovirus test

Echovirus test positive

Ecthyma

Eczema herpeticum
Eczema impetiginous
Eczema infected
Eczema vaccinatum
Ehrlichia test

Ehrlichia test positive Elephantiasis nostras

verrucosa

Embolic pneumonia Empedobacter brevis

infection

Empedobacter test

positive

Emphysematous cholecystitis

Emphysematous

cystitis

Emphysematous pyelonephritis Empyema Encephalitis

Encephalitis allergic Encephalitis australia Encephalitis brain stem Encephalitis california

Encephalitis cytomegalovirus Encephalitis eastern

equine

Encephalitis enteroviral Encephalitis fungal

Encephalitis haemorrhagic

Encephalitis influenzal Encephalitis Japanese B Encephalitis lethargica

Encephalitis
meningococcal
Encephalitis mumps
Encephalitis post

immunisation Encephalitis post

measles

Encephalitis post

varicella

Encephalitis protozoal Encephalitis rickettsial Encephalitis toxic Encephalitis venezuelan

equine

Encephalitis viral Encephalitis western

equine

Encephalomyelitis Encephalomyelitis

rubella

End stage AIDS

Endemic syphilis Endocarditis

Endocarditis bacterial Endocarditis candida

Endocarditis enterococcal

Endocarditis gonococcal

Endocarditis haemophilus

Endocarditis helminthic

Endocarditis histoplasma Endocarditis meningococcal Endocarditis pseudomonal

Endocarditis Q fever Endocarditis rheumatic

Endocarditis staphylococcal Endocarditis syphilitic Endocarditis viral

Endometritis

Endometritis bacterial Endometritis decidual

Endometritis decidade
Endometritis
gonococcal
Endophthalmitis
Endotoxaemia
Endotoxic shock
Enteritis infectious
Enteritis necroticans

Enterobacter bacteraemia

Enterobacter infection

Enterobacter pneumonia

Enterobacter sepsis Enterobacter test

positive
Enterobacter
tracheobronchitis
Enterobiasis
Enterococcal
bacteraemia

Enterococcal infection Enterococcal sepsis Enterococcus test

positive

Enterocolitis AIDS
Enterocolitis bacterial
Enterocolitis fungal

Enterocolitis helminthic Enterocolitis infectious Enterocolitis viral Enterovirus infection Enterovirus test Enterovirus test positive

Eosinophilia myalgia syndrome

Eosinophilic cystitis

**Ependymitis** 

Epidemic pleurodynia Epidemic polyarthritis

Epidemic typhus Epidermodysplasia

verruciformis **Epididymitis Epididymitis** blastomyces

Epididymitis mumps

**Epididymitis** tuberculous **Epididymitis** ureaplasmal Epididymo-orchitis

gonococcal **Epiglottitis** 

Epiglottitis haemophilus Epiglottitis obstructive Epstein-Barr viraemia Epstein-Barr virus

antibody

Epstein-Barr virus antibody positive

Epstein-Barr virus antigen positive Epstein-Barr virus associated lymphoma Epstein-Barr virus

associated

lymphoproliferative

disorder

Epstein-Barr virus

infection

Epstein-Barr virus test Epstein-Barr virus test

positive

Erosive balanitis

Eruptive

pseudoangiomatosis

Erysipelas Erysipeloid Erysipelothrix infection Erysipelothrix test

positive

Erythema induratum Erythema infectiosum Erythema migrans

Erythrasma Escherichia bacteraemia

Escherichia infection Escherichia

pyelonephritis Escherichia sepsis

Escherichia test

positive

Escherichia urinary tract infection Escherichia vaginitis Eubacterium infection

Exanthema subitum

Exserohilum infection

External ear cellulitis Extradural abscess Extrapulmonary tuberculosis

Eye abscess Eve infection Eye infection bacterial

Eye infection

chlamydial

Eye infection fungal Eye infection gonococcal

Eye infection helminthic

Eye infection intraocular Eye infection staphylococcal

Eye infection syphilitic Eye infection

toxoplasmal Eye infection viral

Eyelid boil Eyelid folliculitis Eyelid infection Faecal-oral transmission of

infection

Fallopian tube abscess Fascial infection

**Fascioliasis** Fasciolopsiasis Febrile infection Female genital tract

tuberculosis Femoral hernia gangrenous **Filariasis** 

Filariasis lymphatic Filovirus infection Filovirus test positive Flavivirus infection Flavivirus test positive

Flavobacterium infection

Flavobacterium test

positive

Flea infestation **Folliculitis** Foot and mouth

disease

Francisella test positive

Fungaemia

Fungal abscess central

nervous system Fungal cystitis Fungal endocarditis Fungal infection Fungal labyrinthitis Fungal oesophagitis Fungal paronychia Fungal peritonitis Fungal retinitis Fungal rhinitis

Fungal sepsis Fungal skin infection

Fungal test

Fungal test positive Fungal tracheitis Fungating wound

**Funisitis Furuncle** 

Fusarium infection Fusobacterium infection Fusobacterium test

positive

Gallbladder abscess Gallbladder empyema

Gangrene

Gangrene neonatal Gangrenous balanitis Gardnerella infection Gardnerella test

positive

Gas gangrene
Gastric infection
Gastric ulcer
helicobacter
Gastritis bacterial
Gastritis fungal
Gastritis helminth

Gastritis helminthic Gastritis herpes

Gastritis viral
Gastroenteritis
Gastroenteritis
adenovirus
Gastroenteritis
aerobacter
Gastroenteritis
aeromonas
Gastroenteritis

astroviral Gastroenteritis bacillus

Gastroenteritis bacterial Gastroenteritis

caliciviral Gastroenteritis clostridial Gastroenteritis

cryptococcal Gastroenteritis cryptosporidial Gastroenteritis enteroviral

Gastroenteritis Escherichia coli Gastroenteritis norovirus

Gastroenteritis paracolon bacillus Gastroenteritis proteus

Gastroenteritis pseudomonas Gastroenteritis rotavirus

Gastroenteritis salmonella Gastroenteritis sapovirus

Gastroenteritis shigella

Gastroenteritis staphylococcal

Gastroenteritis vibrio Gastroenteritis viral Gastroenteritis yersinia Gastrointestinal

anthrax

Gastrointestinal bacterial infection Gastrointestinal

candidiasis

Gastrointestinal fungal

infection Gastrointestinal gangrene Gastrointestinal

infection Gastrointestinal

mucosal necrosis Gastrointestinal

necrosis

Gastrointestinal protozoal infection Gastrointestinal viral

infection

Generalised vaccinia Genital abscess

Genital candidiasis

Genital herpes Genital herpes simplex Genital herpes zoster

Genital infection Genital infection

bacterial

Genital infection female Genital infection fungal Genital infection

helminthic

Genital infection male Genital infection viral

Genital tract inflammation Genitourinary chlamydia infection Genitourinary tract

gonococcal infection Genitourinary tract

infection
Genotype drug
resistance test
Genotype drug
resistance test

abnormal Genotype drug

resistance test positive Geotrichum infection Gerstmann Straussler Scheinker syndrome Gianotti-Crosti

syndrome Giardia test

Giardia test positive

Giardiasis

Gingival abscess

Gingivitis Gliosis

Gnathostomiasis Gonococcal pelvic inflammatory disease

Gonorrhoea

Gradenigo's syndrome

Graft infection Gram stain

Gram stain positive Granuloma inguinale Granulomatous dermatitis

Granulomatous liver

disease

Granulomatous pneumonitis Groin abscess Groin infection

Group B streptococcus

neonatal sepsis
Guillain-Barre
syndrome
Gynaecological
chlamydia infection
H1N1 influenza
Haematoma infection

Haemophilus bacteraemia

Haemophilus infection Haemophilus sepsis Haemophilus test

positive

Haemorrhagic fever Haemorrhagic fever with renal syndrome Haemorrhoid infection Hand-foot-and-mouth

disease

Hantaviral infection Hantavirus pulmonary

infection

Hantavirus test positive

**HBV-DNA** polymerase

increased

Helicobacter gastritis Helicobacter infection

Helicobacter sepsis Helicobacter test

Helicobacter test

positive

Helminthic infection Henipavirus test

positive

Hepatic amoebiasis

Hepatic candidiasis Hepatic cyst infection

Hepatic echinococciasis Hepatic infection

Hepatic infection

bacterial

Hepatic infection fungal

Hepatic infection helminthic

Hepatic infiltration eosinophilic Hepatic necrosis

Hepatitis Hepatitis A

Hepatitis A antibody Hepatitis A antibody

abnormal

Hepatitis A antibody

positive

Hepatitis A antigen

positive

Hepatitis A virus test Hepatitis A virus test

positive

Hepatitis acute Hepatitis B

Hepatitis B antibody

Hepatitis B antibody abnormal

Hepatitis B antibody

positive

Hepatitis B antigen Hepatitis B antigen

positive

Hepatitis B core

antibody

Hepatitis B core antibody positive

Hepatitis B core antigen

Hepatitis B core antigen positive

Hepatitis B DNA assay

Hepatitis B DNA assay

positive

Hepatitis B DNA decreased

Hepatitis B DNA increased

Hepatitis B e antibody

Hepatitis B e antibody

positive

Hepatitis B e antigen Hepatitis B e antigen

positive

Hepatitis B surface

antibody

Hepatitis B surface

antibody positive Hepatitis B surface

antigen

Hepatitis B surface antigen positive Hepatitis B virus test Hepatitis B virus test

positive Hepatitis C

Hepatitis C antibody Hepatitis C antibody

positive

Hepatitis C RNA Hepatitis C RNA

decreased

Hepatitis C RNA fluctuation Hepatitis C RNA increased

Hepatitis C RNA

positive

Hepatitis C virus test Hepatitis C virus test

positive

Hepatitis chronic active

Hepatitis chronic persistent

Hepatitis D Hepatitis D antibody Hepatitis D antibody

positive

Hepatitis D antigen Hepatitis D antigen

positive

Hepatitis D RNA Hepatitis D RNA

positive

Hepatitis D virus test Hepatitis D virus test

positive Hepatitis E

Hepatitis E antibody Hepatitis E antibody

abnormal

Hepatitis E antibody

positive

Hepatitis E antigen Hepatitis E antigen

positive

Hepatitis E virus test

positive Hepatitis F

Hepatitis fulminant

Hepatitis G Hepatitis H

Hepatitis infectious Hepatitis infectious mononucleosis Hepatitis mumps Hepatitis neonatal Hepatitis non-A non-B Hepatitis non-A non-B

non-C

Hepatitis post transfusion

Hepatitis syphilitic Hepatitis toxoplasmal

Hepatitis viral Hepatitis viral test Hepatitis viral test

positive

Hepatitis virus-

associated nephropathy Hepatobiliary infection

Hepatosplenic candidiasis

Hernia gangrenous

Herpangina

Herpes dermatitis Herpes oesophagitis Herpes ophthalmic Herpes pharyngitis Herpes sepsis Herpes simplex

Herpes simplex colitis
Herpes simplex DNA test positive Herpes simplex encephalitis Herpes simplex

gastritis Herpes simplex hepatitis Herpes simplex meningitis Herpes simplex meningoencephalitis

Herpes simplex meningomyelitis Herpes simplex

necrotising retinopathy

Herpes simplex oesophagitis

Herpes simplex otitis

externa

Herpes simplex pharyngitis Herpes simplex pneumonia

Herpes simplex sepsis

Herpes simplex

serology

Herpes simplex serology positive Herpes simplex virus conjunctivitis neonatal Herpes simplex visceral Herpes virus infection

Herpes zoster Herpes zoster cutaneous disseminated Herpes zoster disseminated

Herpes zoster infection

neurological Herpes zoster meningitis Herpes zoster meningoencephalitis Herpes zoster meningomyelitis

Herpes zoster necrotising retinopathy Herpes zoster oticus

Herpes zoster pharyngitis

Heterophyiasis Hirudiniasis

Histiocytic necrotising lymphadenitis Histoplasmosis Histoplasmosis

cutaneous Histoplasmosis disseminated HIV antibody

HIV antibody positive

HIV antigen

HIV antigen positive HIV associated nephropathy

HIV cardiomyopathy

HIV carrier HIV enteropathy HIV infection HIV infection CDC

category A

HIV infection CDC

category B

HIV infection CDC

category C

HIV infection CDC

Group I

HIV infection CDC

Group II

HIV infection CDC

Group III

HIV infection CDC

group IV

HIV infection CDC

Group IV subgroup A HIV infection CDC

Group IV subgroup B HIV infection CDC

Group IV subgroup C1 HIV infection CDC Group IV subgroup C2

HIV infection CDC Group IV subgroup D HIV infection CDC Group IV subgroup E

HIV infection WHO clinical stage I HIV infection WHO

clinical stage II HIV infection WHO

clinical stage III

HIV infection WHO clinical stage IV HIV peripheral neuropathy HIV test

HIV test positive HIV tropism test HIV wasting syndrome Hookworm infection

Hordeolum

HTLV test positive HTLV-1 carrier HTLV-1 test positive HTLV-2 test positive Human anaplasmosis Human ehrlichiosis Human herpes virus 6

serology

Human herpes virus 6 serology positive Human herpes virus 8

test positive

Human herpesvirus 6

infection

Human herpesvirus 7

infection

Human herpesvirus 8

infection Human

immunodeficiency virus

transmission

Human papilloma virus

test

Human papilloma virus

test positive

Human polyomavirus

infection

Human rhinovirus test

positive Human T-cell

lymphocytic virus type

II infection Human T-cell lymphotropic virus

infection Human T-cell

lymphotropic virus type

I infection Hydrocele male infected

Hymenolepiasis Hypopyon

Iatrogenic infection Ileal gangrene Immune reconstitution inflammatory syndrome associated tuberculosis **Impetigo** Implant site abscess Implant site cellulitis Implant site infection Implant site pustules Incision site abscess Incision site cellulitis Incision site infection Incisional hernia gangrenous Inclusion body myositis Inclusion conjunctivitis Inclusion conjunctivitis neonatal Indeterminate leprosy Indirect infection transmission Induced abortion infection Infantile septic granulomatosis Infected bites Infected bunion Infected cyst Infected dermal cyst Infected fistula Infected lymphocele Infected naevus Infected neoplasm Infected seroma Infected skin ulcer Infected varicose vein Infection Infection in an immunocompromised Infection masked Infection parasitic Infection protozoal Infection reactivation Infection susceptibility increased Infection transmission via personal contact Infection via vaccinee

Infectious colitis

Infectious crystalline keratopathy Infectious disease carrier Infectious iridocyclitis Infectious mononucleosis Infectious pleural effusion Infectious thyroiditis Infective aneurysm Infective aortitis Infective chondritis Infective corneal ulcer Infective episcleritis Infective exacerbation of bronchiectasis Infective exacerbation of chronic obstructive airways disease Infective gastroduodenitis Infective glossitis Infective iritis Infective mesenteric panniculitis Infective myositis Infective periostitis Infective pulmonary exacerbation of cystic fibrosis Infective spondylitis Infective tenosynovitis Infective thrombosis Infective uveitis Infestation Influenza Influenza A virus test Influenza A virus test positive Influenza B virus test Influenza B virus test positive Influenza C virus test positive Influenza virus test Influenza virus test positive Infusion site abscess Infusion site cellulitis Infusion site infection Infusion site pustule

Inguinal hernia gangrenous Injection site abscess Injection site cellulitis Injection site infection Injection site joint infection Injection site pustule Instillation site abscess Instillation site infection Instillation site pustules Intervertebral discitis Intestinal fistula infection Intestinal gangrene Intestinal tuberculosis Intrauterine infection Iridocyclitis Iritis Isosporiasis Japanese spotted fever JC virus granule cell neuronopathy JC virus infection JC virus test JC virus test positive Jejunal gangrene Joint abscess Joint tuberculosis Kaposi's sarcoma AIDS related Kaposi's varicelliform eruption Kawasaki's disease Keratitis Keratitis bacterial Keratitis fungal Keratitis interstitial Keratitis viral Keratoconjunctivitis measles Keratosis gonococcal Kerion Kidney infection Klebsiella bacteraemia Klebsiella infection Klebsiella sepsis Klebsiella test positive Kuru **Kyasanur Forest** 

disease

Laryngitis

Labyrinthitis
Lacrimal sac cellulitis
Lactobacillus infection
Lactobacillus test
positive

Laryngitis bacterial Laryngitis fungal Laryngitis viral Laryngotracheitis

obstructive
Lassa fever
Latent syphilis
Latent tuberculosis
Legionella infection
Legionella test

Legionella test positive

Leishmaniasis Lemierre syndrome Lentivirus test positive Lepromatous leprosy

Leprosy

Leptospira test positive

Leptospirosis

Leptotrichia infection Leuconostoc infection

Lice infestation

Ligneous conjunctivitis

Lineal gingival erythema Lip infection Listeria encephalitis

Listeria sepsis Listeria test positive

Listeriosis
Liver abscess
Lobar pneumonia
Localised infection
Lochial infection

Louping ill

Lower respiratory tract

infection

Lower respiratory tract infection bacterial Lower respiratory tract

infection fungal

Lower respiratory tract

infection viral Ludwig angina Lung abscess Lung infection Lung infection pseudomonal Lupus encephalitis Lupus vulgaris Lyme disease

Lymph gland infection Lymph node abscess

Lymph node tuberculosis

Lymphadenitis bacterial Lymphadenitis fungal

Lymphadenitis helminthic

Lymphadenitis viral Lymphangitis Lymphogranuloma

venereum

Lyssavirus test positive

Malaria

Malaria antibody test Malaria antibody test

positive

Malarial myocarditis Male genital tract

tuberculosis Malignant syphilis Marburg disease

Marburg virus test positive Mastitis

Mastitis bacterial Mastitis fungal

Mastitis postpartum Mastoid abscess Mastoid empyema

Mastoiditis Measles

Measles antibody Measles antibody

positive

Measles post vaccine Mediastinal abscess

Mediastinitis

Meibomian gland

discharge Meibomianitis

Meningitis Meningitis aseptic Meningitis aspergillus

Meningitis bacterial Meningitis borrelia

Meningitis candida

Meningitis chemical Meningitis coccidioides Meningitis coxsackie

viral

Meningitis cronobacter
Meningitis cryptococcal
Meningitis echo viral
Meningitis enterococcal
Meningitis enteroviral
Meningitis eosinophilic
Meningitis eosinophilic
Meningitis fungal
Meningitis fungal
Meningitis fungal
Meningitis haemophilus
Meningitis herpes
Meningitis histoplasma
Meningitis leptospiral
Meningitis listeria

meningococcal Meningitis mumps Meningitis neonatal Meningitis

Meningitis pneumococcal

Meningitis salmonella

Meningitis staphylococcal

Meningitis

Meningitis streptococcal Meningitis toxoplasmal

Meningitis trypanosomal

Meningitis tuberculous

Meningitis viral Meningococcal bacteraemia

Meningococcal carditis Meningococcal infection Meningococcal sepsis Meningoencephalitis

adenoviral

Meningoencephalitis

amoebic

Meningoencephalitis

bacterial

Meningoencephalitis

helminthic

Meningoencephalitis herpes simplex

neonatal

Meningoencephalitis

herpetic

Meningoencephalitis

viral

Meningomyelitis herpes Mesenteric abscess

Mesenteritis
Metagonimiasis
Metapneumovirus

infection

Methylobacterium

infection

Microbiology test Microbiology test

abnormal

Micrococcal sepsis Micrococcus infection Micrococcus test

positive

Microsporidia infection Microsporum infection Middle ear operation Middle East respiratory

syndrome

Miliary pneumonia Milker's nodules Minimum inhibitory concentration

Minor cognitive motor

disorder

Molluscipoxvirus test

positive

Molluscum contagiosum

Monkeypox Mononucleosis heterophile test Mononucleosis heterophile test positive

Mononucleosis syndrome

Moraxella infection Moraxella test positive Morbillivirus test

positive

Morganella infection Morganella test positive

Mucocutaneous candidiasis Mucocutaneous leishmaniasis Mucosal infection

Mumps

Mumps antibody test

Mumps antibody test

positive

Mumps deafness
Murine typhus
Murray Valley
encephalitis
Muscle abscess
Muscular sarcoidosis

Mycetoma mycotic

Mycobacterial disease

Mycobacterial infection

Mycobacterium
peritonitis
Mycobacterium
abscessus infection
Mycobacterium avium
complex immune
restoration disease
Mycobacterium avium

complex infection
Mycobacterium
chelonae infection
Mycobacterium
fortuitum infection

Mycobacterium kansasii

infection

Mycobacterium leprae

test positive Mycobacterium marinum infection Mycobacterium test

Mycobacterium test positive

Mycobacterium tuberculosis complex

est

Mycobacterium tuberculosis complex

test positive Mycobacterium ulcerans infection Mycoplasma genitalium

infection

Mycoplasma infection Mycoplasma test Mycoplasma test

positive Mycoplasmal postabortal fever Mycoplasmal

postpartum fever

Mycotic corneal ulcer

Mycotic

endophthalmitis Mycotoxicosis

Myelitis

Myelitis transverse

Myiasis

Myocardiac abscess

Myocarditis

Myocarditis bacterial Myocarditis helminthic Myocarditis infectious

Myocarditis meningococcal Myocarditis mycotic Myocarditis post

infection

Myocarditis septic Myocarditis syphilitic

Myocarditis toxoplasmal Myometritis Myositis

Myositis ossificans Myositis-like syndrome

**Myringitis** 

Myringitis bullous Naegleria infection Nail bed infection Nail bed infection

bacterial

Nail bed infection

fungal

Nail bed infection viral

Nail candida Nail infection

Nairovirus test positive

Nasal abscess
Nasal candidiasis
Nasal discharge
discolouration
Nasal herpes
Nasal vestibulitis
Nasopharyngitis

Natural killer cell count Natural killer cell count

decreased

Natural killer cell count

increased

Natural killer T cell

count

Natural killer T cell count decreased Natural killer T cell count increased Necrobacillosis Necrotising fasciitis Necrotising fasciitis

fungal

Necrotising fasciitis staphylococcal Necrotising fasciitis

streptococcal

Necrotising herpetic

retinopathy

Necrotising myositis Necrotising retinitis Necrotising ulcerative gingivostomatitis Necrotising ulcerative

periodontitis

Neisseria infection Neisseria test positive

Nematodiasis Neonatal candida

infection

Neonatal infection Neonatal infective

mastitis Neonatal

mucocutaneous herpes

simplex

Neonatal pneumonia Neuroborreliosis Neurocryptococcosis Neurocysticercosis Neurological infection

Neurosyphilis

Neutropenic infection Neutropenic sepsis Newcastle disease Newcastle disease virus

test positive

Nipah virus infection Nipple infection Nipple inflammation Nocardia sepsis

Nocardia test positive

Nocardiosis

Norovirus test positive North Asian tick typhus Nosocomial infection Obstetric infection

Oculoglandular syndrome Oesophageal candidiasis

Oesophageal infection

Oesophageal tuberculosis

Oesophagitis bacterial

**Omphalitis** 

Omsk haemorrhagic

fever

Onchocerciasis

Oncovirus test positive Onychomycosis

Oophoritis Ophthalmia neonatorum Ophthalmic herpes

simplex

Ophthalmic herpes

zoster

Opisthorchiasis

Opportunistic infection

Optic neuritis Optic neuritis meningococcal

Oral bacterial infection Oral candidiasis

Oral fungal infection Oral hairy leukoplakia

Oral helminthic

infection Oral herpes Oral infection Oral pustule Oral viral infection Orbital infection Orbivirus infection

Orbivirus test positive

Orchitis

Orchitis mumps

Orf

Organic dust toxic

syndrome Oro-pharyngeal aspergillosis Oropharyngeal candidiasis Oropharyngeal gonococcal infection Oropharyngitis fungal Orthobunyavirus test

positive

Orthopox virus

infection

Orthopoxvirus test

positive Osler's nodes Osteomyelitis

Osteomyelitis acute Osteomyelitis bacterial

Osteomyelitis blastomyces

Osteomyelitis chronic Osteomyelitis fungal

Osteomyelitis salmonella

Osteomyelitis viral Otitis externa

Otitis externa bacterial Otitis externa candida Otitis externa fungal Otitis externa viral

Otitis media

Otitis media acute Otitis media bacterial Otitis media chronic Otitis media fungal

Otitis media haemophilus

Otitis media moraxella

Otitis media post

measles

Otitis media viral Otorrhoea Otosalpingitis Ovarian abscess Ovarian bacterial

infection

Overgrowth bacterial Pachymeningitis Pancreas infection Pancreatic abscess Pancreatitis bacterial Pancreatitis fungal Pancreatitis helminthic Pancreatitis mumps Pancreatitis viral **Panencephalitis Panophthalmitis** Pantoea agglomerans

infection

Pantoea agglomerans

test positive

Papilloma viral infection

Paracoccidioides

infection

Paragonimiasis Parainfluenzae viral laryngotracheobronchiti

S

Parainfluenzae virus

infection

Parametric abscess Parametritis

Paraoesophageal

abscess

Parapox virus infection

Parapoxvirus test

positive

Parasite allergy
Parasite blood test
Parasite blood test

positive

Parasite cervical specimen test positive

Parasite DNA test
Parasite DNA test

positive

Parasite stool test Parasite stool test

positive

Parasite tissue

specimen test positive Parasite urine test

positive

Parasitic encephalitis Parasitic gastroenteritis Parasitic oesophagitis

Parasitic test

Parasitic test positive Paraspinal abscess Parathyroid gland

abscess

Paratyphoid fever Paravaccinia

Paravaccinia virus test

positive

Parechovirus infection

Paronychia Parophthalmia Parotid abscess

**Parotitis** 

Parvovirus B19 test

Parvovirus B19 test

positive

Parvovirus infection
Pasteurella infection
Pasteurella test positive
Pathogen resistance
Peliosis hepatis
Pelvic abscess
Pelvic infection

disease

Pelvic inflammatory disease mycoplasmal

Pelvic inflammatory

Pelvic sepsis Penicilliosis Penile abscess

Penile infection Penile wart

Peptic ulcer helicobacter

Peptostreptococcus

infection

Peptostreptococcus test

positive

Perianal streptococcal

infection

Pericarditis amoebic Pericarditis fungal Pericarditis gonococcal Pericarditis helminthic Pericarditis histoplasma

Pericarditis infective Pericarditis meningococcal Pericarditis

mycoplasmal Pericarditis rheumatic

Pericarditis syphilitic Pericarditis tuberculous Perichondritis

Pericoronitis Perihepatic abscess

Perihepatitis Perihepatitis gonococcal

Perinatal HBV infection Perinatal HIV infection Perineal abscess Perineal infection

Perinephric abscess Periodontal destruction Periodontal inflammation Periodontitis

Periorbital abscess Periorbital cellulitis Periorbital infection Peripheral nerve

infection
Periporitis
staphylogenes
Perirectal abscess
Peritoneal abscess
Peritoneal candidiasis
Peritoneal chlamydia

infection

Peritoneal tuberculosis

Peritonitis

Peritonitis bacterial Peritonitis gonococcal Peritonitis helminthic

Peritonitis pneumococcal Peritonitis syphilitic Peritonitis viral Peritonsillar abscess

Peritonsillitis

Periumbilical abscess Persistent generalised lymphadenopathy

Pertussis Petrositis

Phaehyphomycosis Pharyngeal abscess Pharyngeal chlamydia

infection Pharyngitis

Pharyngitis bacterial

Pharyngitis mycoplasmal Pharyngitis streptococcal

Pharyngoconjunctival fever of children Pharyngolaryngeal

abscess

Pharyngotonsillitis Phlebitis infective Phlebotomus fever Phlebovirus test

positive Pilonidal cyst

Pilonidal cyst congenital Pingueculitis Pinta

Pitted keratolysis

Plague Plague sepsis Plasma cell mastitis Plasmodium falciparum

infection

Plasmodium malariae

infection

Plasmodium ovale

infection

Plasmodium vivax

infection

Pleural fluid analysis Pleural infection Pleural infection

bacterial Pleurisy viral Pneumococcal bacteraemia

Pneumococcal infection Pneumococcal sepsis Pneumocystis jirovecii

infection

Pneumocystis jirovecii

pneumonia

Pneumocystis test

positive Pneumonia

Pneumonia adenoviral Pneumonia anthrax Pneumonia bacterial

Pneumonia blastomyces

Pneumonia bordetella Pneumonia chlamydial

Pneumonia cryptococcal Pneumonia cytomegaloviral

Pneumonia escherichia Pneumonia fungal

Pneumonia haemophilus

Pneumonia helminthic Pneumonia herpes viral Pneumonia influenzal Pneumonia klebsiella Pneumonia legionella Pneumonia measles Pneumonia moraxella

Pneumonia mycoplasmal

Pneumonia necrotising

Pneumonia

parainfluenzae viral

Pneumonia pneumococcal Pneumonia pseudomonal

Pneumonia respiratory

syncytial viral

Pneumonia salmonella

Pneumonia staphylococcal Pneumonia streptococcal

Pneumonia toxoplasmal Pneumonia tularaemia Pneumonia viral

Pneumonic plague Pneumovirus test

positive

Pogosta disease Polioencephalitis

Poliomyelitis Poliomyelitis post

vaccine

Poliovirus test

Poliovirus test positive Polymerase chain

reaction Polymyositis

Polyneuropathy mumps Polyomavirus test

positive Polyomavirus-

associated nephropathy

Pontiac fever Porphyromonas

infection

Porphyromonas test

positive Portal pyaemia Portal tract inflammation

Post abortion infection Post herpetic neuralgia

Post polio syndrome Post procedural

cellulitis

Post procedural infection

Post procedural pneumonia

Post procedural sepsis
Post streptococcal
glomerulonephritis
Post vaccination
autoinoculation
Post viral fatigue

syndrome

Postoperative abscess Postoperative wound

infection

Postpartum sepsis Potassium hydroxide

preparation

Potassium hydroxide preparation positive Presumed ocular histoplasmosis syndrome Primary syphilis Primary transmission Prion agent test

positive

Proctitis bacterial
Proctitis chlamydial
Proctitis fungal
Proctitis gonococcal
Proctitis herpes
Proctitis infectious
Proctitis monilial
Proctitis mycoplasmal
Progressive massive

fibrosis

Progressive multifocal leukoencephalopathy Progressive vaccinia Propionibacterium

infection

Propionibacterium test

positive

Prostate infection Prostatic abscess

Prostatitis

Prostatitis Escherichia

coli

Prostatitis gonococcal Prostatitis trichomonal Prostatitis tuberculous Prostatovesiculitis

Proteus infection Proteus test positive Protozoal corneal ulcer Pseudallescheria

infection

Pseudallescheria sepsis Pseudocroup Pseudofolliculitis

barbae

Pseudomembranous

colitis

Pseudomonal bacteraemia

Pseudomonal sepsis

Pseudomonas

aeruginosa meningitis

Pseudomonas bronchitis

Pseudomonas infection

Pseudomonas test positive

**Psittacosis** Psoas abscess Psorospermiasis Puerperal infection Puerperal pyrexia

Pulmonary echinococciasis Pulmonary mycosis Pulmonary sepsis Pulmonary syphilis

Pulmonary

trichosporonosis

Pulmonary tuberculoma Pulmonary tuberculosis

Pulpitis dental Punctate keratitis

Puncture site abscess

Puncture site discharge Puncture site infection Puncture site oedema

Purulence

Purulent discharge Purulent pericarditis

Purulent synovitis **Pyelocystitis** 

**Pyelonephritis** Pyelonephritis acute Pyelonephritis chronic Pyelonephritis fungal

**Pyelonephritis** mycoplasmal

Pyelonephritis viral Pyloric abscess

Pvoderma

Pyoderma streptococcal

Pvometra **Pyomyositis** Pyonephrosis

Pyopneumothorax

Pyospermia

Pythium insidiosum

infection Pyuria O fever

Queensland tick typhus

Rabies Raoultella

ornithinolytica infection Raoultella test positive

Rash pustular

Recrudescent typhus

Rectal abscess Rectovaginal septum

abscess

Reiter's syndrome Relapsing fever Renal abscess Renal cyst infection Renal syphilis

Renal tuberculosis

Respiratory moniliasis Respiratory papilloma

Respiratory syncytial virus bronchiolitis

Respiratory syncytial virus bronchitis

Respiratory syncytial

virus infection

Respiratory syncytial

virus test

Respiratory syncytial virus test positive

Respiratory tract infection

Respiratory tract infection bacterial Respiratory tract

infection fungal Respiratory tract infection viral

Respirovirus test positive Retinitis

Retinitis histoplasma

Retinitis viral

Retroperitoneal abscess

Retroperitoneal

infection

Retroviral infection Retroviral rebound

syndrome

Reye's syndrome Rheumatic fever Rheumatic heart

disease Rhinitis

Rhinolaryngitis Rhinoscleroma Rhinosporidiosis Rhinotracheitis Rhinovirus infection Rhodococcus infection

Rhodococcus test

positive Rickettsialpox

Rickettsioses not tick

borne Rickettsiosis Rift Valley fever Rocky mountain spotted fever Root canal infection

Roseola

Roseolovirus test

positive

Rotavirus infection Rotavirus test

Rotavirus test positive

Rubella

Rubella antibody

positive

Rubella antibody test Rubella immunity

confirmed

Rubella in pregnancy Rubella infection neurological

Rubivirus test positive Rubulavirus test

positive Salmonella bacteraemia Salmonella sepsis

Salmonella test positive

Salmonellosis

Salpingitis Salpingitis gonococcal Salpingitis tuberculous Salpingo-oophoritis Sapovirus test positive Sarcocystis infection

Scarlet fever

Scedosporium infection Schistosoma test Schistosoma test

positive

Schistosomiasis Schistosomiasis

bladder

Schistosomiasis

cutaneous

Schistosomiasis liver

Scrotal abscess Scrotal gangrene Scrotal infection Scrub typhus Sebaceous gland

infection

Secondary syphilis Secondary transmission Seminal vesicular

infection

Seminal vesiculitis Seminal vesiculitis

gonococcal Sepsis

Sepsis neonatal Sepsis pasteurella Sepsis syndrome Septic arthritis haemophilus Septic arthritis neisserial Septic arthritis staphylococcal Septic arthritis streptobacillus Septic arthritis

Septic embolus Septic encephalopathy Septic necrosis Septic phlebitis

streptococcal

Septic rash Septic shock Septic vasculitis

Seroconversion test

Seroconversion test

positive

Serology abnormal Serology positive Serology test

Serratia bacteraemia Serratia infection Serratia sepsis

Serratia test positive

Severe acute

respiratory syndrome Severe invasive

streptococcal infection Sexual transmission of

infection

Sexually transmitted

disease

Sexually transmitted

disease carrier Shigella infection

Shigella sepsis Shigella test positive

Shunt infection Sialoadenitis

Silicotuberculosis Simplex virus test

positive Sinobronchitis Sinusitis

Sinusitis aspergillus Sinusitis bacterial Sinusitis fungal

Skin bacterial infection

Skin candida Skin graft infection Skin infection Skin infection helminthic

Slit-lamp tests

abnormal

Slow virus infection Small intestinal

bacterial overgrowth Small intestine

gangrene Smallpox

Snowshoe hare virus

infection

Soft tissue infection Spermatic cord

funiculitis

Spermatic cord inflammation **Sphingomonas** 

paucimobilis infection Spinal cord abscess Spinal cord infection

Spirillary fever Spirillum test positive

Spirochaetal infection Spleen tuberculosis Splenic abscess Splenic candidiasis Splenic infection Splenic infection

bacterial

Splenic infection fungal

Splenic infection

helminthic

Splenic infection viral

Sporotrichosis

Spotted fever rickettsia

test positive Sputum culture

Sputum culture positive Sputum purulent St. Louis encephalitis Staphylococcal abscess

Staphylococcal bacteraemia Staphylococcal impetigo Staphylococcal infection Staphylococcal mediastinitis

Staphylococcal osteomyelitis

Staphylococcal parotitis

Staphylococcal pharyngitis

Staphylococcal scalded

skin syndrome

Staphylococcal sepsis Staphylococcal skin

infection Staphylococcal toxaemia

Staphylococcus test Staphylococcus test

positive

Stenotrophomonas

infection

Stenotrophomonas

sepsis

Stenotrophomonas test

positive Sternitis

Stitch abscess Stoma site abscess Stoma site candida Stoma site cellulitis Stoma site infection Stomach granuloma

Stomatococcal infection

Stomatococcus test

positive

Strawberry tonque Streptobacillary fever

Streptobacillus

infection

Streptobacillus test

positive

Streptococcal abscess

Streptococcal bacteraemia Streptococcal endocarditis

Streptococcal impetigo Streptococcal infection Streptococcal sepsis Streptococcal urinary

tract infection Streptococcus test Streptococcus test

positive

Strongyloidiasis Subacute endocarditis Subacute sclerosing panencephalitis Subarachnoid abscess

Subcutaneous abscess Subdiaphragmatic

abscess

Subperiosteal abscess

Superinfection

Superinfection bacterial

Superinfection fungal Superinfection mycobacterial Superinfection viral Suspected transmission of an infectious agent

via product

Sweat gland infection

Sweating fever Svcosis barbae

Syphilis Syphilis anal Syphilis genital **Syphilis** 

musculoskeletal Syphilitic endocarditis of heart valve Systemic candida

Systemic mycosis

Taeniasis

Tertiary syphilis Testicular abscess

Tetanus

Tetanus neonatorum Thornwaldt disease Thrombophlebitis septic

Thymus abscess Thyroglossal cyst

infection

Thyroid echinococciasis Thyroid gland abscess Thyroid tuberculosis Thyroiditis subacute Tick-borne fever Tick-borne viral encephalitis Tinea barbae

Tinea blanca

Tinea capitis Tinea cruris Tinea faciei Tinea imbricata Tinea infection Tinea manuum Tinea nigra Tinea pedis

Tinea versicolour Tongue abscess

Tonsillitis

Tonsillitis bacterial Tonsillitis fungal Tonsillitis streptococcal

Tooth abscess Tooth infection Torulopsis infection Toxic shock syndrome

Toxic shock syndrome staphylococcal

Toxic shock syndrome

streptococcal

Toxocariasis

Toxoplasma serology Toxoplasma serology

positive **Toxoplasmosis** Tracheitis

Tracheitis obstructive Tracheobronchitis Tracheobronchitis mycoplasmal

Tracheobronchitis viral Tracheostomy infection

Trachoma

Transmission of an infectious agent via

product

Transplant abscess Trematode infection

Trench fever Treponema test Treponema test false

positive

Treponema test positive **Trichiniasis** Trichomoniasis Trichomoniasis intestinal

Trichophytic granuloma

Trichophytosis

Trichosporon infection Trichostrongyliasis

Trichuriasis **Trigonitis** 

Tropical eosinophilia Tropical infectious

disease

Tropical spastic paresis

Tropical ulcer

Trypanosoma serology

positive

Trypanosomiasis Tuberculin test

Tuberculin test positive Tuberculoid leprosy Tuberculoma of central

nervous system **Tuberculosis** 

Tuberculosis bladder

Tuberculosis gastrointestinal Tuberculosis liver

Tuberculosis of central nervous system
Tuberculosis of eye
Tuberculosis of genitourinary system
Tuberculosis of intrathoracic lymph nodes
Tuberculosis of

peripheral lymph nodes Tuberculosis ureter Tuberculous abscess central nervous system Tuberculous

Tuberculous endometritis

Tuberculous laryngitis Tuberculous pleurisy

Tuberculous tenosynovitis

Tubo-ovarian abscess

Tularaemia

Type 1 lepra reaction Type 2 lepra reaction Typhoid carrier

Typhoid fever Typhus

Typhus rickettsia test Typhus rickettsia test

positive

Ulcerative keratitis Umbilical hernia gangrenous Umbilical sepsis Upper aerodigestive tract infection Upper respiratory fungal infection

Upper respiratory tract

infection

Upper respiratory tract infection bacterial Upper respiratory tract infection helminthic Urachal abscess Ureaplasma infection

Ureaplasma test positive

Ureter abscess Ureteritis

Urethral abscess Urethral carbuncle Urethral stricture post

infection Urethritis

Urethritis chlamydial Urethritis gonococcal Urethritis mycoplasmal Urethritis trichomonal Urethritis ureaplasmal

Urinary bladder

abscess

Urinary tract abscess Urinary tract infection Urinary tract infection

bacterial

Urinary tract infection

enterococcal

Urinary tract infection

fungal

Urinary tract infection

neonatal

Urinary tract infection

pseudomonal

Urinary tract infection

staphylococcal

Urinary tract infection

viral

Urinary tract inflammation Urogenital infection

bacterial

Urogenital infection

fungal
Urogenital
trichomoniasis
Urosepsis
Uterine abscess
Uterine infection

**Uveitis** 

Vaccination site

abscess

Vaccination site

cellulitis

Vaccination site discharge

Vaccination site infection

Vaccination site pallor Vaccination site pustule Vaccine breakthrough

infection

Vaccine virus shedding Vaccinia test positive

Vaccinia virus infection

Vaginal abscess
Vaginal cellulitis
Vaginal infection
Vaginitis bacterial
Vaginitis chlamydial
Vaginitis gardnerella
Vaginitis viral
Variant Creutzfeldt-

Jakob disease Varicella

Varicella post vaccine Varicella virus test Varicella virus test

positive

Varicella zoster

gastritis

Varicella zoster oesophagitis Varicella zoster pneumonia Vector-borne transmission of

infection

Veillonella infection Veillonella test positive

Vertical infection transmission

Vessel puncture site

infection

Vestibular neuronitis

Vestibulitis

Vibrio test positive

Viraemia

Viral cardiomyopathy Viral corneal ulcer Viral diarrhoea Viral epiglottitis Viral haemorrhagic

cystitis

Viral hepatitis carrier Viral infection Viral labyrinthitis

Viral load

Viral load decreased Viral load increased Viral mastitis

Viral mutation identified Viral myelitis Viral myocarditis Viral myositis

Viral oesophagitis Viral parotitis Viral pericarditis Viral pharyngitis Viral rash Viral rhinitis Viral sepsis Viral sinusitis Viral skin infection

Viral test

Viral test positive Viral titre

Viral titre decreased Viral titre increased Viral tonsillitis Viral tracheitis

Viral upper respiratory tract infection Viral uveitis Viral vasculitis Virologic failure Visceral larva migrans

Visceral leishmaniasis Vitreous abscess

Vitritis

Vorticella infection Vulval abscess Vulval cellulitis

**Vulvitis** 

Vulvovaginal candidiasis

Vulvovaginal human papilloma virus infection

Vulvovaginal mycotic

infection

Vulvovaginal warts

Vulvovaginitis

Vulvovaginitis

chlamydial Vulvovaginitis gonococcal Vulvovaginitis helminthic Vulvovaginitis streptococcal

trichomonal Waterhouse-

Friderichsen syndrome

Weil's disease

Vulvovaginitis

West Nile viral infection Whipple's disease Withdrawal hepatitis

Wound abscess

Wound contamination

Wound infection Wound infection bacterial

Atypical

Wound infection fungal

Wound infection helminthic Wound infection pseudomonas Wound infection staphylococcal

Wound infection viral

Wound sepsis

Yaws

Yaws of bone Yaws of skin Yellow fever

Yellow fever vaccineassociated neurotropic

disease

Yellow fever vaccineassociated viscerotropic

disease

Yersinia bacteraemia Yersinia infection Yersinia sepsis Yersinia test

Yersinia test positive Young's syndrome

Zoonosis

Zoonotic bacterial

infection Zygomycosis

#### **Serious infections**

Aeromona infection

Infections as defined above, assessed as serious

## **Opportunistic infections (excluding TB)**

Aeromonas test positive Allescheriosis Alternaria infection Aspergilloma Aspergillosis oral Aspergillus infection Asperaillus test Aspergillus test positive Atypical mycobacterial lower respiratory tract infection Atypical mycobacterial

pneumonia

mycobacterium pericarditis Bacillary angiomatosis BK virus infection Bronchopulmonary aspergillosis Burkholderia cepacia complex infection Burkholderia cepacia complex sepsis Burkholderia gladioli infection Burkholderia infection

Burkholderia test positive Candida endophthalmitis Candida osteomyelitis Candida pneumonia Candida retinitis Candida sepsis Capnocytophaga infection Capnocytophaga test

positive

Cerebral aspergillosis Cerebral fungal

infection

Cerebral toxoplasmosis Chronic pulmonary histoplasmosis Coccidioides encephalitis Coccidioidomycosis

Colitis herpes

Cryptococcal cutaneous

infection

Cryptococcal fungaemia Cryptococcosis

Cryptococcus test Cryptococcus test

positive Cutaneous

coccidioidomycosis Cytomegalovirus chorioretinitis

Cytomegalovirus colitis

Cytomegalovirus

duodenitis

Cytomegalovirus

enteritis

Cytomegalovirus enterocolitis Cytomegalovirus

gastritis

Cytomegalovirus gastroenteritis Cytomegalovirus gastrointestinal infection

Cytomegalovirus gastrointestinal ulcer Cytomegalovirus

hepatitis

Cytomegalovirus

infection

Cytomegalovirus mucocutaneous ulcer Cytomegalovirus

myelomeningoradiculiti

S

Cytomegalovirus myocarditis
Cytomegalovirus oesophagitis
Cytomegalovirus pancreatitis
Cytomegalovirus pericarditis

Cytomegalovirus

syndrome

Cytomegalovirus test Cytomegalovirus test

positive

Cytomegalovirus urinary tract infection

Cytomegalovirus

viraemia
Disseminated
cryptococcosis
Disseminated
cytomegaloviral

infection Encephalitis

cytomegalovirus Encephalitis fungal Endocarditis histoplasma Enterocolitis fungal

Exserohilum infection Exserohilum test Exserohilum test

positive
Eye infection
toxoplasmal
Fungaemia

Fungal abscess central

nervous system
Fungal oesophagitis
Fungal retinitis
Fungal sepsis
Fungal tracheitis
Fusarium infection

Gastritis fungal

Gastritis herpes Gastroenteritis

cryptococcal
Hepatic candidiasis
Hepatic infection fungal
Hepatitis toxoplasmal

Hepatosplenic candidiasis

Herpes oesophagitis

Herpes sepsis

Herpes simplex colitis Herpes simplex encephalitis Herpes simplex

gastritis

Herpes simplex

hepatitis

Herpes simplex meningitis Herpes simplex meningoencephalitis Herpes simplex

Herpes simplex meningomyelitis Herpes simplex

necrotising retinopathy

Herpes simplex oesophagitis Herpes simplex pneumonia

Herpes simplex sepsis Herpes simplex visceral

Herpes zoster cutaneous disseminated Herpes zoster disseminated Herpes zoster meningitis Herpes zoster

meningoencephalitis Herpes zoster meningomyelitis Herpes zoster

necrotising retinopathy

Herpes zoster
pharyngitis
Histoplasmosis
cutaneous
Histoplasmosis
disseminated
Infection in an

immunocompromised

host

JC virus granule cell neuronopathy JC virus infection JC virus test

JC virus test positive Kaposi's sarcoma AIDS

related

Kaposi's varicelliform

eruption

Listeria encephalitis Listeria sepsis

Listeria test positive Lymphadenitis fungal Meningitis aspergillus Meningitis candida Meningitis coccidioides

Meningitis cryptococcal Meningitis exserohilum Meningitis fungal Meningitis histoplasma Meningitis listeria Meningitis toxoplasmal Meningomyelitis herpes Methylobacterium infection Miliary pneumonia Mucocutaneous candidiasis Mycobacterium avium complex immune restoration disease Mycobacterium avium complex infection Mycobacterium chelonae infection Mycobacterium fortuitum infection Mycobacterium kansasii infection Myocarditis toxoplasmal Necrotising herpetic retinopathy Neurocryptococcosis Neutropenic infection Neutropenic sepsis Nocardia sepsis Nocardia test positive Nocardiosis Oesophageal candidiasis Opportunistic infection Oral candidiasis

Oral hairy leukoplakia Oro-pharyngeal aspergillosis Oropharyngeal candidiasis Oropharyngitis fungal Otitis media fungal Pancreatitis fungal Penicilliosis Pericarditis fungal Pericarditis histoplasma Phaehyphomycosis Pneumocystis jirovecii infection Pneumocystis jirovecii pneumonia Pneumocystis test

positive
Pneumonia
cryptococcal
Pneumonia
cytomegaloviral
Pneumonia herpes viral
Pneumonia toxoplasmal
Polyomavirus-

associated nephropathy Presumed ocular histoplasmosis syndrome

Progressive multifocal leukoencephalopathy Progressive vaccinia Pseudallescheria

infection Pseudallescheria sepsis Pyelonephritis fungal Respiratory moniliasis Retinitis histoplasma Retinitis viral Rhodococcus infection Rhodococcus test positive

Scedosporium infection Sepsis pasteurella Sinusitis aspergillus Sinusitis fungal Splenic candidiasis Splenic infection fungal Stomatococcal infection Stomatococcus test

positive Strongyloidiasis Systemic candida Systemic mycosis Tonsillitis fungal Upper respiratory fungal infection Varicella zoster

gastritis
Varicella zoster
oesophagitis
Varicella zoster
pneumonia
Viral oesophagitis
Yersinia sepsis

Zygomycosis Varicella zoster virus

infection

Meningitis herpes Proctitis herpes Herpes zoster oticus Herpes zoster infection

neurological

Genital herpes zoster Ophthalmic herpes

zoster

#### **Active TB**

Oral fungal infection

Adrenal gland tuberculosis
Bone tuberculosis
Choroid tubercles
Congenital tuberculosis
Conjunctivitis
tuberculous
Cutaneous tuberculosis
Disseminated
tuberculosis
Ear tuberculosis

Epididymitis
tuberculous
Erythema induratum
Exposure to
communicable disease
Extrapulmonary
tuberculosis
Female genital tract
tuberculosis
Joint tuberculosis

Lymph node
tuberculosis
Male genital tract
tuberculosis
Meningitis tuberculous
Oesophageal
tuberculosis
Pericarditis tuberculous
Peritoneal tuberculosis
Prostatitis tuberculous
Pulmonary tuberculoma

Pulmonary tuberculosis Renal tuberculosis Salpingitis tuberculous Silicotuberculosis Spleen tuberculosis Thyroid tuberculosis Tuberculoma of central nervous system Tuberculosis Tuberculosis bladder

Tuberculosis gastrointestinal Tuberculosis liver Tuberculosis of central nervous system Tuberculosis of eye Tuberculosis of genitourinary system Tuberculosis of intrathoracic lymph nodes

Tuberculosis of peripheral lymph nodes Tuberculosis ureter Tuberculous abscess central nervous system **Tuberculous** endometritis Tuberculous laryngitis Tuberculous pleurisy **Tuberculous** tenosynovitis

#### **Latent TB**

Latent tuberculosis Mycobacterium test

positive

Mycobacterium tuberculosis complex test positive

Tuberculin test false negative Tuberculin test positive

## **Herpes zoster infection**

Herpes zoster Colitis herpes Gastritis herpes Herpes oesophagitis Herpes sepsis Herpes virus infection Herpes ophthalmic Herpes pharyngitis Herpes zoster cutaneous disseminated Herpes zoster disseminated Herpes zoster

Herpes zoster meningoencephalitis Herpes zoster meningomyelitis Herpes zoster necrotising retinopathy Herpes zoster pharyngitis Meningomyelitis herpes Pneumonia herpes viral Varicella zoster gastritis Varicella zoster oesophagitis

Varicella zoster pneumonia Varicella zoster virus infection Meningitis herpes Proctitis herpes Herpes zoster oticus Herpes zoster infection neurological Genital herpes zoster Ophthalmic herpes zoster

## **Malignancies**

meningitis

Malignancies (SMQ) (Narrow)

#### Lymphoma

Malignant Lymphomas (SMQ) (Narrow)

## Hypersensitivity reactions (including anaphylaxis and angioedema)

- Hypersensitivity (SMQ) (Narrow)
- Anaphylactic reaction (SMQ) (Narrow)
- Angioedema (SMQ) (Narrow)

## **Gastrointestinal (GI) perforation**

Gastrointestinal perforation (SMQ) (Narrow)

## **Demyelinating disorders**

Demyelination (SMQ) (Narrow)

## Major adverse cardiac events (MACE)

- Ischaemic heart disease (SMQ) (Narrow)
- Central nervous system vascular disorders (SMQ) (Narrow)
- Cardiac failure (SMQ) (Narrow)

#### 17.19 Listing display/contents

All data recorded in the CRF and mapped to Study Data Tabulation Model (SDTM) except for individual scores of SF-36 and CLASI, and individual items of 28-joint Count will be displayed in data listings unless it is recorded as not done; where applicable analysis visit (i.e. visit used in the analysis) will be included in the listings. Data used in the analysis (where there are multiple results for the same analysis visit) will be flagged.

Derived parameters (for example index scores, composites endpoints, change from Baseline, etc.) used in summaries and/or analyses as well as study day will be displayed in data listings. In addition, data imputations where performed for the efficacy endpoints and Baseline records will be displayed and/or flagged in the corresponding listings.

Listings will be sorted by subject identification number, test/parameter (if applicable), date of assessment and analysis visits (if applicable) and grouped by treatment arm.

Missing/partial dates for medications and AEs will be imputed as per imputations rules described in Section 17.15 for the purpose of determining prior, concomitant, treatment failure as well as treatment emergent flags but the imputed dates will not be displayed in data listings.

Dates will be displayed as DDMMMYYYY format in the data listings. In the event of partial date, partial dates where the day only is missing will be displayed as -----YYYY and partial dates where the day and month are missing will be displayed as -----YYYY (i.e. dashes will replace the missing elements).

## 17.20 CTCAE Grades

The rules defined in Table 17-11 will be used to derive the CTCAE grades (the rules are based on the laboratory results and the numeric portion of the definition of AEs per the NCI CTCAE v4.03 guidance).

**Table 17-11: NCI CTCAE Grades** 

| Category | <b>Analyte Name</b> | CTCAE Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|---|
| Blood<br>Chemistry | Alanine<br>Aminotransferase<br>(Serum) | Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Blood<br>Chemistry | Aspartate<br>Aminotransferase<br>(Serum) | Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Blood<br>Chemistry | Creatinine<br>(Serum) | Creatinine increased | >1 - 1.5 x Baseline; >1.5 - 3.0 x Baseline; >3.0 Baseline; | | >3.0 Baseline;<br>>3.0 - 6.0 x ULN | >6.0 x ULN |
| Blood<br>Chemistry | eGFR | Chronic kidney disease | eGFR <lln -="" 60<br="">ml/min/1.73 m<sup>2</sup></lln> | eGFR 59 - 30<br>ml/min/1.73 m <sup>2</sup> | eGFR 29 - 15<br>ml/min/1.73 m <sup>2</sup> | eGFR <15<br>ml/min/1.73<br>m <sup>2</sup> |
| Blood<br>Chemistry | GGT | GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Lipid Profile | Cholesterol<br>(Serum) | Cholesterol high | >ULN - 300 mg/dL;<br>>ULN - 7.75 mmol/L | >300 - 400 mg/dL;<br>>7.75 - 10.34<br>mmol/L | >400 - 500 mg/dL;<br>>10.34 -12.92<br>mmol/L | >500 mg/dL;<br>>12.92 mmol/L |
| Hematology | Leukocytes (Blood) | Leukocytosis | - | - | >100,000/mm3 | - |
| | | White blood cell decreased | <lln -="" 3000="" mm3;<br=""><lln -="" 10^9="" 3.0="" l<="" td="" x=""><td>&lt;3000 - 2000/mm3;<br/>&lt;3.0 - 2.0 x 10^9/L</td><td>&lt;2000 - 1000/mm3;<br/>&lt;2.0 - 1.0 x 10^9 /L</td><td>&lt;1000/mm3;<br/>&lt;1.0 x 10^9/L</td></lln></lln> | <3000 - 2000/mm3;<br><3.0 - 2.0 x 10^9/L | <2000 - 1000/mm3;<br><2.0 - 1.0 x 10^9 /L | <1000/mm3;<br><1.0 x 10^9/L |
| Hematology | Lymphocytes<br>(Blood) | Lymphocyte count decreased | <lln -="" 800="" mm3;<br=""><lln -="" 0.8="" 10^9="" l<="" td="" x=""><td>&lt;800 - 500/mm3;<br/>&lt;0.8 - 0.5 x 10^9/L</td><td>&lt;500 - 200/mm3;<br/>&lt;0.5 - 0.2 x 10^9/L</td><td>&lt;200/mm3;<br/>&lt;0.2 x 10^9/L</td></lln></lln> | <800 - 500/mm3;<br><0.8 - 0.5 x 10^9/L | <500 - 200/mm3;<br><0.5 - 0.2 x 10^9/L | <200/mm3;<br><0.2 x 10^9/L |
| | | Lymphocyte count increased | - | >4000/mm3 -<br>20,000/mm3;<br>>4 - 20 10^9/L | >20,000/mm3;<br>>20 10^9/L | - |
| Hematology | Neutrophils,<br>Segmented<br>(Blood) | Neutrophil count<br>decreased | <lln -="" 1500="" mm3;<br=""><lln -="" 1.5="" 10^9="" l<="" td="" x=""><td>&lt;1500 - 1000/mm3;<br/>&lt;1.5 - 1.0 x 10^9 /L</td><td>&lt;1000 - 500/mm3;<br/>&lt;1.0 - 0.5 x 10^9 /L</td><td>&lt;500/mm3;<br/>&lt;0.5 x 10^9 /L</td></lln></lln> | <1500 - 1000/mm3;<br><1.5 - 1.0 x 10^9 /L | <1000 - 500/mm3;<br><1.0 - 0.5 x 10^9 /L | <500/mm3;<br><0.5 x 10^9 /L |
| Hematology | Platelets (Blood) | Platelet count decreased | <lln -="" 75,000="" mm3;<br=""><lln -="" 10^9="" 75.0="" l<="" td="" x=""><td>&lt;75,000 -<br/>50,000/mm3;<br/>&lt;75.0 - 50.0 x<br/>10^9/L</td><td>&lt;50,000 -<br/>25,000/mm3;<br/>&lt;50.0 - 25.0 x<br/>10^9/L</td><td>&lt;25,000/mm3;<br/>&lt;25.0 x 10^9/L</td></lln></lln> | <75,000 -<br>50,000/mm3;<br><75.0 - 50.0 x<br>10^9/L | <50,000 -<br>25,000/mm3;<br><50.0 - 25.0 x<br>10^9/L | <25,000/mm3;<br><25.0 x 10^9/L |
| PD | Fibrinogen | Fibrinogen decreased | <1.0 - 0.75 x LLN or<br><25%<br>decrease from<br>Baseline | <0.75 - 0.5 x LLN or<br>25 - <50%<br>decrease from<br>Baseline | <0.5 - 0.25 x LLN or<br>50 - <75% decrease<br>from Baseline | <0.25 x LLN or 75%<br>decrease from<br>Baseline or absolute<br>value <50 mg/dL |

## 17.21 Worst on-treatment definition

Table 17-12 display how the worst on-treatment is defined for each laboratory parameter. If a laboratory test is not listed below, no worst on-treatment summary will be provided.

**Table 17-12: Worst on-treatment** 

| Category | Analyte Name | Worst on-treatment |
|---|---|---|
| Blood Chemistry | Alanine Aminotransferase (Serum) | Maximum value |
| Blood Chemistry | Aspartate Aminotransferase (Serum) | Maximum value |
| Blood Chemistry | Creatinine (Serum) | Maximum value |
| Blood Chemistry | GGT | Maximum value |
| Blood Chemistry | Albumin (Serum) | Minimum value |
| Blood Chemistry | Alkaline Phosphatase (Serum) | Maximum value |
| Blood Chemistry | Bilirubin (Serum) | Maximum value |
| Blood Chemistry | Calcium (Serum) | Minimum value; Maximum value |
| Blood Chemistry | Creatine Kinase (Serum) | Maximum value |
| Blood Chemistry | Glucose (Serum Fasting) | Minimum value; Maximum value |
| Blood Chemistry | Potassium (Serum) | Minimum value; Maximum value |
| Blood Chemistry | Sodium (Serum) | Minimum value; Maximum value |
| Blood Chemistry | Lactate Dehydrogenase | Maximum value |
| Blood Chemistry | Urea | Maximum value |
| <b>Blood Chemistry</b> | Total Protein | Minimum value |
| <b>Blood Chemistry</b> | Chloride | Minimum value; Maximum value |
| Coagulation | Prothrombin Time | Maximum value |
| Coagulation | Activated Partial Thromboplastin Time (Plasma) | Maximum value |
| Coagulation | INR | Maximum value |
| Lipid Profile | Triglycerides (Serum) | Maximum value |
| Lipid Profile | Cholesterol (Serum) | Maximum value |
| Lipid Profile | LDL-Cholesterol | Maximum value |
| Lipid Profile | HDL- Cholesterol | Minimum value |
| Hematology | Leukocytes (Blood) | Minimum value |
| Hematology | Lymphocytes (Blood) | Minimum value |
| Hematology | Neutrophils, Segmented (Blood) | Minimum value |
| Hematology | Platelets (recorded as Thrombocytes) (Blood) | Minimum value |
| Hematology | Hemoglobin (Blood) | Minimum value; Maximum value |
| Hematology | Erythrocytes | Minimum value |
| Hematology | Haematocrit | Minimum value |
| Hematology | Absolute Monocytes | Minimum value |
| Hematology | Absolute Eosinophils | Minimum value |
| Hematology | Absolute Basophils, | Minimum value |
| Hematology | Mean Corpuscular Volume, | Minimum value; Maximum value |
| Hematology | Mean Corpuscular Haemoglobin | Minimum value |
| Hematology | Mean Corpuscular Haemoglobin Concentration | Minimum value |
| Efficacy | eGFR | Minimum value |
| Efficacy | Urine protein / creatinine ratio | Maximum value |
| PD | Fibrinogen | Minimum value |
| PD | C3 | Minimum value |
| PD | C4 | Minimum value |
| PD | CH50 | Minimum value |

## 17.22Stratified CMH 95%CI and p-value

The following formula will be used to derived the stratified CHM [15].

Using standard notation, let  $n_{ij}$  be the number of patients that enter stratum i (i=1, ..., s) and are randomized to treatment j (j=0, 1), let  $N_j = \sum_{i=1}^s n_{ij}$  denote the total number of patients on treatment j, and let  $\hat{p}_{ij}$  denote the observed success rate among patients in stratum i on treatment j.

The point estimate of the difference in success rate between the treatments, denoted as  $\delta$ , take the form  $\delta = \sum_{i=1}^{s} w_i \, \delta_i$  where  $w_i$  is the weight assigned to the stratum i,

$$w_i = \frac{(n_{i0}n_{i1})/(n_{i0+}n_{i1})}{\sum_{k=1}^{s}(n_{k0}n_{k1})/(n_{k0+}n_{k1})}$$

and

$$\delta_i = \hat{\mathbf{p}}_{i1} - \hat{\mathbf{p}}_{i0}$$

The statistic for testing  $H_0$ :  $\delta = 0$  is

$$Z_w = \frac{|\hat{\delta}_w|}{\sqrt{\{\sum_{i=1}^s w_i^2 \hat{V}_0(\delta_i)\}}}$$

Where

$$\hat{V}_0(\hat{\delta}_i) = \bar{p}_i (1 - \bar{p}_i) \left( \frac{1}{n_{i0}} + \frac{1}{n_{i1}} \right) \text{ and } \bar{p}_i = \frac{n_{i0} \hat{p}_{i0} + n_{i1} \hat{p}_{i1}}{n_{i0} + n_{i1}}$$

The confidence interval is:

$$\hat{\delta}_w \pm Z_{\alpha/2} \sqrt{\left\{\sum_{i=1}^s w_i^2 \hat{V}(\hat{\delta}_i)\right\}}$$



| Client: | Ablynx |
|---|---|
| Protocol Number: | ALX0061-C204 |
| Document Description: | Final Statistical Analysis Plan |
| SAP Title: | A Phase II Multicenter, Randomized, Double-blind, Placebo-<br>controlled, Dose-range Finding Study to Evaluate the Safety<br>and Efficacy of ALX-0061 Administered Subcutaneously in<br>Subjects with Moderate to Severe Active Systemic Lupus<br>Erythematosus |
| SAP Version Number: | Final version 1.0 |
| Effective Date: | 28-FEB-2018 |

# Author(s):

# Approved by:



SOP-BST-05ar05 Effective Date: 20 September 2017 Page 1 of 2



SOP-BST-05ar05 Effective Date: 20 September 2017 Page 2 of 2



PROTOCOL NUMBER: ALX0061-C204

| Errata | |
|---|---|
| Date | Description |
| | Site 361001 - For subject 2040196, a major Protocol Deviation is missing in the DV dataset (and final PD log on CTMS). "Kit number of study drug dispensed to subject at <u>W36</u> was not the same as kit number assigned by IRT". It has been evaluated if this issue warrants a reopening of the database and after discussion with the internal and external |
| | statistical team, it was concluded no reopening is needed but documentation on the errata list is sufficient. The conclusion was as follows: In the SAP the below is mentioned concerning deviations |
| 09/Mar/2018 | leading to subjects to be excluded from the PP analysis: "Any deviation recorded under "Kit number of study drug dispensed to subject at <specify visit=""> was not the same as kit number assigned by IRT.", where <specify visit=""> is Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 14, Week 16, Week 18, Week 20, Week 22 or Week 24 AND for which (after unblinding) the dispensed kit number corresponds to the incorrect treatment (e.g. kit number should correspond to Placebo but corresponds to ALX0061)." These missing deviations will not have an impact on the PP population as it relates to visits after Week 24.</specify></specify> |
| | Site 001025 - For subject 2040226, a major Protocol Deviation is missing in the DV dataset (and final PD log on CTMS). "Kit number of study drug dispensed to subject at <u>W34</u> was not the same as kit number assigned by IRT". |
| 00/May/2018 | It has been evaluated if this issue warrants a reopening of the database and after discussion with the internal and external statistical team, it was concluded no reopening is needed but documentation on the errata list is sufficient. The conclusion was as follows: |
| 09/Mar/2018 | In the SAP the below is mentioned concerning deviations leading to subjects to be excluded from the PP analysis: "Any deviation recorded under "Kit number of study drug dispensed to subject at <specify visit=""> was not the same as kit number assigned by IRT.", where <specify visit=""> is Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 14, Week 16, Week 18, Week 20, Week 22 or Week 24 AND for which (after unblinding) the dispensed kit number corresponds to the incorrect treatment (e.g. kit number should correspond to Placebo but corresponds to ALX0061)."</specify></specify> |



| | These missing deviations will not have an impact on the PP population as it relates to visits after Week 24. | | | | |
|---|---|---|---|---|---|
| | Site 420001- For subject 2040485, for Adverse Events 4, 5, 6, 7 and 8 the question 'Was the AE related to study drug injection?' was answered as 'Other, please specify: the exact location not known, no reaction was observed during the visit, patient informed us about mild local reaction at the next study visit, she did not remember the exact site'. | | | | |
| 13/Mar/2018 | This is present in SUPPAE as QVAL. However, as the specification is 201 characters long, QVAL has been truncated in these cases to "OTHER, PLEASE SPECIFY THE EXACT LOCATION NOT KNOWN, NO REACTION WAS OBSERVED DURING THE VISIT, PATIENT INFORMED US ABOUT MILD LOCAL REACTION AT THE NEXT STUDY VISIT, SHE DID NOT REMEMBER THE EXACT SIT" where the final "E" is missing. It has been evaluated if this issue warrants a reopening of the database and after internal discussion, it was concluded no reopening is needed but documentation on the errata list is sufficient. After all the specification is still readable. | | | | |
| | Site 052003 – For subject 2040444, Neutralizing antibody results (ISTEST='NAB0061') for two samples (Week 44 and Week 48) were erroneously reported as negative (ISORRES='NEG'). The correct values are: | | | | |
| | | Subject | Visit | Ref ID | ISORRES |
| | | 2040444 | WK44 | Q3820192910 | 0.922 |
| | | 2040444 | WK48 | Q3820323982 | 0.921 |
| 20/Sep/2018 | It has been evaluated if this issue warrants a reopening of the database, it was concluded no reopening is needed but documentation on the errata list is sufficient. Changing the NAb results for these two visits, has no impact on the NAb classification of this subject, as the subject was already classified as "PRE-DOSE NEG -POS ON TREATMENT" based on positive samples at other visits. As such, there is no impact on resulting incidence tables and no need to reopen the database. | | | | |





